**Protocol Title:** A Randomized, Phase II Study of CX-01 Combined With Standard Induction Therapy for Newly Diagnosed Acute Myeloid Leukemia

Protocol Number: CNTX-CX-01-2015-AML-1 (NCT02873338)

**Date:** 20 March 2018

# COVA-

# Cantex Pharmaceuticals, Inc.

# Protocol No.: CNTX-CX-01-2015-AML-I

A Randomized, Phase II Study of CX-01 Combined With Standard Induction Therapy for Newly Diagnosed Acute Mycloid Leukemia

**Covance Study ID: 000000146201** 

## STATISTICAL ANALYSIS PLAN

Version: Final
Date of Issue: 20 March 2018

**Author:** 

Cantex Pharmaceuticals, Inc.

Cantex Pharmaceuticals, Inc. 1792 Bell Tower Lane Weston, Florida 33326 **CovanceClinical Development Services** 

Covance Inc.
210 Carnegie Center
Princeton, New Jersey 08540-6233
USA
Suite 3.02, Level 3
Building A, 97 Waterloo Road
Macquarie Corporate Centre
Macquarie Park
New South Wales 2113, Australia

| Version: Final -,- | l)ate,of Issue: 20_Mars]d018 |
|---|---|
| Caniex Pharmaceuticals, Inc, Proto | ocol No, CNTX-CX-01 2015 AML J Covance Study ID: 000000146201 |

### **APPROVALS**

The undersigned agree that all required reviews of this document are complete, and approve this Statistical Analysis Plan as finaL Programming of the tables, figures imd listings based upon the specifications within this document can proceed.

# Covance Approval: Signarnre Printed Name/Title Contex Phormaceuticals, Inc. Approval: Daw Daw

Printed NmneiTitle

| Version: Final | | | | Date of Issue: 20 March 2018 |
|---|---|---|---|---|
| Cantey Pharmaceuticals Inc | Protocol No Ci | NTY-CY-0 I 2015 AMI | T | Covance Study ID: 00000014620 I |

# **REVIEWERS**

The following reviews of the SAP were conducted:

| Name and Title | Role | Version Last | Company/ |
|---|---|---|---|
| | | Reviewed | Ore:anization |
| | Peer Review Statistician | Draft 01 | Covance |
| | Lead Programmer | Draft 01 | Covance |
| | Senior Manager | Draft 04 | Covance |
| | (Statistics) | | |
| | Senior Medical Director | Draft 02 | Covance |
| | Project Physician | Draft 02 | Cantex |
| M.D./Chief Executive | | | |
| Officer | | | |

# **VERSION HISTORY**

| Version Number | Version Date | Summary and rational of chane:c(s) |
|----------------|--------------|------------------------------------|

# TABLE OF CONTENTS

| A | PPRO | DVALS | 2 |
|---|---|---|---|
| R | EVIE | WERS | 3 |
| V | ERSI | ON HISTORY | 3 |
| G | LOSS | SARY OF ABBREVIATIONS | 6 |
| | | STICAL ANALYSIS PLAN AMENDMENT 1 | |
| I | | URCE DOCUMENTS | |
| 2 | | OTOCOL DETAILS | |
| _ | 2.1 | Study Objectives | |
| | 2.2 | Primary Objectives | |
| | 2.3 | Secondary Ob. iectives. | |
| | 2.4 | Exploratory Objectives | |
| | 2.5 | Overall Study Design | 9 |
| | 2.6 | Sample Size and Power | 12 |
| 3 | EFF | TICACY AND SAFETY VARIABLES | 12 |
| | 3.1 | Primary Efficacy Endpoint(s) | 12 |
| | 3.2 | Secondary Efficacy Endpoints | |
| | 3.3 | Safety Endpoints | 14 |
| 4 | PHA | ARMACOKINETIC/PHARMACODYNAMIC VARIABLES | 14 |
| 5 | AN | ALYSIS POPULATIONS | 14 |
| 6 | DA | ΓA HANDLING | 15 |
| | 6.1 | Time points and Visit Windows | 15 |
| | 6.2 | Handling of Dropouts or Missing Data (where applicable) | 15 |
| 7 | STA | ATISTICALMI THODS | 16 |
| | 7.1 | General Principles | 16 |
| | 7.2 | Subject Disposition and Data Sets Analyzed | 17 |
| | 7.3 | Protocol Deviations | 17 |
| | 7.4 | Demographics and Other Baseline Characteristics | |
| | | 7.4.1 Medical History | |
| | | 7.4.2 Prior, Post treatment (anti AML) and Concomitant Medications | |
| | 7.5 | Measurements of Treatment Exposure and Study Drug Usage Rate | |
| | 7.6 | Efficacy. | |
| | | 7.6.1 Primary Efficacy Analysis | 22 |

| | | 7.6.2 | Secondary Enicacy Analysis | 22 |
|---|---|---|---|---|
| | | 7.6.3 | Sensitivity Analysis | 23 |
| | | 7.6.4 | Subgroup Analysis | 23 |
| | | 7.6.5 | Exploratory Analysis | 23 |
| | 7.7 | Safety | <i>7</i> | 23 |
| | | 7.7.1 | Adverse Events | 23 |
| | | 7.7.2 | Laboratory Evaluations | 25 |
| | | 7.7.3 | Vital Signs and ECOG performance status | 25 |
| | | 7.7.4 | Electrocardiograms | 25 |
| | 7.8 | Interi | m Analysis | 26 |
| 8 | CHA | ANGES | FROM PLANNED ANALYSES IN PROTOCOL | 26 |
| 9 | DA | ΓA ISSU | UES | 26 |
| Ю | REI | <eren< th=""><th>CES</th><th>26</th></eren<> | CES | 26 |
| 11 | APF | PENDIC | CES | 28 |
| ΑP | PEN | DIX I - | SCHEDULE OF EVENTS | 28 |
| ΛP | PFN | DIX II | TARLE FIGURE AND LISTING SHELLS | 34 |

COVANCE INC. CONFfl)ENT!AL

# **GLOSSARY OF ABBREVIATIONS**

| Abbreviation | Definition |
|---|---|
| AE | Adverse Event |
| ALT | Alanine Aminotransferase |
| AML | Acute Myeloid Leukemia |
| ANC | Absolute Neutrophil Count |
| AST | Asparlale Aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| AUC | Area Under Curve |
| BP | Blood Pressure |
| BUN | Blood Urea Nitrogen |
| CBC | Complete Blood Count |
| Cl | Confidence Interval |
| CR | Complete Remission |
| CRi | Complete Remission without recovery of neulrophils and/or platelets |
| CRp | Complete Remission without recovery of platelets |
| DSMC | Data Safety Monitoring Commillee |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| EFS | Event-Free Survival |
| FU | Follow-Up |
| INR | International Normalized Ratio |
| ITT | Intent-To-Treat |
| IWG | International Working Group |
| KM | Kaplan-Meier |
| LDH | Lactate Dehydrogenase |
| LFS | Leukemia-Free Stale/Survival |
| MUGA | Multi Gated Acquisition |
| | National Cancer Institute-Common Terminology Criteria For Adverse |
| NCI-CTCAE | Events |
| NSW | New South Wales |
| OS | Overall Survival |
| PK | Phannacokinetic |
| pp | Per Protocol |
| PT | Prolhrornbin Time |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| soc | System Organ Class |
| TBD | To Be Determined |
| TEAE | Treatment Emergent Adverse Event |
| USA | United States Of America |

Version: FinalDate of Issue: 20 March 2018Cantex Pharmaceuticals. Inc. Protocol No. CNTX-CX-0 I 2015 AML ICovance Study ID: 00000014620I

# STATISTICAL ANALYSIS PLAN AMENDMENT I

NoI applicable

COVANCE INC CONFIDENTIAL

Cantex Pharmaceuticals, Inc. Protocol No. CNTX-CX-01 2015 AML I Covance Study ID: 000000146201

### 1 SOURCE DOCUMENTS

The Statistical Analysis Plan (SAP) was wriUen based on the following documentation:

| Document | Date | Version |
|----------------------|-------------------|---------|
| Protocol | 04 February 2016 | 1.0 |
| Protocol Amendment 1 | 16 September 2016 | 2.0 |
| Protocol Amendment 2 | 13 January 2017 | 3.0 |
| eCRF | 25 July 2016 | 1.0 |
| eCRF Amendment | 16 August 2017 | 1.0.4 |

### 2 PROTOCOL DETAILS

### 2.1 Study Objectives

This randomized, phase II study of CX-01 is designed to assess the effect of adding CX-01 at one of the two different dose levels to standard induction and consolidation therapy for newly diagnosed patients with AML.

### 2.2 Primary Objectives

The primary objectives are:

- To assess whether 2-0, 3-0 desulfated heparin (CX-0 I), administered at any or all studied dose levels in conjunction with standard induction therapy for AML increases the morphologic complete remission (CR) rate based on International Working Group (IWG) criteria.
- To assess the safety and tolerability of CX-01, administered at two studied dose levels in conjunction with standard induction therapy for AML.

### 2.3 Secondary Objectives

The secondary efficacy objectives are:

To assess whether CX-01, administered at any or all studied dose levels in conjunction with standard induction and consolidation therapy fr)r AML improves:

- Event-free survival (EFS)
- Leukemia-free survival (LFS)
- Overall survival (OS)

Cantex Pharmaceuticals, Inc. Protocol No. CNTX-CX-0 I 2015 AML I Covance Study ID: 00000014620 I

- · Colliposite CR rate: incidence of CR+ CRi+CRp
- Duration of morphologic CR
- · 30-day mortality (in the induction cycle)
- 60-day mortality (in the induction cycle)
- 90-day mortality (in the induction cycle)
- Days until neutropbil recovery to? 1,000/ μL
- Days until platelet recovery to? I 00,()00/ μL

### 2.4 Exploratory Objectives

The following items are not specified in the protocol but arc still of clinical importance and will be analyzed:

- Duration of composite CR (if present)
- Days until neutrophil recovery to ? 500/ μL
- Days until platelet recovery to? 20,000/tL

### 2.5 Overall Study Design

This is an exploratory phase II, open-label, rando111ized, 111ulticenter, parallel group trial to deter111ine whether there is evidence that the addition of either or both different dose levels of CX-01 to standard induction therapy (idarubicin + cytarabine) and consolidation therapy has an additive therapeutic effect in newly diagnosed AML patients when co111pared to patients receiving standard induction che111otherapy alone.

To be eligible to participate in the study, patients 111ust meet the following criteria:

- I. Newly diagnosed, de novo or secondary, previously untreated AML
- 2. Age 60 or above
- 3. Eastern Cooperative Oncology Group (ECOG) performance status of Oto 2
- 4. Cardiac ejection fraction 45% (as determined by echocardiography or multi gated acquisition scan)
- 5. Adequate hepatic and renal function determined by the following laboratory values:
- Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) <2.5 x upper limit of normal (ULN)

Cantex Pharmaceuticals, Inc. Protocol No. CNTX-CX-01 2015 AML I Covance Study ID: 000000146201

- Bilirubin <2.5 x ULN
- Calculated creatinine clearance by Cockerofl Gault formula >30 rnL/rnin.
- 6. Able to provide informed consent and have signed an approved consent form that conforms to federal and institutional guidelines.

Patients who meet any of the following criteria will not be eligible to participate in the study:

- I. Patients with acute promyclocytic lcukernia based on the presence oft(15; I 7)(q22;q 12) as determined by karyotyping, fluorescence in situ hybridization or polymerase chain reaction
- 2. Prior chemotherapy for AML (including investigational therapy); prior hydroxyurca to control white blood cell count and a single intrathecal administration of cytarabine for CNS prophylaxis is allowed
- 3. Prior intensive chemotherapy or stem cell transplantation for treatment of myelodysplastic syndrome (prior treatment with hypornethylating agents and lenalidomide are allowed)
- 4. Presence of central nervous system leukernia
- 5. Presence of significant active infection that is not controlled in the opinion of the Investigator
- 6. Presence of significant active bleeding
- 7. History of severe congestive heart failure or other cardiac disease that contraindicates the use of anthracyclines, including idarubicin
- 8. Pre-existing liver disease (such as CHILD-Pugh Class B or C liver disease)
- 9. Renal insufficiency which rnight adversely affect schedule and dose of therapy with cytarabine as well as rnanagement of tumor lysis syndrome
- I0. History of drug addiction within the last 6 months
- II. Known history of positive Hepatitis 13 surface antigens
- 12. Known history of positive test for Human Imrnunodeficiency Virus antibodies
- 13. Psychiatric or neurologic conditions that could compromise patient safety or compliance, or interfere with the ability to give proper informed consent
- 14. History of other active malignant disease within the past 3 years, other than cured basal cell carcinoma of the skin, cured in situ carcinoma of the cervix, or localized prostate cancer that has received definitive therapy. Such prostate cancer patients who are receiving hormonal therapy are eligible
- 15. Patients receiving any form of anticoagulant therapy (heparin flushes for IV catheter permitted)
- 16. Presence of a known bleeding disorder or coagulation abnormality (including but not limited to a PTT >40 seconds) or any condition that requires maintenance of platelet counts at 50,000/"tL or higher
- 17. Pregnant or breast feeding patients
- 18. Patients of childbearing potential not using adequate contraception.

Approximately 75 patients will be randomized in a I: I: I ratio to one of the following study treatment groups:


Cantex Pharmaceuticals, Inc. Protocol No. CNTX-CX-0 I 2015 AML I Covance Study ID: 00000014620 I

- Group I: Idarubicin + Cytarabine, OR
- Group 2: Idarubicin + Cylarabine plus lower dose CX-01 (0.125 mg/kg/hour), OR
- Group 3: Idarubicin + Cytarabine plus higher dose CX-0 I (0.25 mg/kg/hour)

Eligible patients who meet the inclusion criteria and do not meet any of the exclusion criteria and have provided informed consent will be enrolled in the study. Each patient will participate in the study for approximately 18 months from the time of informed consent through final study contact, or until they withdraw from the study or the study is terminated by the Sponsor.

Overall survival data will be collected every 3 months until death or until the end of study by the investigational sites. The end of study will occur approximately 18 months afler the last patient is randomized. Overall survival data will be collected every 3 months until death or until the end of study by the investigational sites. The end of study will occur approximately 18 months afler the last patient is randomized.

A Data and Safety Monitoring Commiltee (DSMC) will meet periodically to review the safety of the study (see Section 6.6.5 of protocol). Details describing the DSMC process and procedures will be outlined in a separate DSMC Charter.

Adverse events (AEs) will be collected from time of informed consent and continue until 30 days after the last study treatment is administered. Longer follow-up and collection of AEs may be required for patients that do not have an absolute neutrophil count (ANC) recovery within 42 days (i.e., until the recovery or the reason for no recovery is diagnosed) after the last induction or consolidation cycle.

A flow diagram of the study design is shown in Figure 2---1.

Cantex Pharmaceuticals, Inc. Protocol No. CNTX-CX-0 I 2015 AML I Covance Study ID: 00000014620 I



Abbreviations: AML=acute mycloid leukemia

Note: It is expected that approximately 90 patients will be screened to identify 75 patients for randomization.

### 2.6 Sample Size and Power

A total of 25 evaluable patients per arm will provide 71.8% power fi:ir each test comparing a dose with control via a Fisher's exact test at I-sided alpha •0.15 to detect a difference between a control proportion 0.55 and an experimental dose proportion 0.80; these tests will be conducted in a fixed sequence: higher dose versus control first and lower dose versus control second, with the second test considered exploratory (failed) if the first test fails.

### 3 EFFICACY AND SAFETY VARIABLES

### 3.1 Primary Efficacy Endpoint(s)

The primary endpoint is the rate of patients in each treatment group achieving morphological CR based on IWG criteria during the induction and re-induction phases  $O\Gamma$  the treatment. Morphologic CR is defined as ANC >1000/;tL, platelet count>100,000/ $\mu$ L, <5% blasts in an bone marrow aspirate sample, no blasts with Auer rods, and no evidence of extramedullary disease (see Appendix A of protocol). Note that a patient is only considered to have achieved morphologic CR if this is documented on or after 21 days from date of randomization and not superseded by a subsequent data entry within 42 days of randomization that indicates treatment failure or progressive disease or persistent disease as indicated by >5% blasts in a bone marrow aspirate sample.

Cantex Pharmaceuticals, Inc. Protocol No. CNTX-CX-01 2015 AML I Covance Study ID: 000000146201

### 3.2 Secondary Efficacy Endpoints

- Event Free Survival (EFS)
  - o Event-free survival (from date of randomization) is measured from the date of randomization until treatment failure (e.g., failure to achieve composite complete morphological remission during the induction or re-induction phase of the study lasting up to 60 days, relapse from CR, or death from any cause, whichever occurs first).
- Leukemia-Free State (LFS)
  - o Leukemia-free survival is only assessed in patients who achieve composite CR and is measured from the date ofleukemia-free state until disease relapse or patient death from any cause, whichever occurs first.
- Overall Survival (OS)
  - o Overall survival is measured from the date of randomization until death from any cause.
- Composite Complete Remissions (CR) rate
  - Complete remission rate includes CR, (on or after 21 days from date of randomization) and CRi and CRp (either need to be on or after 21 days from date of randomization) as defined by IWG criteria (Appendix A in the protocol) during the induction and reinduction phases of treatment. If a patient achieves a composite CR, but followed by PD or treatment failure from day 21 to 42, then the patient did not achieve a composite CR and should be considered a treatment failure.
- Duration of morphologic CR
  - o Duration of morphologic complete response is measured from the achievement of CR to detection of relapse. A relapse is defined as progressive disease or death from clinical disease progression
- Duration of composite CR (if available)
  - o Duration of composite complete response is measured from the date of achievement of composite CR to detection of relapse. A relapse is defined as either progressive disease or death from clinical disease progression.
- 30-day, 60-day and 90-day mortality
  - o Thirty-day, 60-day, and 90-day mortality are the rate of death during 30 days, 60 days, and 90 days, respectively, from the first day of induction treatment.
- Neutrophil and Platelet Recovery
  - o Time to neutrophil recovery (from date of randomization) is measured from the date of randomization until ANC recovers to> 500 and>1000/μL respectively.


Cantex Pharmaceuticals, Inc. Protocol No. CNTX-CX-01 2015 i\ML I Covance Study ID: 000000146201

Time to transfusion-independent platelet recovery (from date of randomization) is measured from the date of randomization until the first day that the platelet count recovers to> 20,000 and>100,000/ tL respectively (provided it is not as a consequence of platelet transfi.1sion and provided platelets are then maintained at> 20,000 and >100,000/μL respectively for the five subsequent clays without platelet transfusion).

### 3.3 Safety Endpoints

Key safety endpoints will be assessed by review of summaries of A Es which will include only treatmentemergent AEs (TEAEs), unless otherwise stated. Adverse events will be categorized by System Organ Class (SOC) and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA) dictionary (version 14.1), and will be graded according to NCI-CTCAE version 4.03.

### 4 PHARMACOKINETIC/PHARMACODYNAMIC VARIABLES

Details to be provided by Biocascade in a separate PK SAP.

### 5 ANALYSIS POPULATIONS

The analysis sets that will be used for statistical analyses are as follows:

<u>Intent-To-Treat (ITT)</u>: This includes all randomized patients. Patients will be analyzed according to the treatment to which they are randomized. The ITT Population will be the primary analysis set for the efficacy variables.

modified-Intent-To-Treat (m!TT): This includes all randomized patients who received at least one dosage of study drug. Patients will be analyzed according to the treatment to which they are randomized.

<u>Per Protocol (PP)</u>: Supporting analyses will be conducted on the PP Population, comprising all patients randomized and treated without major protocol deviations during the trial. This population will he documented before final database lock. PP Population will be analyzed according to the treatment lo which they received.

The following are considered protocol deviations for the purpose of identifying the per protocol set:

- 1. Patients who were subsequently found to be not complying with the inclusion and exclusion criteria
- 2. Patients who are not compliant with study restrictions (eg. use of prohibited medication (generic drug name) or prohibited treatment therapy)
- 3. Patients who continued in study but should have been withdrawn according to withdrawal criteria
- 4. Patients who are not compliant with study drug treatment dose modification or stoppage rules (either temporary or permanent).
- 5. Patients who took incorrect study drug (CX-01 or other) dose, frequency, timing or method of drug delivery (e.g. subject <u>overdosed with study drug, incomplete</u> study drug administered).

- 6. Patients who took different study drug than the study drug to which they were randomized.
- 7. Patients who do not have post baseline data anywhere in the system.

!terns I to 5 are routinely monitored in the study as part of the study monitoring plan.

<u>Safety</u>: All patients who received at least one dose of study treatment. Patients will be included in the analyses according to the treatment they received. The Safety Population will be used in the analyses of all safety endpoints.

### 6 DATA HANDLING

### 6.1 Time points and Visit Windows

Day I is defined as the day of randomization visit. Relative days after Day I are calculated as (assessment date... Day I date)+ I. Relative days prior to Day I are calculated as (assessment date Day I date). The day prior to Day I is Day -1.

All data will be analyzed using nominal study visits as defined in the Study Schedule and eCRF. No visit windows will he applied for summary and analysis.

In determining the baseline, if assessment on date of randomization is unavailable, then the last scheduled or unscheduled assessment before first study drug/randomization will be used instead.

### 6.2 Handling of Dropouts or Missing Data (where applicable)

For ITT analysis, patients with partial or missing data to determine morphologic complete remission on the eCRF form will be considered as not having met the criteria morphologic complete remission. For PP analysis and elsewhere, only the complete cases will be analyzed and no missing value imputation will be carried out.

Incomplete AE-related dates will be handled as follows:

- In cases where:
  - o the onset date is completely missing or
  - o the onset is in the same year (only the onset year is available) as the start of study treatment or
  - o the onset is in the same month and year (only the day is missing) as the start of study treatment or
  - o either the onset day or month is missing but the year is not before start of study treatment then the onset date will be replaced by the minimum of start of study treatment and AE resolution date.
- In all other cases the missing onset day or onset month will be replaced by first day or January.

- Incomplete stopping dates will be replaced by the last day of the month (if the day is missing only), unless this will result in a date after the date of death. If the imputed date will exceed the date of death, the date of death will be used as the stopping date. No imputation is needed if the event is ongoing.
- In all other cases the incomplete stopping date will not be imputed.

To impute missing day of follow-up dates (such as safety long term follow up) or Disease History, the missing day will be taken as the 15th of the month, as long as month and year is available. In all other cases missing or incomplete dates will not be imputed.

In patient listings, the documented date from cCRF will be reported (e.g. .May2016 in case where the day is missing, but month and year are available).

### 7 STATISTICAL METHODS

### 7.1 General Principles

All data processing, summarization and analyses will be performed using the Hosted SAS Environment Version 9.3 (or later) of the SAS' statistical software package.

Unless specified otherwise, data will be displayed using the following treatment group labels, in the order presented:

- Control,
  - o those who are on Idarubicin + Cytarabine therapy only
- Low CX-01,
  - o those who are on Idarubicin + Cytarabine + plus lower dose CX-01
- High CX-01,
  - o those who are on Idarubicin + Cytarabine + plus higher dose CX-01
- Overall

All data collected will be presented in listings by treatment group, site, subject and visit (where applicable), unless otherwise specified.

Data will be presented in snmmary tables by treatment group, and visit (where applicable). The category "Missing" will be presented if the number missing is greater than zero for at least one treatment group.

Descriptive summary statistics for continuous variables will include the number of subjects (N), mean, standard deviation (SD), median and range.

Descriptive summary statistics for categorical variables (such as gender, race) will include frequency counts and percentages [n (%)]. Unless stated otherwise in the table shells, the denominator for percentage calculations for a particular variable will be the number of subjects with non-missing data.

Dates will be displayed as DDMMMYYYY.

All significance tests will be two-sided and use a 5% significance level except for primary outcome, which is tested at I -sided at 15% level of significance.

### 7.2 Subject Disposition and Data Sets Analyzed

Subject disposition will be listed and summarized by treatment group and overall and will include the number and percentage of subjects:

- screened;
- randomized;
- randomized and not treated;
- treated;
- available at each study visit (treatment period, 30 day safety follow-up, long term follow-up at every 3 months until approximately 18 months or deaths of all patients, whichever is earlier);
- included in each study population (ITT, PP, Safety).

In addition, the number and percentage of subjects who complete the study and who discontinued early, including a breakdown of the primary reasons as reported in the eCRF for early termination, will be presented for all analysis populations (ITT, PP, Safety). Additional summaries frir safety follow up (reasons for not completing safety follow up) and long term follow up (status of long term follow up, cause of death recorded at long term follow up) will be provided for each treatment arm for the JTT, PP and safety population.

A summary of patient enrollment by site will also be provided by treatment group and overall for the ITT population.

A summary of the reasons for screen failure as well as the number of subjects screened but not randomized will be produced. No other informati, In for screen failures will be presented.

### 7.3 Protocol Deviations

All protocol deviations will be listed and summarized by treatment group for the ITT population.

All important protocol deviations leading to exclusion from the PP population (see Section 5) will be listed and summarized by treatment group for the ITT population.

### 7.4 Demographics and Other Baseline Characteristics

Demographic and baseline characteristics will be listed and summarized by treatment group and overall for all analysis populations (ITT, PP, Safety). Standard descriptive statistics will be presented for the continuous variables of:

- Age at screening (years) [calculated as (informed consent date date of birth)/365.25 and reported as whole years;
- weight (kg);
- height (cm);
- BMI
- Time since diagnosis
- Baseline blasts in bone marrow(%)
- Baseline LDH

The total counts and percentages of subjects will be presented for the categorical variables of:

- age group (years) (grouped as <70 and 2: 70);
- sex;
- race;
- ethnicity;
- AML type (de novo or secondary);
- Baseline peripheral blasts (Yes/No)
- ECOG performance status
- Time since diagnosis(<= 30 days,> 30 days)

No formal tests of statistical significance will be performed on the demographic and baseline data.

Other baseline measurements, such as bone marrow aspirate/biopsy, pregnancy test result, lab parameters, vital signs, ECG and ECOG, will be summarized by treatment group with the post-baseline measurements.

### 7.4.1 Medical History

Medical history will be coded using the latest available Medical Dictionary for Regulatory Activities (MedDRA). All medical history will be listed, and the number and percentage of subjects with any medical history will be summarized for some analysis populations (ITT, Safety) by system organ class (SOC) and preferred term (PT) for each treatment group and overall.

Cantex Pharmaceuticals, Inc. Protocol No. CNTX-CX-0 I 20 I 5 \ML I Covance Study ID: 00000014620 I

### 7.4.2 Prior, Post treatment (anti AML) and Concomitant Medications

Medications received prior to or concomitantly with treatment will be coded using the WHO Drug Dictionary [March 2016 132 version] Anatomical Therapeutic Chemical (ATC) Classification codes.

Prior, post treatment medications and concomitant medications are defined as follows:

- Concomitant medications are those with a start date on or after the first dose date of study treatment,, or those with a start date before the first dose date of study treatment and a stop date on or after the first dose date of study treatment.
- Prior medications will be defined as non-study medication with a stop date prior to the first dose of study treatment.
- Post treatment medications are those with start date after the last dose of study drug.

Concomitant medications will be further divided according to whether they were started before (both prior and concomitant) or after (concomitant-only) the first dose of treatment.

If a medication cannot be classified as "prior" or "concomitant" after applying imputation rules for missing/incomplete dates, it will be classified as concomitant.

Prior anti-AML treatment medications and concomitant medications will be listed and summarized separately for ITT analysis population. Post treatment medications will be listed only.

The number and percentage of subjects using each medication will be displayed together with the number and percentage of subjects using al least one medication within each therapeutic class (ATC-Level 2), chemical subgroup (ATC-Level 4), and generic term.

### 7.5 Measurements of Treatment Exposure and Study Drug Usage Rate

Extent of study treatment exposure will be summarized for the entire study treatment period and by cycle. Exposure variables will include duration of study treatment, number of dose reductions, number of treatment delays (interruptions), number of treatment cycles, and dose intensity relative lo dose levels specified in the protocol.

There are three types of treatment cycles: induction cycle, re-induction and consolidation cycles. For each cycle, the exposure for each drug (Jdarubicin, Cytarabine, CX-01) is taken as the sum of duration of drugs for drug taken within that cycle. For drugs that started and ended on the same day, it will be regarded as I day, for drugs that started and ended on different days, the duration will be calculated as date of last dose minus date of first dose + 1 day for the period which the drug was administered. Proportion of patients who are exposed to the full expected duration for each component of the study drug will be presented for each cycle.

The study drug usage rate calculation for the induction cycle is as follows, where the expected number of days is the number of days the <u>patients were expected to take</u> the drug, up to the point of study


Cantex Pharmaceuticals, Inc. Protocol No. CNTX-CX-01 2015 AML I Covance Study ID: 000000146201

discontinuation. If a patient was scheduled to lake 7 days of drug but only took the drug for 5 days because of early withdrawal, then the expected number of days would be 5.

The calculation of BSA will be based on the best possible results for study drug usage (closest to 100% and below) from Mostellar, Dubois and Gehm, formulae as outlined below.

### DuBois[ I]

BSA (11f) = 0.007184 x Height(cm)  $^{0.725}$  x Weight(kg)  $^{04.25}$ 

Gehan/2]:

BSA  $(111^2)$  =, 0.0235 x lle ight(cm)  $^{042246}$  x Weight(kg)  $^{0.51456}$ 

Mostellar/3]:

BSA  $_{(111)}^{2} = ([\text{Heigh!(cm)} \times \text{Weight(kg)}] / 3600)^{0.5}$ 

### **Group |: Idarubicin + Cytarabine**

Idarubicin: Actual total dosage per 1112/(12 mg/1112 x expected number of days) [Maximum expected number of

days=3

Cytarabine: Actual total dosage per 1112/( I 00 mg/1112 x expected number of days) [Maximum expected number of

days=7]

### Group 2: Idarubicin + Cytarabinc + plus lower dose CX-01

Initial CX-01 4 mg/kg, (0 or 100%)

CX-01: Actual total dosage per kg/(3 mg/kg/dayx expected number of days) [Maximum expected number of

days=7]

ldarnbicin: Actual total dosage per 1112/(12 mg/1112 x expected number of days) [Maximum expected number of days,-

31

Cytarabine: Actual total dosage per 1112/( I 00 mg/1112 x expected number of days) [Maximum expected number of

days=7]

### Group 3: Idarubicin + Cytarabinc + pins higher dose CX-01

Initial CX-01 4 mg/kg, (0 or 100%)

CXOI: Actual total dosage per kg/(6 mg/kg/dayx expected number of days) [Maximum expected number of

days=7]


Page 20 of 34 ST-\D-008 version 02

Version: Final Dale of Issue: 20 March 2018

Canlex Pharmaceuticals, Inc, Protocol No, CNTX-,(:X-01 2015 AML I Covance Study ID: 000000146201

Idarubicin: Actual total dosage per 1112/(12 mg/1112 x expected number of days) [Maximum expected number of

days=3]

Cytarabine: Actual total dosage per 1112/(100 mg/1112 x expected number of days) [Maximum expected number of

days=7]

The study drug usage rate calculation for the re-induction cycle under 5+2 regimen is as follows:

### **Group 1: Idarubicin + Cytarabinc**

Idarubicin: Actual total dosage per 1112/(12 mg/1112 x expected number of days) [Maximum expected number of

days 002]

Cytarabine: i\ctual total dosage per 1112/(100 mg/1112 x expected number of days) [Maximum expected number of

days=5]

### Group 2: Idarubicin + Cytarabinc + plus lower dose CX-01

Initial CX-01 4 mg/kg, (0 or 100%)

CXO1: Actual total dosage per kg/(3 mg/kg/day x expected number of days) [Maximum expected

number of days=S]

Jdarubicin: Actual total dosage per 1112/ (12 mg/1112 x expected number of days) [Maximum expected

number of days=2]

Cytarabine: Actual total dosage per 1112/ (100 mg/m2 x expected number of days) [Maximum expected

number of days=5]

### Group 3: Idarubicin + Cytarabinc + plus higher dose CX-01

Initial CX-01 **4** mg/kg, (0 or 100%)

CXOJ: Actual total dosage per kg/ (6 mg/kg/dayx expected number of days) [Maximum expected

number of days=5]

ldarubicin: Actual total dosage per 11121 (12 mg/1112 x expected number of days) [Maximum expected

number of days=2]

Cytarabine: Actual total dosage per 1112/ (100 mg/m2 x expected number of days) [Maximum expected

number of days=5]

The study drug usage rate calculation for the consolidation cycle is as follows:


Cantex Pharmaceuticals, Inc. Protocol No. CNTX-CX-01 2015 AML I Covance Study ID:000000146201

### **Group 1: Cytarabinc**

Cytarabine: Actual total dosage per m2/ (2 g/ m2x expected number of days) [Maximum expected number of days=3]

### Group 2: Cytarabine + plus lower dose CX-01

Initial CX-01 4 mg/kg, (0 or 100%)

CXOJ: Actual total dosage per kg/(3 mg/kgx expected number of days) [Maximum expected

number of days=5]

Cytarabine: Actual total dosage per 1112/(2 g/ rn2x expected number of days) [Maximum expected

number of days=3]

### Group 3: Cytarabinc + plus higher dose CX-01

Initial CX-01 4 mg/kg, (0 or 100%)

CXOI: Actual total dosage per kg/(6 mg/kgx expected number of days) [Maximum expected

number of days-,5]

Cytarabine: Actual total dosage per 11<sup>2</sup>/(2 g/ nix expected number of days) [Maximum expected number

of days=3]

### 7.6 Efficacy

### 7.6.1 Primary Efficacy Analysis

Fisher exact test will be used to compare the proportion of CRs between each dose and control for the ITT population using one sided test at 15% level of significance along with a 70% CI. These tests will be conducted in a fixed sequence: higher dose versus control first and lower dose versus control second, with the second test considered exploratory (failed) if the first test fails.

### 7.6.2 Secondary Efficacy Analysis

The primary efficacy analysis will be repeated using the PP Population as a supportive analysis along with CRi and composite CR for ITT and PP. Complete response rates and composite complete response rates and confidence intervals will also be reported for key subgroups (De-novo *vs* secondary AML at diagnosis, Age< 70 vs Age 2 70, ECOG performance status:::: 1 vs ECOG performance status =2). The following secondary analyses will be performed on the ITT population. Analyses of EFS, LFS, time to neutrophil and platelet recovery, and OS will be descriptive. Kaplan-Meier (KM) estimates will be used to estimate the survival distribution for each arm and KM plots will be produced to accompany these analyses. 95% Confidence Intervals will be reported for medians and KM estimates. Duration of response will be analyzed using a similar approach; the survival distributions will be estimated as cumulative incidence functions.

M01iality rate at Day 30, Day 60, and Day 90 will be reported using descriptive statistics in a manner similar lo the reporting of the morphologic CR rate. The time to neutrophil and platelet recoveries will be reported using the following descriptive statistics: N, mean, SD, median, minimum, maximum, and the 1st and 3<sup>rd</sup> quartiles.

### 7.6.3 Sensitivity Analysis

None.

### 7.6.4 Subgroup Analysis

Descriptive statistics for the primary efficacy variable (CR) and composite CR and 95% confidence intervals will be provided of the following subgroups for ITT population provided there is sufficient number of patients in total within the subgroup across the treatment arms:

- Age groups (<70 and 2: 70)
- AML at diagnosis (de novo, secondary)
- ECOG performance status (:S 1 Vs ECOG=2)

### 7.6.5 Exploratory Analysis

Additional efficacy analyses will be performed as exploratory analysis for the following variables, summarized by treatment groups and analyzed in the same way as secondary analyses above.

- Duration of composite CR (if present)
- Days until neutrophil recovery to 2: 500/ LL (from date of randomization and from date of first study drug)
- Days until platelet recovery to 2: 20,000/ LL (from date of randomization and from date of first study drug)

### 7.7 Safety

### 7.7.1 Adverse Events

All adverse events (AEs) recorded on the eCRF will he coded using the MedDRA dictionary [Version 14. 1] and classified as either pre-treatment AEs or treatment - emergent AEs (TEA Es) as follows:

- Pre-treatment AEs are events that stail prior to the date of first dose of study treatment.
- Treatment-emergent AEs (TEAEs) arc events with start date and time on or after the date and time of first dose of study treatment (and up to 30 days after date of last dose of treatment) with

start dale prior to the dale of first dose of study treatment whose severity worsens on or after the dale and time of first dose of study treatment.

Assessment of AE severity will be based on the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE, version 4.0.3).

All AF data will be listed by treatment group including Pre-treatment AEs and TEAEs. The number and percentage of subjects reporting each treatment AE and TEAEs will be summarized for each treatment group and overall, by System Organ Class (SOC) (sorted alphabetically) and Preferred Term (PT) (sorted by descending overall total) for Safety populations.

In addition, corresponding listings of serious AEs (SAEs), AEs leading to discontinuation of treatment, AEs causing interruptions from study treatment, AEs causing dose reduction from study treatment and study treatment-related AEs causing dose reductions are provided.

An overview table will summarize the number and percentage of subjects with at least one of the following AEs/TEAEs, where subjects with more than one AEs/TEAE in a particular category are counted only once in that category:

- any AE;
- any TEAEs;
- treatment-related TEAE;
- any AE by maximum NCI-CTCAE grade; treatment-related TEAE by maximum NCJ-CTCAE grade;
- AE leading to treatment interruption;
- treatment- emergent AEs leading lo treatment interruption;
- AF leading to treatment reduction;
- treatment- emergent AEs leading to treatment reduction;
- AE leading lo treatment discontinuation; treatment-emergent AEs leading to discontinuation from the study;
- SAE;
- treatment-emergent SAE;
- SAE leading to death;
- treatment-emergent SAE leading to death;
- SAE leading to treatment discontinuation;

The number and percentage of subjects reporting each TEAE will be summarized by System Organ Class (SOC) and Preferred Term (PT) for the Safety population. Tables will be sorted alphabetically by SOC. !'Ts will be sorted by descending overall total; if the number and percentage are the same for different PTs, the PTs will be listed in alphabetical order (within the SOC). The following summaries will be produced:


Cantex Pharmaceuticals, Inc. Protocol No. CNTX-CX-01 2015 AML I Covance Study ID: 000000146201

- TEAEs by SOC and PT;
- TEAEs by PT;NCI-CTCAE Grade 3 or higher TEAEs by SOC and PT;
- NCI-CTCAE Grade 2 or lower TEAEs by SOC and PT;
- TEAEs related to treatment, by SOC and PT;
- TEAEs by maximum NCl-CTCAE grade, by SOC and PT;
- Treatment--related TEAEs by maximum NCI-CTCAE grade, by SOC and PT;
- TEAEs causing discontinuation from treatment, by CTCAE and worst CTCAE grade;
- TEAEs related lo treatment causing discontinuation from treatment, by CTCAE and worst CTCAE grade;
- Serious TEAEs, by SOC and PT;
- NCI-CTCAE Grade 3 or higher Serious TEAEs, by SOC and PT;
- NCI-CTCAE Grade 2 or lower Serious TEAEs, by SOC and PT;
- Serious TEAEs related lo treatment by CTCAE and worst CTCAE grade;
- TEAEs leading to death, by SOC and PT

In the above summaries, subjects with more than one AE/TEAE within a particular SOC are counted only once for that SOC. Similarly, subjects with more than one AE/TEAE within a particular PT are counted only once for that PT. For summary by maximum severity, subjects with multiple AE/TEAEs within a particular SOC or PT will be counted under the category of their most severe AE/TEAE within that SOC and PT.

### 7.7.2 Laboratory Evaluations

Clinical laboratory assessments will be summarized using frequency tables, shift tables, and descriptive statistics. Frequency tables and shill tables will be presented by NCI-CTCAE grade. Laboratory variables with no NCI-CTCAE group will be presented in shift tables with respect to normal range. All laboratory variables will be presented in tables of descriptive statistics (mean, SD, etc.) and graphs will be presented for PT/INR, aPTT, anti-factor Xa, fibrinogen, D-dimer, and platelet count.

### 7.7.3 Vital Signs and ECOG performance status

Vital signs variables and ECOG performance status will be summarized using descriptive statistics at screening visit and start of consolidation cycle (vital signs only).

### 7.7.4 Electrocardiograms

Counts and proportion of patients with clinically significant abnormal results at screening and Day 7 will be reported.

Cantex Pharmaceuticals, Inc. Protocol No. CNTX-CX-0 I 20 I 5 AML I Covance Study ID: 000000 I 4620 I

### 7.8 Interim Analysis

A Data Safety Monitoring Committee (DSMC) will be instituted for this study according to a separate DSMC Charter in order to ensure ongoing safety of study subjects.

No other interim analysis is planned.

### 8 CHANGES FROM PLANNED ANALYSES IN PROTOCOL

A new analysis population m!TT is added as per client request aner the first DSMB meeting.

For primary objective, the time component required (on or after 21 days from date of randomization) for the recognition of morphologic CR is added in the definition.

For secondary objective, the time component required (on or after 21 days from date of randomization) for the recognition of CRi and CRp is added in the definition.

For secondary and exploratory objectives, the following variables are additional to the protocol:

- Duration of composite CR, with the definition of composite CR being clarified as CR or CRi or CRp.
- Days until neutrophil recovery to 2: 500/ ,tL
- Days until platelet recovery to 2: 20,000/ ,tL

For Leukemia-Free State (LFS), the definition is now changed to from date ofleukemia free state, because the protocol definition from date of randomization is not correct.

Repeat of CRi and composite CR in the same fashion as primary efficacy analysis and addition of composite CR for subgroup analysis.

Compliance is termed as study drug usage rate in the SAP.

Competing risk of death analyses will not be performed.

Post treatment medications will only be listed and not summarized as per client request.

### 9 DATA ISSUES

Not applicable.

### 10 REFERENCES

[I] DuBois D, DuBois DF. A formula to estimate the approximate surface area if height and weight be known. Arch Int Med 1916;17:863-71.


Cantex Pharmaceuticals, Inc. Protocol No. CNTX-CX-0 I 20 I 5 AML I Covance Study ID: 000000 I 4620 I

12] Gchan EA, George SL. Estimation of human body surface area from height and weight. Cancer Chemother Rep 1970;54:225-35.

[3] Mosteller RD. Simplified calculation of body-surface area. N Engl. I Med 1987;3 17: I 098.

Covance Study ID: 000000 J 4620 J

Date 9 f\_lssue: 20 March 201Jl

### 11 APPENDICES

# **Appendix I- Schedule of Events**

Table 11-1 Induction/Re-induction Cycle Schedule of Study Procedures

| Examination | Scree<br>n<br>Visit<br>D<br>-28- | DI | D2 | D3 | D4 | DS | D6 | D7 | D<br>8-13 | D<br>14-21 | At count recovery & Weekly from D21 | Early<br>Term Visit | Safety FU visit<br>(30 days after<br>last dose of<br>treatment) | Long Term FU contact (every 3 month |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | until<br>count<br>recovery<br>or D60 <sup>15</sup> | | | sup to<br>death, or<br>EoS) <sup>16</sup> |
| Informed consent <sup>1</sup> | X | | | | | | | | | | | | | |
| Demographic and medical history | X | | | | | | | | | | | | | |
| Eligibility criteria | X | X | | | | | | | | | | | | |
| Randomization | | X | | | | | | | | | | | | |
| Idarubicin <sup>2</sup> | | X | X | X | | | | | | | | | | |
| Cytarabine <sup>3</sup> | | X | X | X | X | X | X | X | | | | | | |
| CX-01 Bolus <sup>4</sup> | | X | | | | | | | | | | | | |
| CX-01 <sup>5</sup> | | | | | | | | | | | | | | |
| continuous infusion | | X | X | X | X | X | X | X | | | | | | |
| ECOG status | X | | | | | | | | | | | | | |
| Vital signs (BP, | X | | | | · | | · | | | | | | | |


Covance Study ID: 00000014620 I

Date of Issue: 2J) March 201 !1

Table 11 1 Induction/Re-induction Cycle Schedule of Study Procedures

| Examination | Scree<br>n<br>Visit<br>D<br>-28-<br>1 | DI | D2 | D3 | D4 | D5 | D6 | D7 | D<br>8-13 | D<br>14-21 | At count recovery & Weekly from D21 until count recovery or D60 <sup>15</sup> | Early<br>Term Visit | Safety FU visit<br>(30 days after<br>last dose of<br>treatment) | Long Term FU contact (every 3 month sup to death, or EoS) 16 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| heart rate, height and weight) <sup>6</sup> | | | | | | | | | | | | | | |
| Physical exam | X | | | | | | | | | | | | | |
| 12-lead ECG | X | | | | | | | X | | | | | | |
| Echocardiography orMUGAscan | X | | | | | | | | | | | | | |
| Hematology <sup>7</sup> | Х | X | X | X | X | X | X | X | X | Х | Х | X | Х | |
| Anti-factor Xa, 89 | Χ | Χ | Χ | X | X | X | X | X | x9 | | | X | | |
| PT/INR, aPTT <sup>8</sup> 10 | X | X | Х | Χ | X | X | X | Χ | xio | X | X | X | X | |
| Chemistry <sup>11</sup> | X | X | X | X | X | X | X | X | X | Х | X | X | X | |
| PK sampling <sup>12</sup> | | | | X | | X | | | | | | | | |
| AE Assessment | | | | | | | | | ( | Continuo | usly | | <del>, i</del> | |
| Previous medications | X | ! | | | | | | | | | | | | |
| Concomitant medications | | | | | | | | | ( | continuo | usly | | ,' | |

Covance Study ID: 000000146201

Date of 1\$!Oe: 20 Marrl! 2018

Table 11-1 Induction/Re-induction Cycle Schedule of Study Procedures

| Examination | Scree<br>n<br>Visit<br>D<br>-28-<br>1 | DI | D2 | D3 | D4 | D5 | D6 | D7 | D<br>8-13 | D<br>14-21 | At count recovery & Weekly from D21 until count recovecy or D60 <sup>15</sup> | Early<br>Term Visit | Safety FU visit<br>(30 days after<br>last dose of<br>treatment) | Long Term FU contact (every 3 month sup to death,or EoS) 16 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Fibrinogen,<br>D-dimer | X | | | | | | | | | | X | X | X | |
| Serum or urine pregnancy test <sup>13</sup> | X | | | | | | | | | | | | X | |
| Bone marrow<br>aspirate/<br>Biopsy <sup>14</sup> | x14 | | | | | | | | | xi4 | x14 | | | |
| Relapse and survival data | | | | | | | | | | | | | | X |

**Abbreviations:** AE=adverse event, ALT=alanine aminotransferase, ANC=absolute neutrophil count, anti-Xa=anti-factor !0a, aPTT=activated partial thromboplastin time, AST=aspartate aminotransferase, BP=blood pressure, BUN=blood urea nitrogen, CBC=complete blood count\_ CX-01=2-O, 3-0 desulfated heparin, D=day, ECG=electrocardiogram, ECOG=Eastern Cooperative Oncology Group. EoS=end of study, FU=follow-up, INR=international normalized ratio, IV=intravenous, LDH=lactate dehydrogenase, MUGA=multi gated acquisition. OS=overall survival, PK=pharmacokinetics, PT=prothrombin time, Term=termination.

| l. | Informed | l consent | t must t | oe obtained | befo | re any | stud | ly-rel | ated | proced | lures | are | cond | ucte | d |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

Version: Final
Cantex Pharmaceuticals, Inc. Protocol No. CNTX-CX-0 I 2015 AML I

Covance Study ID: 00000014620 I

Date Offssue: 2JLMarch 201

- 2. Idarubicin administered at a dose of 12 mg/m²/day by slow (10 to 30 minutes) IV injection/infusion daily on Days 1, 2, and 3.
- 3. Cytarabine administered at a dose of 100 mg/m²/day as a continuous 24-hour IV infusion on Days 1-7. Patients who do not achieve leukemia-free state (<5% bone marrow blasts) on bone marrow aspirate performed between Days 14-21 may receive a reinduction cycle with the same regimen ("7 + 3" ± CX-01). Ifin the Investigator's opinion, the patient is not fit to receive full reinduction cycle of "7 + 3" ± CX-01, at the Investigator's discretion the patient may receive "5 + 2" ± CX-01 which is 5 days of cy1arabine (Days 1-5) and 2 days of idarubicin (Days 1 and 2).
- 4. CX-01 administered at a dose of 4 *mg/kg* as an initial bolus on Day 1 only, 30 minutes after completion of administration of the first dose of idarubicin.
- 5. CX-01 administered at a dose of 0.125 or 0.25 mg/kg/hour as a continuous 24-hour IV infusion on Days 1-7.
- 6. Height obtained at Screening only. Actual body weight will be measured at the beginning of each cycle to calculate treatment doses.
- 7. Hematology **must** include the following: hemoglobin, ANC, and platelets. All other hematology assessments should be performed only if standard of care and/or clinically indicated. Hematology samples will be collected daily until discharge and weekly thereafter until recovery.
- Note: blood samples for PT/INR, aPTT and anti-Xa levels will be collected 12 hours after the bolus dose of CX-01.
- 9. Anti-Xa samples ,vill be collected only on Days 1-8.
- Io. PT/aPTT will be collected daily on Days 1-8, and on Day 9, Day 1 L and Day 13.
- 11. Chemistry (and comprehensive metabolic panel) includes BUN, serum creatinine, total bilirubin, ALT, AST, and alkaline phosphatase. Samples will be collected daily until discharge.
- 12. At selected sites, blood samples for steady-state PK analysis will be collected during the induction cycle from the first six randomized patients assigned to CX-01 on Days 3 and 5 at a single time point.
- 13. For females of childbearing potential only. All female patients will have a urine pregnancy test at Screening; positive urine tests must be confirmed by a serum pregnancy test.
- 14. Bone marrow aspirates and/or biopsies are not performed weekly. If the patient's peripheral blood is negative for persistent AML: a bone marrow aspirate and/or biopsy will be performed (once) between Days 14-21 to determine the need for re-induction. Bone marrow biopsy may be necessary if sufficient spicules are not available on aspirate. Bone marrow aspirate at baseline and follow-up should include analysis by flow cylometry and cytogenetic analysis. Bone marrow (or peripheral blood if bone marrow is unavailable) should be sent to the institution's local cylogenetic laboratory for analysis. For patients with documented CR, confirmatory bone marrow aspirate slides will be submitted to the Sponsor or designee. If count recovery has not occurred by Day 42, a bone marrow aspirate/biopsy will be performed to evaluate disease status, unless presence of persistent AML in peripheral blood.


Version: FinalDa Jeof Issue: 21:1 iVlarch 201 1!Cantex Pharmaceuticals, Inc. Protocol No. CNTX-CX-01 2015 AML 1Covance Study JD: 000000146201

- 15. Count recovery is defined as ANC of>  $1000/\mu$ L and a platelet count> $100,000/\mu$ L.
- 16. During long term follovi-up, relapse and survival data will be collected every 3 months until death or until the end of study. The end of study will occur approximately 18 months after the last patient is randomized.


Cantex Pharmaceuticals, Inc. Protocol No. CNTX-CX-0 I 2015 AML I

Covance Study ID: 00000014620 I

Table 11-2 Consolidation Cycle Schedule of Study Procedures

| <u>Table 11-2 Consolidation Cycle Schedule of Stud</u> | ту г | 1000 | uur | JS , | | |
|---|---|---|---|---|---|---|
| Examination | l) | I) | I) | I) | l) | Weekly |
| | 1 | 2 | 3 | 4 | 5 | from D6 |
| | | | | | | until |
| | | | | | | count |
| | | | | | | recover |
| | | | | | | у8 |
| Hematology <sup>1</sup> | X | X | X | X | X | X |
| PT/INR, aPTT, and anti-X a <sup>2</sup> | X | X | X | X | X | |
| Chemistry <sup>3</sup> | X | X | X | X | X | X |
| Vital signs (BP, heart rate, height and weight) <sup>4</sup> | X | | | | | |
| Cytarabine <sup>5</sup> | X | | X | | X | |
| c·X-01 Bolus <sup>6</sup> | X | | | | | |
| CX-01 <sup>7</sup> continuous infusion | X | X | X | X | X | |
| Concomitant medications | continuously | | | | | |
| | | | | | | <del>,</del> |
| Adverse events | continuously | | | | | |
| | | | | | | • |
| Bone marrow aspirate/ | | | | | | x9 |
| Biopsy | | | | | | 22.7 |

**Abbreviations:** aPTr-"activated partial thromboplastin time, anti-Xa=anti-factor IOa, BP<sup>®</sup> blood pressure; CBC=complete blood count, D=day, INR=international normalized ratio, PT=prothrombin time.

- 1. Hematology **must** include the following: hemoglobin, ANC, and platelets. All other hematology assessments should be performed only if standard of care and/or clinically indicated. Hematology samples will be collected daily until discharge and weekly thereafter until recovery.
- 2. PT/aPTT and anti-Xa blood samples will be collected 12 hours alter the bolus dose of CX-01.
- 3. Chemistry (and comprehensive metabolic panel) will be collected daily until discharge.
- 4. Actual body weight will be measured at the beginning of each cycle to calculate treatment doses.
- 5. Cytarabine administered at a dose of 1.0 g/m<sup>2</sup> over 3 hours, every 12 hours on Days 1, 3, and 5.
- 6. CX-01 administered at a dose of 4 mg/kg as an initial bolus on Day 1, 30 minutes after completion of the first 3-hour infusion of cytarabinc, followed immediately by a continuous CX-01 24-hour IV infusion.
- 7. CX-01 administered at a dose of 0.125 or 0.25 mg/kg/hour as a continuous 24-hour IV infusion on Days 1-5 for a total of 120 hours of continuous CX-01 infusion.
- 8. Count recovery is defined as ANC of> 1000/μL and a platelet count>100,000/ tL.
- 9. Bone marrow aspirate/biopsy is not done weekly. If the patient's peripheral blood is negative for persistent AML and count recovery has not occurred by Day 42 (of Consolidation cycle), a bone marrow aspirate/biopsy will be done to evaluate disease status.

|---|
| Cantex Pharmaceuticals, Inc. Protocol No. CNTX-CX-01 2015 AMI, I |

Cantex Pharmaceuticals, Inc. Protocol No. CNTX-CX-01 2015 AML I Covance Study ID: 00000014620 I

# **Appendix 11 - Table, Figure and Listing Shells**

The tabk, figure and listing shells and corresponding Table of Contents. are available as a separate file.
## TABLES, FIGURES, AND LISTINGS SHELLS

## A Randomized, Phase II Study of CX-01 Combined With Standard Induction Therapy for Newly Diagnosed Acute Myeloid Leukemia

TFL Status: Final TFL Date: 20 I 8-03-08T07:32:05

Study Drug: CX-0 I

Sponsor Reference: Covance Study No: 00000014620 I

#### I. INTRODUCTION

The table, figure, and listing (TFL) shells presented in this document arc mock-ups and may be subject to minor format modifications once the actual data are used. The data represented in this document arc used for example purposes only and do not reflect the actual study data captured. The overall contents in any individual TFL shell will not change, although additional tables may be added if necessary, thus changing the table number scheme. Significant changes will be approved by the responsible Covance Clinical Pharmacology project team member and communicated to the Sponsor.

## 1.1 General Programming Specifications

All TFLs will follow the following rules:

Papersize will be A4, with the following margins in Inches:

Every TFL will have a footnote containing program location, name, run date and run time (optional), listing source, the name of the last person who ran the program, and the status of the output: Dry run - Draft-- Final Draft- Final (others as needed)

Dates will be presented in the format yyyy-mm-dd

The presentation order of the statistics will be:

Mean, SD, median, minimum, maximum, N. The abbreviations Med, Min, Max may be used, if necessary.

Rules for significant digits in safoty data tables are as follows: if the raw value has x decimal places, then the mean and the median will have x decimal places, the standard deviation will have x+I decimal places.

N will be presented as whole numbers.

#### 1.2 Derived Parameters

Individual derived parameters (e.g. pharmacokinetic parameters) and appropriate summary statistics will be reported to three significant figures.

## 1.3 Tables Summarizing Categorical Data

Tables that summarize categorical data will be created per these specifications:

- I. If the number of events is zero, data will be presented as "0".
- 2. If the categories of a parameter are ordered, all categories between the maximum possible category and the minimum category will be included, even if tF0 for a given category.
- 3. If the categories arc not ordered, only those categories for which there is at least one subject represented will be included.
- 4. A "missing" category will be included for any parameter for which information is missing. This will ensure that the population size totals are consistent across different parameters.

## 2. TJ:.BLE Cf CC?<)'?SN'IS

| 10.000 |
|---|
| IC |
| 12 |
| 13 |
| 14 |
| 14 |
| 14 |
| 14 |
| on in |
| ¥7 |
| 22 |
| 22 |
| 23 |
| 74 |
| 1984 - De 1984 - All General II. (1984 - All 1984 - All 1984 - All 1984 - All 1984 - All 1984 - All 1984 - All |
| 1988 - |
| 90 |
| 23 |

| Table 14.1.26 | Summary of Study Drug Usage Rate Induction Cycle Safety Population | 30 |
|---|---|---|
| Table 14.!.27 | Summary of Study Drug Usage Rate Re-induction (7+3) Cycle Safety Population | 31 |
| Table 14.1.28 | Summary of Study Drug Usage Rate Re-induction (5+2) Cycle Safety Population. | 31 |
| Table 14.1.29 | Summary of Study Drug Usage Rate Consolidation Cycle I Cycle Safety Population | |
| Table 14.1.30 | Summary of Study Drug Usage Rate Consolidation Cycle 2 Cycle Safety Population | |
| Table 14.1.31 | Summary of Treatment E::posure by Cycle Safety Population | 32 |
| Figure 14.2.1 | Overall Sun iYal plot ITT Population | 37 |
| Figure 14.2.2 | O\earli Su01\all plot \\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ | 37 |
| Figure 14.2.3 | O\crall Sur\ 1\al plot PP Populatmn | 37 |
| Figure 14.2.4 | ( [F plot for e\enl tree sutvl\al (from date of random 2.atlon) IIISpf: !flation | 38 |
| Figure 14.2.5 | CIP 1 · C · C · TV 1 (C · 1 · C · 1 · C · VEED D · 1 · C | 39 |
| Figure 14.2.6 | | 39 |
| Figure 14.2.7 | | 39 |
| Figure 14.2.8 | | 39 |
| Figure 14.2 9 | CIE plot for platelet (>20000) recovery (from date of randomization) ITT Population | 3.6 |
| Figure 14.2 JO | CIF plot for neunophil (>1 000) recovery (from date of randomization) ITT Population | 39 |
| Figure 14.2.11 | CJF plot for platelet(>100000) recovery (from dai,:;. of randomization) ITT Population | 39 |
| Figure 14.2.12 | OIE 1 ( | |
| Figure 14.2.13 | CIF plot for relapse (composite CR) ITT Population | 30 |
| Figure !4.2.14 | CIF plot for relap:>e (composite CR) MITT Popular ion | 39 |
| Table 14.2.1 | Primary Outcome-CR ITT Population | 40 |
| Table 14.2.2 | Primary Outcome-CR M!TT Population | 40 |
| Table 14.2.3 | Primary Outcome-CR PP Population | 40 |
| Table 14.2.4 | Secondary Outcome-CRi [TT Population | 40 |
| Table 14 2.5 | Secondar: Outcome-CRi MJTT Population <sub>B</sub> | 40 |
| Table 14.2.6 | Secondary Outcome-CRi PP Population | 41 |
| Table 14.2.7 | Secondary Outcome-Composite CR ITT Papplatation | 41 |
| Tabie 14.2.8 | Secondary Outcome-Composite CR MJTTIPppplatition | 41 |
| Table 14.2.9 | Secondary Outcome-Composite CR PP Popplishion | 41 |
| Table 14.2.10 | Mortality Day-30 iTT Population | 42 |
| Table 142.11 | Mortality Day-60 ITT Population | 42 |
| Table 14.2.12 | Mortality Day-90 !TT Population | 42 |
| Table 11-2.13 | Nortality Day-30 M11 1 Population | 42 |
| Table 14.2.14 | !\fortality Day-60 MITT Population: | 42 |
| Table 14.2.15 | \fortality Da;,'-90 t\ffIT Population | 42 |
| Table 14.2.16 | l\fortality Da:,-30 PP Population | 42 |
| Table 14.2.17 | Morality Day-60 PP Population | 42 |
| Tab!c 14.2.18 | Mortality Day-90 PP Population | 42 |
| Table 14.2.19 | Summary of Overall Survival ITT Population | |

| Table 14.2.20 | Summary of O\-eral! Survival MITT Population | 4 |
|---|---|---|
| Table 14.2.21 | Summary of Overall Survival PP Population | |
| Table 14.2.22 | Summary of OYerall Survival KM Estimate !TT Population | |
| Table 14.2.23 | Summary of Overall Survival KM Estimate MITT Population | |
| Table 14.2.24 | Summary of O'"erall Sun:i\al KM Estimate PP Population | |
| Table 14.2.25 | Time to EYent Free Survival - Days ITT Population | |
| Table 14.226 | Time to faent Free Survival - Days IVHTT Population | 1 |
| Table i4 2.27 | Time to Leukemia Free Survival - Days (from randomization) ITT Population | 4 |
| Table 14.2.28 | fime to Leukemia Free Survival - Days (from randomization) MITT Population | 4 |
| Table 14.2.29 | Time to "Keutrophil Recovery (>500) - Days (from randomization) ITT Porulation | 4 |
| Table 14.2.30 | Time to platelet Recovery (>20000) - Days (from randomization) !TT Population | 4 |
| Table 1-U.31 | Time to Neutrophil ReCO\"ery (> 1000) - Days (from randomization) ITT Population | 4 |
| Table t-+.2.32 | Time to plateiet Reco\ery (>100000) - Days (from randomiz.ation) ITT Population | 4 |
| Table 14.2.33 | Time to reiapse (duration of morphologic CR)- Days ITT Population | |
| Table 14.2.34 | Time to relapse {duration of composite CR) - Days fTT Population | |
| Table 14.2.35 | Time to E\enl Free Survival - Days (from randomization) PP Population | |
| Table 14.2.36 | Time to Leukemia Free Sun; ival - Days PP Population | to the state of th |
| Table 14.2.37 | Time to::eutrophii Recovery (>500)- Days (from randomization) PP Population | 14 |
| Table 14.2.38 | Time to diatelet K. covery (>20000)- Days (from randomization) PP Population. | 1 |
| Table 14 2.39 | Time to Neutrophii Recovery(>!000) - Days (from randomization) PP Population | 1 |
| Table 14.2.40 | Time to platelet Recovery(>100000) - Days (from randomization) PP Population | And the second s |
| Table 14.2.41 | Time to readse (duration of morphologic CR)- Days PP Population | |
| Table 14.2.42 | Time to relapse (duration of composite CR) - Days PP Population | 4 |
| Table 14.2.43 | Subgroup Analysis-CR ITT Population | 4 |
| Table 14.2.44 | Subgroup Analysis-Composite CR ITT Population | |
| Table 14.3.1.1 | O\·erall Summary of Adverse Events Safety Population | |
| Table 14.3.1.2 | Summary of Treatment related Adverse faent ([darubicin] Safety Population | 4 |
| Table 14.3. I.3 | Summary of Treatment related Adverse Event (Cytarabine) Safety Population | 5 |
| Table 14.3.1i | Summary of Treatment related Adverse Event (CX01) Safety Population Summary of Adverse Event due to underlying disease or other drugs or chemicals Safety Population | 4 |
| Table 14.3.1.5 | Summary of Adverse Event due to underlying disease or other drugs or chemicals Safety Population | 5 |
| Table 14.3.J.6 | Overall Counts of Adverse Events Safety Population . | |
| Table 14.3.1.7 | Summary of TEAEs by MedDRA System Organ Class and Preferred Tenn Safety Population | |
| Table !4.3.1.8 | Summary of TEAEs by Preferred Tern, Safety Population. | |
| Table 14.3.1.9 | Summary of NCI-CTCAE Grade 3 or higher TEAEs by MedDRA System Organ Class and Preferred Term Safety Population | 165 |
| Table !4.3.1.J0 | Summary of NCJ-CTCAE Grade 2 or lower TEAEs by MedDR.i\ System Organ Class and Preferred Tenn Safety Population | |
| Table 14.3.1.11 | Summary of Treatment-Related TEA Es by !'>,1edDRA System Organ Class and Preferred Tenn Safety Population | 5 |
| Table !4.3.1 i2 | Summary of TEAEs by Relationship to Study Treatment by MedDRA System Grgan Class and Preferred Tenn Safety Population | 5 |
| Table 14.3.1.13 | Summary of TEAEs by Maximum NCI-CTCAE Severity. System Organ Class and Preferred Tenn Safety Population | |
| Table 14.3.1.!4 | Summary of Treatment-Related TEAEs by Maximum NCI-CTCAE Severity, System Organ Class and Preferred Term Safety Population | |

| Tabie 14.3.1 15 | Summary of TEAEs Causing Discontinuation from Study Treatment by CTCAE and worst CTCAE grade Safety Population | |
|---|---|---|
| Table 14.3 i !6 | Summary of Treatment-Related TEAEs Causing Discontinuation from Study Treatment by CTCAE and worst CTCi\E grade Safoly Population | |
| Table 14.3 1 17 | Summary of TESAEs/Serious TEAEs by MedDRA System Organ Class and Pret"erred Term Safety Population | 51 |
| Table 14.3.i.18 | Summar: • of NCI-CTCAE Grade 3 or higher TESAEs/Serious TEAEs by MedDRA System Organ Class and Preferred Tenn Safety Population | |
| Tabie 14.3.1 19 | Summar;,- ot NCI-CTCAE Grade 2 or lower TESAEs/Serious TEAEs by MedDRA System Organ Class and Preferred Tenn Safety Population | 5. |
| Tab!e 14.3.1.20 | Summary ol"Treatment-Related TESAE/Serious TE/I.Es by CTCAE and worst CTCAE grade Safety Population | |
| Table !4.3.1.21 | Summary of TEA Ec Leading to Death by MedDRA System Organ Class and Preferred Term Safet) Population | |
| Table 14.3.2.1 | Death Listing Safety Population | TO MAKE THE PROPERTY OF THE PR |
| Table 14.3.2.2.1 | Summar;,- of Laboratory Test Results and Change from Baseline by Visit-Bone MaITO\\- Safety Population | |
| Table 14.3.2.2.2 | Summary of Laboratory Test Results and Change from Baseline by Visit-Hematology \\rith CBC Safety Population on | £1 |
| Table 14.3.2.2.3 | Summary of Laboratory Test Results and Change from Baseline by Visit-Coagulation Safety Population | |
| Tabk 14.3 2.2.4 | Summary of Laboratory Test Results and Change from Baseline by Visit-Serum Chemistry Safety Population | |
| Table 14.32.2.5 | Shifl: Tabie of Laboratory Test Results (counts) by NCJ_CfCAE grade Hematology \\"ith CBC Safety Population | 69 |
| Table 14.3.2.2.6 | Shirl Table of Laboratory Test Results (counts) by NCl_CTCAE grade: Coagulation Safety Population | //123 |
| Table 14.3.2.27 | Shitl Table of Laboratory Test Results (counts) by NCJ_CTCAE grade: Scrum Chemistry Safety Population | |
| Table 14.3.2.2.8 | Shift Tab!e of Laboratory Test Results ( 'G) by NC!_CTCAE grade: Hematology with CBC Safr:t:s Population | |
| Table 14.3.2.2.9 | Shift Tabie of Laboratory Test Results(%) by NCJ_CTCAE grade: Coagulation Safety Population | The state of the s |
| Table 14.3.2.2.10 | Shill Tabie of Laboratory Test Results(%) by NCI_CTCAE grade: Semm Chemistry Sater:- Population | |
| Table 14.3.2.2.11 | Shift Tabk: of Laboratory Results (coums) Hematology with CBC:Hemoglobin Safety Population . | |
| Table 14.3.2.2.12 | Shift Tabk or Laboratory Results (counts). Coagulation: Anti-Factor Xa Safety Population | |
| Table 14.3.2.2.13 | Shitl Table of Laboratory Results (counts): Serum Chemistry: Albumin Safety Population | |
| Table 14.3.2.2.!4 | Shiti. Tabk of Laboratory Results(%) Hematology \\"ith CBC.Hemoglobin Safety Population ion | |
| Table 14.3.2.2.!5 | Shift Tabk of Laboratory Results(%) Coagulation:Anti-Factor Xa Safety Population | |
| Table 14 3.2.2.16 | Shift Table of Laboratory Results(%) Serum Chemistry: Albumin Safety Population | |
| Figure 14 3.2.2.17 | PT/fNR over time Safety Population | |
| Figure 14 3.2.2.18 | :\PTT m·er time Safety Population | |
| Figure 14.3.2.2.19 | :\nli-factor Xa over time Safety Population | |
| Figure 14.3.2.2.20 | fibrinogen O\ver time Safety Population | |
| Figure 14.3.2.2.21 | D-dirner over time Safety Population | |
| Figure 14.3.2.2.22 | Platdel count over time Safety Population | 74 |
| Table !4.3.3.1 | Summary of ECOG Status at Screening and Vital Signs at Screening and State of Consolidation Cycle Safet) Population in | 74 |
| Table 14.3.3.2 | Shift of ECG Results Safety Population | |
| Listing 16.2.1 | Subjects Screened | |
| Listing 16.2.2 | Subject Disposition | Per |
| Listing 16.2.3 | Suliiect Treatment Aliocation | |
| Listing 16.2.4 | Protocol Deviations | |
| Listing 16.2.5 | Inclusion Criteria | 83 |
| Listing 16.2.6 | Exclusion Criteria | |
| Listing 16.2.7 | Study Population | |

| Listing 16.2.8 | Demographics and Baseline Characteristics | 9/1 |
|---|---|---|
| Listing 16.2.9 | Medical History | 97 |
| Listing 16.2.10 | Prior ;,viedication | 99 |
| Listing 1 6.2.1 1 | Concernitant Medication Post Adjection | 90 |
| Listing 16.2.12 | Post kdication | Qr. |
| Listing 16.2.13 | Study Drug Usage and Exposure | |
| Listing 162.14 | Efficacy pan 1 | A CONTRACTOR OF THE PARTY OF TH |
| Listing 16.2.15 | Efficacy part 2 | |
| Listing 16.2.!6 | Adverse E'l"ents Safety Population | 94 |
| Listing 16.2.17 | Adn:rs<: E\"ents Causing Discontinuation from Study Treatment Safety Population | 99 |
| Listing 16.2.18 | Advcrse Events Causing Interruption from Study Treatment Safety Population | 95 |
| Listing 16.2.19 | ,\dvcrse E\ents Causing Dose Reduction from Study Treatment Safety Population | 95 |
| Listing 16.2.20 | Treatm.:nt-Related Adwrse Events Causing Dose Reduction from Study Treatment Safety Population on | 6.5 |
| Listing 16.2.21 | Serious Adverse hents Safety Population | 11. |
| Listing 16.2.22 | Laboratory Findings - Bone I'vlarro\\ Safety Population | 97 |
| Listing 16.2.23 | Laborator:, Findings - Hematolog;, \\int CBC Safety Populatior. | 98 |
| Listing 16.2.24 | l,aboratory Findings - Coagulation Safety Population | 99 |
| Listing 16.1.25 | Laboratory findings - Serum Chemistry Part 1 Safety Population | 100 |
| Listing 16.2.26 | !.aboratory Findings - Scrum Chemistry Pa.rt 2 Safi':ty Population | 101 |
| Listing i 6.2.27 | PK listing Safety Population | 102 |
| Listing 16.2.28 | Vital Signs Safety Population | 103 |
| Listing 16 2.29 | ECG Results Safety Population | 104 |
| Listing i 6 <b>2</b> 30 | Physical Examination Results Sater;, Population | 105 |



### Overall Preface Tables, Figures 2nd istings

| @ | Patient :Sxcludeci from Safety ?o;;;12::ion |
|---|---|
| S | Patier.t txcl_uce.o. fro2, Ir;c:er,::-to- reat Populatio:1 (ITT) |
| & | Patient E:zcluded fro:n Per-Protoc:o.: Populatio,c |
| {?.) | Repeat: Visit |
| {W) | Patient ,:,Jithdre,-; |
| ;:, | Patient clisra:1dornized |
| c'i | lot Applicable |
| NC | Not Calculated |
| ND | Net Do:-1.e |
| NK | Not K:r.own |
| ? <ir< td=""><td>Not Recorde::i</td></ir<> | Not Recorde::i |

Page x c,f

Date Ge'l.e.::ateci.:

?rograE Nazne: Listing Source:

?aDle :;..4. Su,c;;;:ary of S::udy Co:;r:pletie>r-, and Withdra·dal

| | Cont: | :-ol | <u>-0.•</u> . | rv-o. | :-!igh | CX-01 | Tot | al |
|---|---|---|---|---|---|---|---|---|
| Patients Screened | | | | | | | XX;,: | |
| Patie,. s Rando::nized [a] | XXX | | xxx | | XXX | | >:Z:-: | xx.x% |
| ?.andom zeC ar,d not tr,::oated [bj | ZXX | xx.z%' | :,;::x | ;:x. :,;:-'i., | XXX | <u>&gt;.A. &gt;.I,</u> | ; xx | xz.:9- |
| Rar:do'''- zed ar:d -::.reateci lb} | XXZ | XZ. | ::-:ZX | X}:. Xi·, | XXX | xx.x'ic.) | XXX | x :.z::, |
| ITT ?op' <lat [b<="" en="" td=""><td>xxx</td><td>xx.x&gt;,;</td><td>xxx</td><td>xx.x%::</td><td>:.;xx</td><td>xx.x%)</td><td>xxx</td><td>XX.</td></lat> | xxx | xx.x>,; | xxx | xx.x%:: | :.;xx | xx.x%) | xxx | XX. |
| ?er ?rotoco ?opulation. [bj | x;-:x | xx.x% | XXX | X:-: | ;-:xx | xx, | XXX | xz.;-:i;) |
| Safety Pcµu atio,, [b] | XXX | xx.x°:" | XZX | xx.x ,• | XXX | xx.x0) | xzx | xx.x%) |
| Completed St:c,.d '.b] | :G{X | xx.:,J, | ;,;xx | xx.x | XX}: | ;,:x.xco) | ·,:xx | xx.xS;\ |
| Entered XXX Cy le Jl .c'is!t [bJ | XXX | xx.x'i | XXX | xx.; | XXX | ( xx.x%) | XXX | XX.X '' |
| repeat ::ora::. visi::s fro2 Dl | xxx | xx.x':1 | XX;· | <u>:</u> < | :u:x | i xx.xS) | XXX | ( xx.x%) |
| Primary ?eason fer Ea:-ly Disconti::.uation [c] | | | | | | | | |
| Reasor. | x:c: | xx.x':c' | XXX | zx.xrs | x:o: | xx.x'o | xx;,; | xx. x'o) |
| Reason 2 | :o:x | XX.X | zx:,; | XX. | XXX | xx.x'i,; | XXX | xx. x'2) |
| Reaso:i. 3 | xxz | xx.x | XXX | xx.x%) | XXX | xx.;,:S | xxx | ( xx.x%) |
| etc | XXX | :,;:x.x | x;;x | :-:x.z''' · | XXX | xx.x% | :-:xx | xx.z'2) |

<sup>[</sup>a: The den0:r,ir,ator for percentage ca cu ation s !:lase::i er, rl:J.."1lber of patien"...s sc::::eened.

Progrc.m Ne.me: D2.te Ge::.e:::-2te1:

Listing Source:

Page z 0£ y

<sup>[</sup>b] The deriorriline tor f-1]r percentage calculation s based ert. n; i, -::ber of patrier:tis rati-ticiomized ir: each gree:p.

<sup>[</sup>c] The denominate::- for percentage ca cu a-:::ion s based c., the nu."1\De::: of pa-::::.e,;ts ;...,ho did r.ot comp.Lete t:"::e study for each gro-clp. P.t:09't6:minit1g::Notes:
'Obtain··reasons £,or :early· di'SC\_onti nua:ti()n from. CRF.

#### Table 2.'<c..2.2 Surnxo.ary of Wi tC'.dra-,.•al ITT ?opc1lation

| | Co:n-<br>'.N<br>C | ∷rol<br>XXX) | | CX-JI<br>xx)<br>6; | Eigr.<br>'t = :,::xx] | cx-o::.<br>} | Overa<br>X<br>n ( ; | XX) |
|---|---|---|---|---|---|---|---|---|
| Primary Reason fo.:c Ea.:c::.y Discoc:tinuatio"<br>[aJ | | | | | | | | |
| Reasor; | x;,:x | x;;, | X:-:Z | X);. Z | XZX | XX. X;,, | XXX | XX.X |
| Reason 2 | XXX | xx. x%'• | XXX | XX. | XXZ | xx. | XXX | XX.X |
| ?easor: 3 | ZXX | xx. x'1", | XXX | XZ.X | XXX | ;,:z ,. | xx;.: | XX.X |
| etc | :-:xx | x. x-"'- | XZZ | xx.:-:"' | xxx | XX. | :,:xx | xx.x% |

[aJ ::i.e denominator for percer:tage ca.'...culatic:-. is based on :nu.:sb,2r of patie:-.::s i:n the vr:,;;n1.'.a-::io:-, set :,rithin each group.

Pi:o'g i- ing: Notes:

\_\_Obtain·.reason·s foi -.earl:,/ \_discontinua\_tiO:ri· fi-o:m CRF.

Program Name:

Listing SoJrce:

Date Generated:

Page x of y

?,epeat for the fol-2.owir,g displa :s:

Table: ':.4. l. 2. 3 Su.Tu"tlary of Wi thdra: ..-a::. PP Population

.;dd:

Footnote: la; "e denominator for :=,ercer,tage calculc.-:::io:-i is based on ;,;;.sber of patierats

t:'le ?? ?opulation set , ithin each groc:p.

Delete:

Footnote: La; The denomir.ator for per:::e::tage calculation is based on n:.......Ther of patie,;ts · :::, e:::-: Population se::: 1,,,ithi::1 each group.

Table 14. 1. 2. 4 SUJ.-:-.mary of \\*Ii thdra'.12.1 Safet'::/ Population

Footnote: [aJ The deno;r,inator for percen.-;:age calculatioD is based or. nu.-r.ber of pa.tier.ts ....-, .:::;-::e Safety Populatior:: set ,....;it.J.ir. each grou?,

Delete:

Footnote: [aJ The denominator for percentage calcu::.ati.on is based on nu.T<Der cf pac::ier,ts in ::he

Population se:: within each gro;ip.

#### Table 14.1.2.5 S·u..,--r:TI',ary O:: Screen Fai2-11::::es :='.n,olled Population

| - | rota.! | |
|---|---|---|
| Patients Sc:reened | xx;-; | |
| ?atier,ts Rancio:2.:i.2ed [a] | XXX XZ | .:,0) |
| Patients Screened bu;:: not Randcenized [a; | xx:-: XX | . Z <sup>1</sup> ⁄2 |
| Screen a ::re :reasor. LbJ<br>Sc.:::een a :1re reason :: | | :.z'i:)<br>:.x', |
| Screen a ;;.re reason LOJ | | . xS,, |
| etc | | |

No e: If a pc. ient has rrrc.ltiple sc.:::een :: ilu::::e easor,s, t'.ne patient is cou:--,ced under each screer: faiL:re reascr:. la The deno;n nator for perce:1tage calcv. a;::2.or-: s baseci or, nurrcbe!."" of patie:its enrolled.

[b Theder,om nator for percentage calc'..t at.ion s Daseci on the number of patients who got screened bL<:: r.ot rar,cio:.r.iz.eC.
?rogram c'lame:
Listing Source:

Date Gene::::ated:

age of

# Tc.ble ,::. .c.2.6 :::;urr,rrtary of Subject Disposition. - Safe":y ?ollow-up :::.:- Popula":.ion

| Dispositicr:: | :or;.trol<br>(IS co x;,::,:)<br>r, | $Low CZ-O1$ (J = z:-:z\ | ( i hx Gl | Q;rerall<br>(N xxx)<br>n (%) |
|---|---|---|---|---|
| Safety ::cllc;,-,1p perf,-:,r:;rced Dici not ccrt,plete safe fello-,-up | xxx xx.x'o)<br>xxx X'X".') | XXX <b>xx.x;/</b> xxx ;-:x.x" i | ;-: :-:X.X'c | xxx xx.x i·,<br>xzx xx.x%'. |
| orimc.r y ?.eason [aJ<br>Rease:,. | x;:x (::o:.x't) | XXX ;-::-:.·,•'i•' | xxx xx.x':i | xxx zx.x%) |
| Reason<br>?.eascn. | xxx xx. x'SI | XXX | XXX (X*:.;-:½' | x::-:x xx.xf,) |
| r.cascii. | x:·c-: | x:o:<br>x;,:x | xxx ;-:x.x'.;·,<br>xzx x:-:.x | xx;,: xx.z%)<br>xxx xx.z%) |
| Other Ongoing ;-:i th safety follow-up | :-:xx | xxx | XXX XX.::;<br>XXX :-:x.x | xxx xx.x':,,'<br>xxx xx.x%) |

The deno.r,i;:atol:' for perce::-ltages ::.s the nwcher cf patien.ts ::..r. the IT;:' Pcp,::laticr, for each Trec.t:ser:t group.

For [aJ, U:e Cenominator for percentage calco::lation is based 0:1 the r-,u..,--;.ber of patients ,,ho Cici not complete safety follo:,;; '--'P for each group. Progra Cla,ne:

L st--i--,g SO"""C"""

Page x of

#### Repeat fer the fcllow:cng dis::;,lays:

TabJ.e 10....2. 7 Sllic.:7:lary of S\;bject Disposition - Sa'.:ec:y Follow-up ?P ?c:;:;c1latio:1

Fooc::-iote: The deno:mi:1ator fer perce:1tages is the Cl..hc'..ber cf patier,ts i:1 ::he PP Populat::.on for eac:'. TreatE,ent group. Delete:

?ootnote: ?he der:omi:cator .:or percen:::ages is t'."'.e n.uillber of patier-.ts in ::he Pop'..:la::ior: for each Treat:;rrent grou.p.

Table 1 . .e:.8 Su.rr.ncary of Sc.:bject Jis;,ositio;-i - Sa::"ety Follo,,'-up Safety Population .Sdd:

Foo::rwte: '?he deno:;r;i:iator ::er percem:.ai;es is the m.;\_\_;lber of patier,ts ,..., the Safec:y ?cp;..;2.ation for each Treatr:",ent gro,.:p. Delete:

::'00-::10-ce: '.'he denomiriator for perce:-ic:ages is the r:urnber of patients " c::he :TT Pop1...;.2.ation for eech Treat:nent i;roup.

:'able 14.1.2.9 S T01a:ry of Subject Disposition:: - Long Te:er:1 FolJ..o •:--crp: !':onth X --""7 Pop--1latior,

| Ji S∷0 <sup>™</sup> ************************************ | ::c:,t:r<br>= | ol<br>XXX) | :.o'-'.'<br>(N =<br>,, !' | | $ \text{High C} \\ (K = XXX) \\ \mathbf{n} $ | :.,;- <b>C</b> ::. | o·,,rer<br>('.') | rall<br>xxx} |
|---|---|---|---|---|---|---|---|---|
| Patients with long te:rrr, fol::.ow-t.:p La) | xzx | xx.xS) | xxx | xz.x%) | :-:;-:x | '. | XXZ | )-:':' |
| ::,ong ter:n follow-up stac.t.:s '.DJ | | | | | | | | |
| Death | x ::< | :-:x.xS) | X;-:;-;: | xx.x | XXZ | _;.:;-;_;.:;) | XXX | zx.x'i |
| Ali·,se | | xx.x%) | xx;-: | xx.x | x:;:x | .:-:x.x\' | :o:x | xz.x';;c |
| Recu:::-rer::ce | :-::-;:;;: | x:-::.x":) | ;.c;:x | x; .x | XXX | Y.X.Z-, | XXX | xx. x'::' |
| | ;:;-:y | zx.x'c) | XXX | x:,:. x%) | XXX | xx.z -) | XXX | X:O<. X',; |
| For ;:atients ;,;ho died p:::-irr,ary ca.use of dea::h [c] | | | | | | | | |
| Res.so:: | XXX | XX.X | x;;:x | xz.x | XXZ | :,:x.z'C | XXZ | X;,-:. ZS |
| Reason 2 | XT" | x;-:.:(%) | xx:,: | xx.zC | XXX | xx.;-;SC | z;-:x | ;,-;x. :;o) |
| | :,:zx | xx.x%) | XXX | xx.x% | XXX | x:, · .z"., | XXX | xx.x•t' |

Foe'.' a the de;;,,o:m nator o::: pe:::-centages is t:'.e ,, "".'<Der of patie::1.ts in the ITT Populatior. for ea..ch Treat:r,er,t group.

"::he denom nator or percentage c2lculation, is :Jased on r,...; r, ber of people wi::h recorded long term fol low w status.

E''er c ::he deno:m nator or percentage calculation is based on the mucher of patients ::10 died.

D"...." s'o""e at"""" Page z of

::,ist::.r.g Source:

Repeat for the follow.ng disc:a,s:

Table "L 1.2.10 Su.mrr.ary o:: Subject Disposi tio'1 - "-'0:1.g "Ier:rr: Follow-up: I:ionth X ?P Populatio;;

Add:

For him the denorr.inac; or fo:::- percer.tages is the ::c::.cc.ber cf patients in the ?P Population for each TreatG.ent group.

'or [a], the cieT10:minac:o:::- fo:r percentages is the "7.ber cf patier,ts." the Populatior. for eac:1 Treatment grc;.:p.

Table 14.. 2. ScL--:-mary of Subject Disposition - Lo;-:; Term Follow-up: Moc:th x Safety Populac:ion F-.dd:

For [aJ, the derwc:-,inator for percer:,tages is the :1;-1,\_--:-ber o-: patier,ts ::..r, the Safety ?cpulation for each Treatmer,t g::::-o'...p. Delete:

For [a), title denominator for percenteiges is tille nurrber oil, pat2-e:1ts in the .ITT ?opulatii.or, for each !:!reat:ne::t g::::-oup.

# Table 14.1.2.12 Swill--rsary of Protocol De-v-∴ations ITT Populatior,

| ?rotocol Deviatio:c | :ontrol<br>(N = XXX)<br>n (%) | Low CX-01<br>$(N = \chi \chi \chi)$<br>n (%) | High CX-01<br>{N = xxx)<br>n {%} | Overall (N = xxx) n (%) |
|---|---|---|---|---|
| At Least l Major !?:rct :col Dev.:.at.:.0:1 | xxx ( xx.x:;) | xxx <b>xx</b> .:-:%\ | xx.z%'. | ;:xx x%) |
| 1-:ajor ?rotocol De,,iat0:1 l | xxx xx.x%) | xxx x: .:-:t1 | ;{;,;:{ zx.x% | xzz <u>···· i·o</u> ': |
| etc | | | | |

?rosr-am Name: Listing Sou:rce: Date Ge:1erate-'.:i: Page x of

Table 14.:.6
Su.i"-<-r.ary of Demograph:.,,,,....... ?opu.lati.on

| | :or,trol | Lo;-: CX-01 | Eigh CX-01 | 07erc.ll |
|---|---|---|---|---|
| | (N = xxx) | = xxx.: | N = ZXX | |
| | | !'. ( % ) | n | |
| Age Categories ea.rs n (%) | | | | |
| N | :-:xz | xxx | XXX | X>-:X |
| <category 70="" <="" e.g.=""></category> | ·-::-:;-: :,;x. | XXZ XX.X'O | XXX XX.X | XX:•· XX.X |
| <cc.tegory 2,="" :c:7c="" e.g.=""></cc.tegory> | XXX XX. | ;,:xx xx.xi} | ·-:;-:x xx.x | :-:x ·,:X.X |
| etc. | :0::: xz.zf,'• | XXX x%) | zxz xx. | ZX.X |
| ";ge ;yea.rs) | | | | |
| n | >-:xx | XZX | x;-;:x | XXX |
| w.ec.n :_s.6. | xx.x $xx.xz'$ | ZX.X XX. XX) | (xx.xx | :n:.;,;x ( ::x |
| medi.C <c:< td=""><td>;c-;:.x</td><td>xx.:-:</td><td>zx.z</td><td>; :;,:. xz</td></c:<> | ;c-;:.x | xx.:-: | zx.z | ; :;,:. xz |
| rEin | xx.x | ::x. x | $\mathbf{x}$ | Z |
| :cc.:-: | ::X | XX. | :-sx.x | X}:.;-;:x |
| Ger,der n | | | | |
| t; | :0:ZX | XXX | ;-:Z)'. | X:,, |
| 112le | :-:xx X. X'5 | ;-:xx xx.x½) | xxx x:.x) | ;-:;-:x zx. zf,) |
| Ferne.le | x:-:x | ;,:xx x x x x oo\ | xzx xx.x'i:) | XXX ;,:X. ·Sc' |

:::rote: De::,o::n.inators for percentages are based or, t:'le m:u--:-J::;er of pat.::\_ents ;, ith r,on-ITcissing dac:a in ec.cr. ?reatme;o,t g::m.ip £or t:'.e relevant -,,a:::iable.
[a] Age is ca:culated as calendar years £::::om. birth to ir:!forrr-\_ed consent

'l'a:Cle 14.1.6 SIJ . TfLar; <u>r. u.:? g. o.1:-'.v</u> IT? Populat:.on

| | :ontrol | | Lo>·i C | X-Gl | High ( | cx-n:: | Q,;erc | .::1 |
|---|---|---|---|---|---|---|---|---|
| | (N = xxx) | ( | N = XX | X) | ::::= :: | ):x) | ()i | XXXi |
| | :1 <i>i ")</i> | | n | | · ''' | e/ | | |
| MI (kg/m:) | | | | | | | | |
| n | XXX | : | :xx | | xx:;: | | :::XX | |
| meac \S .d. ·, | x; | xx.xx) | xx.x | xx.;.:.x) | X{. > | xx.xx: | XX.X | xx (xx.xx) |
| d 2" | XX.X | | XX. | | xx. | | .?::< .z | |
| | XX.X | | xx.x | | XX.Z | z | XX. | XX |
| rr,ax | xx.x | | XX. | | XX.X | ζ | zx.x | |
| ace Categories | | | | | | | | -, - |
| | :.:xx | X | XX | | XXZ | | ;.;,o: | |
| <cac:eg-ory ,="" asias="" e.g.=""></cac:eg-ory> | XXX XX. | .x% :0 | D:X | xx.:- | >:xx | xx.x ) | :-:xx | xx.x |
| <category 2,="" e.g.="" slack=""></category> | ;c-;x xx. | .x% ;- | :xx | xx.x\'· | :•:x>: | xx.zl | XXX | xx.x |
| c | ;c:x xx.x | x':: x | XX | :.:x.x'o | XXX | X1/.X%) | :o:x | XX.X |
| thnicity r, | | | | | | | | |
| N | XZX | X | :-сх | | XXX | | ;,::-0: | |
| <:,Jot 2ispc.::ic or L2tino> | :.: <b>xz</b> XX | X'S X | XX | xx.;,:%/ | X:-:X | :c,.:-c1•, | :c-:z | zx.:,:%) |
| <eispa ic="" latino="" or=""></eispa> | XXX XX. | .χ%'. χ | XX | xx.;.:'; | ;.;;-;.; | xx.x':;) | ::XZ: | xx.z%) |
| etc | ;,:XX XX | %:< X | XX | xx | xx:,: | xx. z2,', | XXX | xx.:-:%) |
| L n (%) | | | | | | | | |
| | ·0,X | X | XZ | | | | XXZ | |
| <de no·v·o=""></de> | i <xx td="" xx.<=""><td>.x%) x</td><td>XX</td><td>xx.z&gt;·'</td><td>X:-:Z</td><td>;-:x. x½)</td><td>;,:::,::z</td><td>xx.x%)</td></xx> | .x%) x | XX | xx.z>·' | X:-:Z | ;-:x. x½) | ;,:::,::z | xx.x%) |
| <secor.dary></secor.dary> | :-;xx xx. | X | :0: | xx.zS·' | x:n: | xx.x%:- | XXX | xx x%) |

Tote: Denominators form percentages are Cased on the nUJ--ibey of patie:--.ts idtl1 nor.-rr,issir.g data in each. Timeatment gro-u.p form the limit of variable. at Age is callinguished as calendar;\_tears frow, birth to .:nformed consen-r

Program Name: Listing SouYce:

Date Generat.eci:

Page z of

Table 14.1.6 Summary of Demography IIT Population

| | :<br> T T T T T T T T T T | I I I'; ;: X (.) :::::::::::::::::::::::::::::::::::: | <br>X X,<br>.;<br>b> II,<br>.f r. | ,-IX-<br>,-IX<br>I\I :=:'<br>H<br>gJ 1:<br><b>t</b> ; 10: | |
|---|---|---|---|---|---|
| | | | : | | |
| ۲, , | | X<br>::;<br>X | XXX | XXX | |
| 1 | ;;;<br>;;:<br>;<: | X | XXX | | |
| | <b>&gt;</b> C:>C | 'X' ;;; > X'; X | 2222 | XXX | |
| | : | X | KOCK | (,;;,<br>2000 | |
| 01<br>t)><br>,-i<br>QJ | | į | | S": | |
| r: l | 222 | Į. | XXX | XX | |
| '0<br>1;;<br>m 1 | xx.x | X | | XX.XX XX.XX | XXX |
| r.!<br>₩<br>₹<br>fil | жж.ж | X ><br>X :::<br>XX | 22.2 | XX.XX | |
| min | хх. х | ( :<<br>X | XX.X | XX.XX | |
| max | 26<br>26<br>26 | | XXX.X | 88.88 | |
| Height (SE) | | | | | |
| sJ | : ; ; ; ; | x<br>i | :<br>X<br>:-:: | | |
| Theat; (g o | <br>27 | X :< | X<br>X<br>; :,; | × >: | |
| median | ы | | X :- | X | |
| 17 | * >: | x<br>>: | .: X | 55<br><br>X | |
| EST | #4<br>:;; | | <br>X | XX | |
| e since ave do made | | | | | |
| 41 | 428 | XXX | X<br>X<br>:,: | XXX | |
| 'O d 3 8 8 8 | 23.33 | xx.x | X<br>X<br>X<br>Z< | :"i | |
| r.: | 22.22 | xx.x | (X:<br>:<<br>X | X ;;; | |
| | XX.X | XX.X | | | |
| | 0 00 | > >> | <b>X</b> | | |

nostate of the section of the number of patients with non-missing ' = ा: each Treatment group 19. the relevant variable of the relevant variable

Table 14.1.6 s cr,ar-:,i o:: De:r,ography .- "Oru:a.-...,

| | :or:-:::rol<br>(N""xxx;<br>n ( % i | OW CX-e::<br>(fl "' xxx)<br>::"l('i;: | High CX-Ol<br>(N " XXX)<br>r, ( % ) | o·,·e:rall<br>xxx)<br>n {%) |
|---|---|---|---|---|
| Firr,e s::nce Al·!!L dia-:;nosis n If:;\ | | | | |
| | KXX | ZXX | xxx | XXZ |
| <less 60="" days="" equa.l="" o::="" to=""></less> | :{×× xz.x%' | ;en: XZ.}:".i | XXX ZX.X) | XX:.,: XX.?:%) |
| <gre2::.er 60="" days="" than=""></gre2::.er> | ;.:XX ×};./;}' | xx.x'2' | zxx xx.x%l | :•:ZX x;,:. |
| Baseline peripheral D:ood blast ao e | | | | |
| ['7 | XXX | xxz | XXX | xxx |
| '£es | XXX XX.XS., | xzx zx.>-:'i·' | xzz: $zx.x?$ | ;-:xz: ( xx.x9;) |
| No | xxx xx.x':'s'- | xxx xx.;,:::; | xx;{ xx.x%'.· | xxx xx.x'6) |
| Baseline blasts i2 D-::::-ce marrD",.' | | | | |
| | :,:xx | XZZ | xx:•: | XXX |
| w.ean ;s.d. | xx.x ( xx.z:' | xx.x (z•:.xx; | xx.xx xx.xx) | xx. xx ( xx. x;,:) |
| :necii2:-:: | xx.x | z;c | xx.x | XY.XX |
| :T,1 <b>n</b> | xx.x | :<'.x. | XX.Z | XJ: |
| :r:ax | xx.x | xx.x | )OS. | XX.XX |
| Baseline ;:i | | | | |
| r, | XXX | XXJ: | xxx | xx;,; |
| ::r:ear. is " | xx.x ( xx. | xx.z :-:x:: | zx.xx $xx.xx$ | z;,:.x;,: xx.xx) |
| :nedia:1 | xx.x | ×{.× | ;-::x.x | XX.XX |
| rr:::n | X:{.X | ;,::,:.x | xx.x | x;,:.xx |
| rnax | XX.X | xx.;,: | J:X. X | xx.xx |

Note: Deno i::ators £0::: percentages are based on the r:.ucc:be::: cf patients with no:1-rr,issing data ' each 'Ireat:ciec,t group for ::he relevant: vari2D2.e. [a) Age is calc;;,la-::.ed as caler:dar year:s f::i-c,rr bi:cth to info:c-rr;ed consen.-::.

Prograr:t ?-iar;,.e: =-.istir:.g Source:

Date Generated:

Page of y

Repeat for '::.l e foJ.los-, ng displays:

Table 14.1 Summary - Demography FF Population

October 6 to the symmetry of propagation of the state of

Table 14. 9 s,.;;.c..,.c\ary of 1,Je:iical History IT'I ?opulation

| | :ontro | ol | Low C | X-01 | High C | X-01 | Overal | 1 |
|---|---|---|---|---|---|---|---|---|
| | (N.= X | XX) | (N = xx) | x:) | (N = XX) | k) | (N = xxx) | :) |
| | n (% | b) | n {%} | ) | n (%) | | n (%) | |
| Patie:ts Any Med."'cal histo.:::y? | | | | | | | | |
| No | XXX | :s:;,:. x'C; i | XXX | .:-:x. | XXX | xx.x'i | xxx | ,,,,, |
| Yes | XXX | :;.x.x%) | XXX | :,,:x.x | XXX | ;,:x.x<" | XXX | xx.z% |
| Medical E:'story | | | | | | | | |
| s:;,,-sterr, C-rgar: Class 1 | xxx | z·,, | XXX | xx.;,:;,; | ;,:xx | xx.x'c,,) | xxx | x:,;:. Y ' |
| ?r2fA "Pci. Term l | XXX | :,:z.x%) | XXX | xx. xi) | >:xx | xx.x | xxx { | xx.x':C) |
| c;;-:-,=,ferred Term | XZX | xx.x%} | XXZ | xx. x) | xxx | xx.x | xxx | xx.z'o |
| ?referred Term 3 | XXX | .x% | xx;,: | x;,; | XXX | XX.X'J | XXX | XX.X'0• |
| Preferred Term 4 | X:-::X | | XX>: | xx. x) | XXX | X}:. x;;} | XXX | zx. >> |
| yste;:,, Orgar-, Class l | XZX | XX.X'i;, | xxx | X?' | xxx | XX.X | XXX | XX. |
| ?re:'.erred Term l | x:o: | 3555 | xxx | x;,:,-'.•. | XXX | xx.;,: | x:-:::x | xx.x2·, |
| ?referred Term 2 | XXX | zx.zS) | xxx | xx.x't' | ;;_xx | XX.X | xxx | xx.x"c; |
| Prefer::ed Terrr, | XXX | ZX.Z': | XXX | xx.x"s) | XXX | xz.zfj) | xx:-: | Z:-::: |
| ?referred Term 4 | XXX | xx.z'i;' | xxx | xx. c) | x:o: | ZX_Z,, | xxx | x .x'c |

The der, orr, icator for percentages is ".:he m.:rrber of patients i::i the ITT 1?opc.:,la-::ion for each T.:::eatrr,ent g!!."ol.:p

Note: This table co:1t2ir:s CO'-!.n:::s of patients. a pac:.ien-: had rt.ere than o:-e r::edical history '.-,i t;'lin a preferred tenr:., ::he patient is col.ln-:.:eci only orcce ,-:ithin 2 prefeYred terE. If a patient had rr,ore -;:t'.an one ::r;edical '.'",istor:,: within a system orga:1 class, the patient is col.::lted once for each prefer:::ed term aGd 0:-1.ce fo::!', ::he sys-::em organ class.

Note: '.edD?A Version used for coding.

ProgracTL Ja"'-e: ::::ate Ger,e.::-a.ted:

Listing Source:

Repeat :'.:or the '::ollow:'..ng displays:

?age x of Y

Table 14. 1. IO Su.7.rr:.ar of 1,;edical History Safety Popc1lation Delete:

Footnote: The de:ior:i.ir,at:cr for percentages is the nurrber of patier.c:s ,,, the IT: ?cpulatic," fer each ?reatffi•"r:t group

Footnote: r::cte: T :is c:ab2.e co:1tains co:o.nts of patients. :;:fa patier::: had :nore ::han or.s- rr,edical :--listory :,;ithin a preferred term, the patient is cccml.:e:i. only cr:ce :--ithin.a p:referred te:::m. ::: a patient had more than one med.ical his::or/ within a syscier:-, o::::gan class, the patier.t is cc::.nteci once ::hor each prefe:rred c:e::n: an-::". once for the syste.cc, organ class.

;iote: i:-1:eO:J?..n. Version '..i.sed £0:::: coOir:g.

Table 14. 1. 2.1 s,.1,.Tu ,ary of Prior l'-'.eciications-f.'.!'-E, ITT Population

| WHO ATC Level 2 (Therapeutic Cl2ss) Generic Tenn ([a;) | $ \begin{array}{l} \text{::::entrel} \\ (N = xxx) \\ n (\%) \end{array} $ | Lew CX-01<br>(N = XXX)<br>n (%) | High CX-01<br>{N = XXX}<br>n (%) | Overall {N = xxx) n (%) |
|---|---|---|---|---|
| Patients with prio:::: ;,,2dicatior,- | | | | |
| _c1.1-JI | :<:-:x >:x.:,;:%·, | xzz xx.x%} | ×××·,:. X-"., | xx; |
| A'!C :Level 2 T rm | ;,;:XZ | xzz xx.z't,) | xx;: :,-:x.xS"\ | x:z. x·c |
| Ger,eric Med cation | :,;:xx | x;{;;; xx.x S) | xxx zx. ;.:% | XXX X;{.X°3 |
| Ger,eric 1•1ed cat on | z ;-:x.x%) | xx.xi ';:) | XXX XX.Z | ××× xx.x½ |
| Gere:::ic Med ca-;:_ 0:1 | xxx ;,:x.;,: | ;,;xx x;,:.x%) | XXX ZX.;,-i•' | :x:>:" <b>xx</b> . |
| Ger,eric Med cat on | ·-:xx | xzx zx.x' | XXX ZX. ;,;?,', | xx;,: xx.x% |
| ATC :.,ev-el 2 T rm 2 | xx.xi | xxz zx.x'o) | zxx xx. z'' | XXX X>" |
| Ger,ec:ic Med catio,;_ | zx.x·} | zx·,• xx.x%j | zxx zx. xS) | xxx xx.x'i-' |
| Ge,,e:::ic Med cat on 2 | XXZ xx.x% | xxx xx.x%) | zxx ( | :on: xx.xc•· |
| Gene.::ic Med cat 0:1 | XXX XX. | xxz xx.x% | XXX XX. Z".' | XXX Z.X'.'. |
| Gene.::ic Med cat on | xxx xx.z%) | xxx xx.x"o) | xxx <b>x:•:.</b> | ××× ;; X , |

The de:wminator for ::> reentages is the nu.'7ber of patients in t:';.e :::'T Po;:,ulation for each Treatrr,ent g.::oup.

Note: P:::ior sedicatio;,,s are defined as Eedications take:1 w.:.th a sta::::t and s-::.op date prier:::o the first dayof stc:dy Treat:rr,ent.

i,;ote: P. patient Eayhave ::aken :rcore than: or.e ::ceCication. Therefore, '::he sun', of nedicatio;-, counts and pe::::cent.ages ::na::, ;-,o-;: equal th',e total counts. :f a patient had :r,ore than one :meciicaticr: in a c2tegor-y, the patient is cour'.!teC or'.!ce ir. that cates,ory.

'.a] ';JEC J::::c:g Dictiona::::y (Ver-sior. xx) was used for coding.

Program, ling :NotEis-:

Note that ':thfr first rowill chan,;;e depen\_d\_ing\_o\_i\_th-e\_-ti\_t\_lE'. If- the ti"t\_l-i\_:|s'-...pr\_-or\_-medi6at:ion:...A.l-lL, -then it i.s tp\_c0;mpute\_any--priot: lML medicat-io-ris;- If- the title -is concomitant -medi(;ation-At-1L then- the req:u ired out-put is to compute any- A.ML concon-sitant :m.edication,

Program Kame: l;isting Source:

Date Generated:

Pcge x of

epeat for the followir.g displays:

Table- L1. I. ::.3 Su.,.:;r:iary of 2::::ior Medicaticr:s-:ior:. A.ML ITT ?opulatic,,

# ?able 14.l.\_:\_c: Sur.cr.arv of Cor.cor:--,i tant edica ticns-AML> I::'T Populatior

| WHOIC Level 2 ,:Ther<[_ )et:tic Class:<br>Ger,eric Te , ([a]' | ::ontrol<br>(N = XXX)<br>n {%) | Low CX-01 $\{N = xxx\}$ $n (\%)$ | High CX-01<br>(N=x=c)<br>n (%) | Overall (N=xxx) n (%) |
|---|---|---|---|---|
| Pa::ients with Cemce:":ti •,ar::.t tledica-;:io'.7 | xzx xx.x?;.) | xzx xx.x%) | :-:xx >:x.x\ · | ZXX x:>:::.X'/2' |
| A C Level 2 Te::::-I:1 | X:, xz.z%) | xxx (xx.xS) | :•:xx | xxz xz.x%'. |
| Generic Med.icat on | xxx xx.z%} | x:-:x xx. x'.,) | .z(, | ;-:xx ·-··,· >:';) |
| Generic Medioat o:-, | xxx xx.x%:, | XXX ( XX.X <sup>0</sup> i | xx.x - | ?:zx xx.xi' |
| Generic cleCicat on | :-::-:x ( xx.x%\ | x:-:x ( xx.x% | xzx :, x. x | x;t. x'ii) |
| Generic Medicat o;;. | XXX ( XX.}:'z\ | zx.x'!c | X::;, <b>XX</b> . | xz:: xx.x%) |
| A'∵C :Se·v·el 2 T rrr. | :,:xx xx.x%) | xxx ( xx. | :{. | XXX :O:.Z |
| Ger.eric 1,1ed cac: on | xxx :-:): | XXX XX.X | ·•:ZX XX.X | XXX X.Y.X |
| Generic ("Jed cat on | xzx :{ <b>×</b> .}:%) | :-:zx (xx.x%) | z:-:;-: xx.;,; | :o:x ;o•:.x |
| Generic edicatiou | xxx xx. x%) | XXX XX.X% | z;-:;.· X>:.X | zxz :,x. x?;\ |
| Ger::eric [,Jedicatio;; | XXX XX.Xi;' | XZX ZX.X'S | ZZ:< xx.;-;%' | <b>xx:{</b> X}:. x'S) |

r:,e denominator for per:cer:tages is the r. T.De,c of patients ir. tr'.e ITT J?opulatior, fer each Treatrr,er..-t gro:...p.

Note: Concomitant me,::::::\_ca-:ior,s are those ;;it:1 a star-;: date o:1 or after t.he first dose date of Treatr::ie:1t, or t:-wse t, ith c. start dat.e before the ::"irst dose date C-:: Treat::nent 2::ci c. stop date or-, or afte:::: the first dose date a:: Treatc:-ie;-,t.

Note: A patient may h2ve taken more that comparison of the compari

#### Pro9"ramtr.i11:g:Jr:ckes':

Note, that,- the first rowwill change de'pendin;/ On the title. :cf -:t e<\_titli::> is, ',Prio:t -m d.i\_cat;i\_on-:AML--,then ft is 1:\_6 o)riq:;ute \_any \_P\_i:ibr ?.ML meclicki'tion's-. If the title -is concomitant medication-AHL -then/the r-equired output is -to c\_ompute-\_any AML concomitaNt.- medication-.

Program Name: Date Gene::"ated: ?age x of y

Listir:.g Source:

Repeat for the fo:'..lo,-.:i.ng displays:

!able 14.1.14 Sur:-,r:,ar- of Concomitant Medicatior.s-non ,ruV;L ::. p-.'a-:-ior-

Table 14.1.1S

SLlirh<,ary O∷ St'-.:Cy Qrug Usage Ra-::e Ir:ductior, Cycle

ITT Populatior:

| | <u>ot-vr.</u> :<br>(N = :n: | Low CX-01 = xxx) | $i-'ligh CX-C)l$ $\{N = xxx\}$ |
|---|---|---|---|
| | | | Ce (1;) |
| Inciuc-::.ion Cy-c2.e Compl.::_ar,ce ?.ate | | | |
| *, | :-:: <b>xx</b> | ZXX | XXX |
| Initiel CX-01 | xxz xx.:<'!:) | :-:XX XX.X'i', | X:X XX.X |
| <u>C''' C'</u> , | XXX <b>xx.</b> ;-;:':; | x:::x | xxx <b>xz.z</b> |
| Cy-::.arabine | xxx x;-::. x': | xxx xx.x"i) | XZX XX.X |
| :::X-0: | x;-::x x;,·. x':, / | XXX ( z:,;. | XXZ XX.X |

-he der,ominator fer 9-2rcentages is the r.u.,2::er of patiewts ,;:it:'. nor:-rr,issing da-::.a ir, tl'''.e ITT ?OfYcllatior, for each Treatr:-,ent g-rc,::p. Study Dru.g T]sage Rate is defined as percer,tage of patiel"...ts ,;i::::. ICG½ dr...ig usage '.-:hile en the stud-y.

#### P:rcjrara,,-rting N6tes:

For:things that -::lo .hot apply; inSert

e.g. for Idarubicin + CS,tarabibe arir,,. -t-XDI:.artct initial CX0-1 would-riot :apply.

?rog::.-an Nar:-,e: Date Generated: Listing Source:

Page x cf y

?.epea:: for the fellowing displays;

:=-0.n e ·''' : .:6 S..m<l"nac; of Study Drug Usage Rate !nd,.::ct.ion Cycle ;,;;:-:r: Pop'-.:la::ion

Footnote: 1.r,e den, Jc::,ina:.or for per-ceritc.:.ges is tie nLl.a,be::: of. patients :,.,ith now-:,-.issing data ir, the :-:=r-r Population fer eacr'. Treatnent g.::-cup.

#### Delete:

Foo-::::lote: Tte ::ien-::i:;,inator for percer::tages is the "-'-'-'her of patier,::.s ;-;ith :''',ori-::n.iss.ing da:::a in the ='='T ?opulaticr, for eac::L T:.-:eau;ier.t gro,..::p.

Ta;)le : 1 2-7 S;;;,c""ary of Study Drug Usage ?..e-indvctio:1 (7+3) Cycle Safety Population Add:

.:'n'1c.no::e: The de:-.:::r:-.iwator for percentages is L;e:n;,..,ber:.,-' :: pat.ien-::::s ·;,ith non-"'-iss.ing data in the Safety Fopula-::::io:--, ::or eac'."'. Trea;:::nent gre-c.1p.

#### Delete:

Footnote: The der,...Jcc,ina::or for percentages is t:?.e n·c:...,tber of p.?.tiewt;s with :--,on-rr,.i.ssing de.ta .in the :T':! Populati.on fer -:?ac:, Treatment gro;;;.p.

Table 14.1. '1 sw,s-1.s.r:: of Study Drug Usage Rate Re-inductio::i (5+2; Cycle :11 ?o;n:.lation

Table 14.. IS Surrer:-,ac-: of St-:::Cy Drc:;g Gs age Rate Consolidation Cycle 1 Cycle ?opulation P.dd:

:'JeJte to ?rog:::ars--rte . Re:rc,cve Idar:..::bicin. For !lings that cior.ot appl:: insert "-" e.g. £or::::darubicin + Cytarabine a.::E,, CXOl and initial CXO:. would not apply.

Delete:

::-icte to ?rogra::--,.e;:: For thir.gs tl'.:at do not apply, i;-;sert "-" e.g. for ::::dar-:::.Oicin + Cytarc.bir,e ar;r., CXCl and initial CXCl ;;could ;-;o:: c.pply.

Table 14.1.2D S:...,c::1ar... of Study )rug <)sage Rate Censolidatio::i Cycle 2 Cycle I'='T Popc1latio:::.

Notice to ?rc-gittarubic.i.r,. For things that do :wt apply, insect "-" e.g. fey IciaL1bicir, + Cyt.aYabir.e a::.-rr., cxo:. and initial CXGl would not appli."

Dele::e:

Note to ?::.-ogr2rr.:::e:::-: For ::::',ir,-;s t:'.at cio not apply, i:::se::.-t "-" e.g. for :dar<J.bici:n + Cyt.arabir,e a.:::r,, CZOl and initi2: CXOl woc....ld cot app::\_y\_

Table- 4 l. 21 Su..., ar - of Stt., dy Drug T)sa.ge Rate Inductic)n Cycle ?? ?opula::io:-,

Add:

Footr::ote: T:'.e cienominator fc:::- perce:-.tages is the number of patients ;-..-ith non-rr,issir,g da-cia tl-:e ?? ?op-ulation for sea\_h T ci...cc e" g:::o'\_:;p.

Delete:

Footnote: The cienc-,-: linator fo::: percentages is t.he nurrbe;:: of patients ;;it.h :-,cn-missir,g G.at2 in t:-',e ITT Population for each Treatrr,er.t groc.:p.

Tab.le · 4 22 Sc.u,c;r,ar,.· of S::,;.ciy Drc.1-q Usage Rate Re-in:foct.ion (7+3) Cycle P??cpc:.lation

Add:

Delete:

Foo::note: Tr',e G.e:::omin2tor fer percentages is the 1;.urrbe-r of patients ',rit:'1 :::on-rnissir-,g cia::a .:.n tr',e ""77 Popc.-::lation for each Treatment gro-cp.

Table 14.1.23 SU:.1irr,ar; of Study Dr;;,,g Usage Rate ?.e-ind:..::ctio:-i. (5+2) Cycle ?P Populatior.

Add:

Footnote: Tt'.e denominator fc.::- percen::.ages is tt:e r:c1.-r.ber of patients :-:;ith :-::on-nissir,g data "" t:".e pp ?opulatio:c for each Treatment grc:.1p.

#### Delete:

Foo::.r,ote: 'Ele ds: •:.ir.: --ate:::- fo::::- =,er-cen.tages is t:-:e ::',c.i...-nber cf patients :;1ith n.'.)r:-r:,issing Cata :::he IT:- Po:!:"u'at-i., for each Treat:,rien; grot.::p.

?able """ . 24 Su.-rmar-,, cf Study Drug Usage ?..ate Cor,solid2tion Cycle Cycle ?P Popu2.a":ion P.dd:

}; ote to ?rogra,rEne.:;,:: Remove :i:daru:Cicir.. For tl'.ings t;:-;at :io not apply, insert"-", e.g. for Idarc:c~c-\_, Cytarac\_\_,e ar-, CXO=. a,1d i,1.:'.tia:.. CXOl >•muld not apply.

Footnote: The deno;ninator for percentages is ti-je r,-1:-i-bel!." ,;;f patients wiii.h nor, missing data. ::::-: the ?P Population ::'or eaci: Treatme:-:t grcc:p. Note: Duratior, of exposure calcula":eC as (date of las:: dose - date of firs::. dosei + 1.

#### Delete:

Note to Progra.rm:1er: For tilir,gs t:"",a.-:.. do not apply, .'...;er:: "-", e.g. for ::darv.bicin + Cy::arai::ine arrc,, CZO: a:-:.d initial CX-!.}l-.w-:;ld-:".ct a::.,p2.y. Footnote: The denominator for percentages is the r::.L--:-.ter of patients ,,,ith :--,-:m-missic1g dat.2 ir: the .,,,,,, Popula icr, for each Trea::.:nen.:: grot:.p. St;;;dy Drug :Jsage Rate is defined as percer,tage of pa":ie;--;ts ,rith 100'6 drc:;g usage while c;; t!"",e s::c:.ciy.

Table 14.1.25 Su,-nmary of Study Drug Usage Rate Conso.lidation Cycle 2 Cycle PP Pop;;.la.tion Add:

Note 'c.o ?rograr::c,,er: Remove Idarc:bicir:. For ti'.ings that do not apply, insert "-" e.g. ::or Idart::.bicic "" Cytarab.'.:.ne ar-rr,, CXOl arni initia::. CXOl ...;ould not apply.

Footnote: The denominate!' for percentages is -::-he nu,c-be::- patients, .. itr. r.cr,-missing data ::\_;, ::!',e ?P Population for eacr. Treatme:::it gx-0'-lp.

#### Delete:

;;ote to Prograr!",me,:: For things ::'.":a:: do :-r.ot apply, insert "-", e.g. for Id&r'-lbicin + Cytara;Jine ar;;-, cx,:::.. and i:ritial CXOl would r.o:: apply. Footnote: Tie deno,nina-cor for per.cectages is the n,.:.,-ber o:: patie:-r.ts ,,ith nor,-:nissing data i:1 ::he ITT Population fer- each ':'reat:..:ent group.

TaDle 14. 1.26 Sinnrary of Study Urug 'Js2ge Rate I:-::ciuctior, Cvcle Safety- Populac:ion

Footnote: The denor, inator for percer::t.ages is ::he nu.rr.ber c, f patien-::.s wi-:::-I', non.-rr:.issing date. -~ ::r.e Sa::'ety ?o;:n..:2-c.t.icr1 fo-r each Trea'c.r:o.eut group.

#### Delete:

Footnote: The deno;ni;iator for percentages is the nu:-r.ber of patients with :::o:,-missing date :::ri -:he ITT ?opulatio:1 for each Treat:nent gro-c;...p.

Tab:ce 14 \_\_2; Sur,t..-nar/of S'c:udy Drug Usage ?.ate ?.e-ir,duction !7+3/ Cycle Safety Population Add:

Foot::io::e: The denominator i'cr per-centages is the nu."":'l::er of pa-::ients.....; th :-ion-missing da::a : n the Safety Population for eac:-', Treatrc.er.-:: group.

#### Delete;

Foo:::cocie; :r:e denomination ::"or percen"::ages is the r:u.,--:\ber oy: patien:;".:s ,,ith ;:;on-missing data the :T? Pop'..llation for eac:J. Treatme:-,t grou::::•.

?able 2.4.. 28 Sill:crr-,ar.- of Study Dr1..;g Usage Rate ?.e-i::.d:J.ctio:1 (5+2;, C: cle Safety Population

Foctr,ote:\_".e derwminator for percentages is the r:ur:-,ber 'Jf pat::.ents ',rit:h ::-'.or:-:rro.issing da-::a ir: the Safety Popula:::ion fo::: each ' rea::rr,e;;.t group.

#### Delet:e:

Fc,otnote: ne denu:ninato;:- for percen::ages is the r:..;:-,be:::: of patients -;i;;:h non-Eissir:;g data ..., the ITT PopGlatiou ::"or each TreatEer,t g:roup.

Table 29 Su."'-0-a:::y of Stud;:- Drug Usage Rate Cor;soli6.ation Cycle Cycle Sa::"ety Pop:..;2.atioc:

c'<ote to ?::::og::::a;:-t!t.e1:: ?.eEc;te :da:::ubicir:. For things t:'1at do ::-,ct apply, ir:s,:c::::t "-", e.g. :/::sr Ida:::"Jbicin + Cy::arabine arm, CZOl aud ::.ni..tic.l CXC.l would net a.pp.:::--

"oo;;::1cte: T:',e denc::,inater for percentages is the :,u:'i'J:,er of patie:r:ts ,..;it:, r:;on-;r,issi..r:g data in ;;:he Safety Pepu.:.a":.icn fo.::: each Treatr::er:t grou)?.

#### Delete

Note to ?..::og.can-;,,er: For things ti-',at do not apply, ir,sert "-", e.g. for Ida::::'.lbicin + c:rta.::abir:;e an:1, C:-'.Ol a::.d :i.:-:itial CXGl ,,oul6. no:: apply. Foot,:ote: The denomir:atcr for.c percentages is the ;,umbe;:- cf patier,ts ;,,citi-', r:;on-recissing data ./c:-, ::he ITT Population fo::: each TreatE,er:c:: g::::oup.

Table 14\_;\_\_3Q SulG.:nary of S-:1.:ciy Drug Usage Rate Consolidation Cycle 2 Cycle Safety ?opulatior, .:6.d:

Note :::c ?ro;;::a:r:rr:e1:: Remove ::darubicin. Fo:::: things that do r,ot apply, ir-;se;:"-::: "-" e.g. fo:::::ci.arubicin + Cytarabi-:-,e arcn, cxc::. ar,d initia.:. CXGl ...;ould not apply.

?oct:note: '='he denominator for percentages is tr.e r:;u...,-nl:..:er of pa.tients ,'it!'. nor,-rr,issir:..; de.ta .... ::he Safety Pop;;;.latior: for eac:'"I T::::eat,c,er,t group .

#### Delete:

•lote to ?.cograrr.me;;; ?or ::hings t:1.at de r:ot apply, ir-:sert "-", e.g. for ::cia.rt:.bicin + Cyta.:::abine arcn, CXOl a,,c i:-,itial CXCl would sot app:y. Foo::no:::e: '::he denc-Einator ::c::: pe::::centages is the r,u.7.be:::: of patients, ..;-ith non-,c,issir,g dat2. in the ::r:r Pop'..llatior\_ for each T::::eatrr.e0.t group.

Tab::.e l,G.1.31 S1.1c-;:.,..ary of Treetmen-c Exposuce by Cycle Safety Population

| | ::or,t:::ol | Low e>::-Ol | ;:.,; gh CX-0" |
|---|---|---|---|
| | (N = xxx) | $(0: = xx;\{)$ | (N xzx) |
| | | | 0 |
| :nd'.lction Cycle T::::eatr.,e:1.t Ez3x-s·_;_re (Days) | | | |
| n | · ····· | XXX | x;-:x |
| r:-:ean 1, s . d . ) | x>:.x ( .:-::-:.xx) | xx.x ;,;y. xx) | xx.xx xx.xx; |
| mediar, | x.x | xx.x | xx.:,; |
| Din | xx.;,: | xx.x | xx.x |
| rrcax | XX.X | xx.x | XX.Z |
| ?a.tient with any dosage ::.nterrup'.::io" Proportio;, of patier::ts -",::c ::eek | xxx :,:x.:,:1;) | :-:xx xx.x;,·1 | xxx xx.xS', |
| Idar,.;bici:r. for less than 3 days | Y.XX XZ. ;,;:\; | XXX xx.x% | XXX |
| Proportion of pat.ients ,,,;-,o toc-k | | | |
| Cytarabine for less t?:an days Proportion of patients o did net | :S:XX ;.;;;.;;% | xx:,,: :-:x.;z;; | XXX ZX.x·'1 |
| take initial CXOl | xxx ( x;:. x"o ·, | XXX XX. | xxx xx.;:'o' |
| ?ro_portion of patients ,:io -::ook CXOl for .:.ess than 7 days | xx.x%1 | xxx xx.x%) | XXX XX.X-'O; |
| Proportion of pat::.ents ,,,,:o took less medicatio:r, in terr,, of recr.;.ired du.:::-ation (any of :;: a.rubici:1, | MA XX.X/01 | AAA AA.A/0) | AA.A-0, |
| Cytarabine, initia cx-o::: '3.nd cxJ:::; | xx.x'01 | ; xx xx. | ;-:xx xz. y; |

The denomi, ator for percent2ges is the nu.,-rJJer cf pa.ti.er:.".:s w:..th:10:1 rr:issir,g- data in the S2fet::,, ?opulation fo::: each '::"reat.ment group.

Note: Durat...on of ezpcsure within a period is ca.lcu ateci as ida:::e of las"..: dose - date of:'i:::s--: dose) -"- 1 for t:'wse d:::ug that ;;;e:::e ad,;i.nistereci across different ciays ar:.ci as .- day for c.hose- dr...;g a-'.i."niniste:::ed and finished within the sa:ne day. The swc: of these duration expcs;;,re within a period would form the d0::-a'..:ion of ezpos,;,re '.-lit"c.in a cycle.

Program :,;Jame: Da'.::e Generated: ?age of y Listing Source:

Table 14.1.31 St'..L-rr,arv of Treat,ner:t :Sxposure by Cycle Sccfety ?Opcilatior:

| | ::ontrol | Lo,.,,- CX-Dl | Hig;", CX-Gl |
|---|---|---|---|
| | | (N = xxx:, | \:'\1 = xx:s:· |
| | ····;-; | ('i') | { % ) |
| Re-i::1ci1.:ction (7+3) Cycle Treatrr,ent | | | |
| S>:;:-os re :Days'. | | | |
| | ;-:xx | xxx | XZX |
| near, !s.d.) | XX•X <u>Z≥1./</u> | :•:>: :{x.xx:, | XX. X;-:: .XX) |
| mediar> | xx.: | X:-:. Y. | XX.X |
| L,::_r: | XY. ;{ | :-:: <b>x</b> .x | XX.X |
| nax | xx. x | XX.Y | xx.:; |
| ?a::ie::It with any ciosag-e interr-,;.ptio:1<br>?rc-por::ior: of pat:: er,ts who took | XXX?: | xxx x;s:. x'i'.· | xxx |
| ICaru.bi_cin :'or less tha:1 3 days<br>?rop<:;rtio;:-, of pat.i.er:ts ,ho ::ock | <b>xx</b> : >:x. xi) | xzx | XXX xx. |
| C::rtarabine fo:r less tha:1 7 days ?:roportic:-: of patie:cts s-;hc did not | :-:x;,;: xy .z%i | xz:: | XXX XZ. |
| 2 A i ti=l rvo1<br>?rcpc.::-ticn of patients ;;to took CXOl | :-:;s:z | <b>xx</b> :: xx. | ;:::X:-:: Z . X, <sup>7</sup> · |
| for less than days ?:r::>portion of patie,1ts whotook .:.ess medication i::, terrr.s of eqciired | ∷XX XX.Z,, | XXX XX. | XXX X>:. x%; |
| dureticr, (a::iy of Idarub cir:, (':/tc.rabine, initial <b>ext</b> and CX-01) | xxx :•:x.x%) | xxx ;-:z.x'o) | XXX <b>xx.x%</b> ' |

The denor::inato:::: for 90rcentag-es is t',e m..L"CT.be::: of 9a-::ie:1-:::s -\_\_,:th nor: 2issir:g da:::a ir. the Safe::y Popt:.lation fo::: eacr:! Treat;-r:.ent grou,:::-.

Note: C•uratior. of exposure wit:-::ir. a period is ca:::c,:lated as (da 7::e o:: ':.ast dose - Cate of fi.::st. dose) + :: fc:::: -:::h8se d::::clg c.hat ·"·ere c.d,;inistered across diffe=ent days ar.d as 1 day fer tr'.ose drug ad.7ir:istered a:1d fi,,ished withi:1 tl":e same day. The sum c:' these duratior. expos"Ll.re ·w·it:"lir.

c. pe:://iod wc/.lld fo:::-r:, the ff0.l.""ation of exposure witl"".i:1 a cycle.

Progrell'. 1".c.;-r,e: Da o Ge...ora.-od Page x of

Listing Scu.:::ce:

#### 7able 14.1.31 Sur:unary of T.::::eatrr,ent E:xposure Cy Cycle Safety Pop"-"lat.ion

| | :::or,t.:: | :::ol | .:,C | '' CX-01 | '-<' <u>§</u> | gh CX-Oi |
|---|---|---|---|---|---|---|
| | (N "" x | xx) | $_{(N}=$ | XXX) | | xxx) |
| | | | n | (%/ | | , |
| ?.e-inductio-r;. 15+2) Cycle T.:::ea-cment | | | | • | | |
| E>:poso:re (Days) | | | | | | |
| n | xxx | | :u:z | | XX>" | |
| :-r,earc (s.d. | x:-:.: | X ZYY.Z) | ; Y | xx.xx) | X.Z | x x::.xx) |
| median | xx. | X | xx.x | | | , |
| t.""c:n | | | XX.X | : | 3 | ζ. |
| max | xx.:,. | : | XX.:- | • | x:-:.x | |
| Pat.ier1t;,:::th &n_y dosage ir.::er.:::0p-:.ion | xx;.: | xx. x%) | X:-:;: | :-::.,:_z:.;; | ;_;.,;y | X:-: |
| ?roport.io:1 of pat:.ent.s ,,:no took | | | | | | |
| IC.arub.::.cir:. to.:::: less tt:ar, 2 days | :,:xx | xx.x%} | XXX | x,:.xs; | XXX | |
| P.:::-oportion of pat1.e;-its ·,-,::to toof: | | | | | | |
| Cytarabine fo.:::- le:ss -:ta;; 5 days | :0;:;-; | XX.X | XXX | XX. )C'.' | XXX | XY.z\: |
| ?.:::opor::ion of pat .er1t.s ,,r:_o d.id r::ot | | | | | | |
| c:.ake i;-iit.ial CXO1 | | xx.x%\ | XX.•- | xx. | XX.X | XXx%\ |
| ?roportion of pat .e:-J.t.s ;-,c ".:oak CXGI | | | | | | |
| fo.:::: less than S days | '.×× | xx.x'b) | xxx | :-:x.x'o·, | xx:,: | XY |
| Proport.ior:. of patc.er,ts ,,,io -coo:-: less | | | | | | |
| medication in te::'.T.: cf equi.:::ed | | | | | | |
| duration (any cf ::: a.::::ub c1.:i, | | | | | | |
| Cytarabir::e, ini ti2. ex- ::. a:::.d CX-Gl) | xxx | :-::x.x"c) | XXX | x::.;.:%' | x;-::-: | x:,:.;-:-"c' |

Tt:e der:;ominat.or for percer:::ages is t:"",e nu.r,:cer o:: patients with r:on sissing da::a. in tt:e Safe::/ ?opc.:latior, for eaci Treatment group.

?rograra Name: Date Generated: Page of y Listing S01...rce:

Table 2-4.1.31 \$;..m',:riary of Treatment ,:posure by Cycle Safety Popul tio,,

| | - or.t:!'. | 'ol | O"w | - CX-01 | Big | -:"i. CX-01 |
|---|---|---|---|---|---|---|
| | $_{1}IJ = :,:x$ | c;-:) | \i:S = | XXX) | (1) | $_{N} = _{XXX}$ : |
| | | | n : | !%i | n ( | 'o' |
| Cor,soliOation Cycle 1 Tr:-eatrcent Sxposure{Days) | | | | | | |
| n | :o::x | | ZXX | | XXX | |
| mean is.d.' | z;,: | xx.xx | x:<. | (xx.xx) | :in:.x | xx ( xx.xx |
| median | ,,.,.,.,, | | :-:x. | | ZX. | |
| in | :-:z.x<br>XX.X | | XX.X | | XX. | |
| Pcctient with a:,.y ciosage interruption<br>Proportion of pa::ients who tock | :,:: <x< td=""><td>xx.;,,;∙,</td><td>:o:x</td><td>xx.x;:,·,</td><td>XZX</td><td>:-:x.x%)</td></x<> | xx.;,,;∙, | :o:x | xx.x;:,·, | XZX | :-:x.x%) |
| Cytarabine for less t!",arr 3 days<br>Proportion of pac:ients who did :wt | ·-:x;: | xx.'.{',: | XXX | xx.x'?) | ;:zx | ·-:x. xt |
| take ir.itial CXOl ,.opor:-tion of pc.tients ·,;ho took CXOl | :,:;,;x | }G:,x'i_,' | | xx.x% i | XXX | xx.xz,; |
| for less thaw 5 dc.ys | | xx.xi) | XXX | xx.x% | XXX | |
| ?roportior. of patients whotook less rr.edicac:ion in terms 0::. equired duration (ar.y of I-iar"J.D cin, | | | | | | |
| Cytarabine, initial ex-1 and cx-0:1 | '{×× | :-:x.xS) | x;oc ( | xx.x%) | XXX | ;.:x.x%) |

T:le denominator for percentages is the n...l..."o'.'her of patie; 1ts ,..iit'.', non missing data in ti:.e Safety ?opulatior, feJY ,22ch Trea:::mec'.t group.

Note: Dur:-ation of expos;...re within 2 period is calc'..llated as (Gate of last ciose Cate of first: dosej +1::.or t.hose drug t:',at ,;ere ad,c,inistered across differ:-en:: deys and 2s 1 d2y fer tl1ose drug acc,ir;istered a:.d finished wit:'!ir. the same day. Ihe su...; of these durc.tior:. exposure witf::ir, a period would form tl":e dura:::io;, o: e\*:pos'-'re wit:::in a cycle.

?rograrr: Ncme: Date Genera-::ed: Page ;z of

Li s -i-.g <::ou...ce

Table 14.1.31
su.,:rr,ary of Treatr:ient E:.-:posc.:re by Cycle
Safety ?opo\_.:.lc.'.:ion

| | :or.trol | Low CX-Cl | Ei;h CX-Cl |
|---|---|---|---|
| | (N "' ;,:xx) | iN " XXX;, | $\{1 = xxx1$ |
| | n (%) | n (%) | (%) |
| Consolidation Cycle <u>r"'-a """""</u> | | | |
| Szposure (Da::is) | | | |
| | KXX | %XX | x;-:z |
| r:'.ea:r, (S.d.': | XX.X X;.,;,:X;, | XX.X XX) | ;-:x.xx { xx.xx) |
| 17.edia.,, | xx.x | XX.X | ;-:-:.X |
| | xx.x | .x | :::X:.·-· |
| IT.C.X | xx.::: | ::X. | XX. |
| ?atie:n:: •,;ith ar,y Gcsage interr,1pticn | x:,;x xx. x%) | ·-::-:x xx.x'.i; | xx;.: xz.x':,J |
| Propo.rtior:. of patients who'.:ook | | | |
| Cytara:Oine for less tha,i 3 days | xxx xx.x%) | xxx :;x.xs·, | x:-:;,: x;-:. |
| ?roportion of pac:.:: er.ts ;;ho did r:ot | | | |
| <u>akA i " ia!</u> cxo | xxx x::.x'c | xxx $xx.x$ ": | x;,:>: xx.x%l |
| Proportior:: cf pc:.t:'.ents ;-,;ho took C:;{Ol | | | |
| for less "c.han 5 days | xxx xx.x:) | zx:,: xx.x-?\ | xx.x\·: |
| Proportion of pati.ents whoc:ook .less | | | |
| :r,ed.:cation ir:.terr:s of equired | | | |
| duration (any of :.darub cic, | | | |
| Cytarabine, ini'.:ial CZ- ; a:1d CX-01) | XXX XX. | zx:s: xz.z's) | :o::s: Z. |

,..;e der).cr:;icator for p'C:rcer>.c:ages is the m.:,,cDer of patie:1ts s-:.it;; r,o:n missir::g da:::a .:.f:: the Sc.fe::::y Populatior. for each Trea-.::icen-:: g::-ou;:.
:(c-te: Dura.tier; of exp:-s'.....re ,,;:ithin a period is calculated as 'Oat e c-f last dose - Gate of first dose: 1 for those drc.:g c.hat ,,-ere adrrdr::.is::.ered a.cross ci.iffe::-e:--.-:: days ar,d as l day for tt:ose drug ad.--:-,i:-:;istered ar,\_6. fir.isied ·,:ithi:-: the same day. The SW-'7. cf these du::at.ion exposure wit:h.i:--2 perioci. wc;;;lld f2r2. the du::-aticr, of e;,:pc;sure witr.i::1 a cycle.

Program Name: elate Ger, erated: Page x of
Figure 14.2.l Ove.:::all Sur,rival plot '<"T' Populatio,,



 ?rogram Name:
 Date Genera::eci:
 ?age x of y

 !.-isting Source:
 \*age x of y

Repeat for the following displays:

Figure 14. 2. 2 Overal Survi;ral plot :.'ETT ?opulatior,

Fig"Jre 14.2.3 Overal.'.. Survival p::..ot ?P ?opc:.latio,,

CIF plo': fo.::- e-,,en.:: f.::-ee s;.::rvival (f.-::orr: date of randc ization) """ Population



Prcgra:r:-, Name:

Da e Gene:ca..::ed;

?age z of

Listir:.g Sou: cce:
Repeat :for t:"le follm,ing displays:

 $-vJ''_{i}$   $f, ''_{i}$  S,5 3/2 if If

Fig.:.....1L.?:::: c::F plot for event f.cee surv-ival, '.fro; r: Gate of :::-ar:do:nization/ Q' 1?op,tlatio;:,.

Figure "1 2. 5 CIF p::.ot ::':or lec1ke:aia free s:.1rvival IIT Populatic:•L

Figu;:e 14.2.' CIFpiot. ::':or le:.1kemia free survival ?opulatio::1

Figure J..4.2.8 CIE' plot fer r.eutrophil (>500) recoste:::-y (frmn date of rar.do:r,iz2-::ion) I':"T Pop:.ila's::ic:i;,.

t=.gure ::.4. 9 CIF:pJ.ot for platelet ">2000C} recovery (from date of rando2ization) I':.-7 Pop·ula-;::i:::r Figu:::-e J.4.2.

10 CIF plc.t f.er ::eu::rophil (>1000) recogery (.fro:2. date of :::a:1ck:2.i::aticr,;, :rT Pop1.1latio"

Figure 14 CIF plc,t for pla.telet f>100000; recovery (f.co.:1 date of rar.Co,c,i=a.::icr,) ;;;,opulat::.on

Figur-2 CE' plct:'.or Ye:l.apse rs,orphelogic C?:\ ''''' - c;iw.::.a:

E"igu.re  $n.2.\sim 3$  CIF plct fey relapse 1c omp c s ....t e CR) I':T ?opulatior,

Figl:.:::-e 14.2. "L: CIF plct. ::er relapse 'corr.posi.te CR) tC'f:"'/?cp,..ilation

Table 14.2.1
Primary Outcor:-,e-CR
-,--, Ovl.'ac '1

?age x of

| | ::antral<br>(N = xxx)<br>n (%) | LowCX-01<br>(N = xxx)<br>n (%) | High CX-01<br>(N = xxx)<br>n (%) |
|---|---|---|---|
| ?chieved CR | XXX <u>X .</u> | :-rnx x. :%) | xzx (x:.z} |
| versus Cent:co:. ?ropoce:ion Difference 70'o C0Efide0ce Interval [a) p-vali.:e [b] | | x.xxx<br>>=.xx, ;;>:x:<br>.xx:•: | X.XXX<br>"Z. ;-c-:, X. X;;;<br>X.XXX |

fa] Based or. Exact. Bir,omial (Cloppec: Pearson) Co:-,fiden:::e :Z::1t.e:::7al

[b] One sided ?ishe:r Exact Test

?rcgrar:: Name: Date Ger,erate:""!

Listing Source:

Repeat fer the fo.llm,1i:::.g displays:

Tab:e 14..c:.3 Prirr, ary Outcoccle-CR ?? ?opulation

Table 14.2.4 Secondary Outco;ne-C:-ti ITT ?opu.lation

Delete:

Footriote: (a] Based or Exact Bir,c ,ial (Clopper ?ea:-sor,) Confidence Inter-9al IbJ One sided Fisher Exact Test

Tab2.e 14.2.5 Secondary Outcome-CRi -IITT Population

Delete:

2'ootnot.e: iaJ 3ased on Exact Bi:-,c::;,ial (Clopper ?earson; Confider::ce ::r::::erval

[b] oesided Fisher Exac:: Test

Delete: Footnote: '.aJ Based on Exact Binomial (Clopper Pea:::soni Confide:c:ce Ir-,::er-val [bl One side-::i Fisher Sxact Test Table . 2. Seco:i.dc.ry Ou-::corr,e-Co:;uposite CR ITT ?opv.lation Delete: Foot::1ote: '.a2 Based on Exact Binomial {Clopper ?ea:::so:1) Confidence I::",::erva.l [bJ One sided :!"isher Sxact Test Table "-'-.2.S Secondc:::::,, Outcome-Co:r,posite CR MITT Popv.lation Delete: Footncte: [aJ 3ased 0:1 2:,:ect 3io.o:-nial {Cloppe.c: ?ea:::-so:--,} Confidence ::::n'Cer-val L.OJ One sided ::'isher 2xact Test Table 14.2.9 Secondary o·c1tco2.e-Co2,posite CR PP Pop:J.lat.io:, Delec:e:

Footno::e: (a] 3ased on :Sxc.ct :Si:cwmial {Clopper ?ea:-so:1) Confidence In-:::e:-va-

Second2.ry Outcome-CRi PP Populc.tio,,

Table 14.2.6

\bJ Cne sided Fishe::: Exact Test

?able 14..2.10 Mo.:::-tality Day-30 ::::T Population

Pase of y

| | :::ontrol<br>{N = xxx)<br>n (%) | Low CX-01<br>(N = XXX)<br>n (%) | High CX-01<br>(N = xxx)<br>n (%) |
|---|---|---|---|
| Death by Day 30 | zxx x:-::.x'i} | xxx xx. | XXX -};" |
| Ve.:::-sus ControJ. Propo:::"tio,, Diffe:::ence 95::, Con::'.de:-,ce Inte.rval [a; p-value [b] | | x.xxx<br>[x.xx, x.xx]<br>x.x:-::x | 7XXX<br>XX,<br>X.X:-:X |

[aj Based en Exact Bir.orr\_ial !Clopper ?earson) Ccnf;,der..ce Interval

[bj Two sided Fisher Exact Test

?.::-ogram :';ase: ::a.te Generate--

listing Source:

Repeat for the follo;, ing displays:

Table 11;. 2. ll Mortality Day-60 rc

rcp''':: "'".:.o'

Table 14. 2 .12 I<lortality Day-SC TIT Population

Table ::\_4. 2 .13 :-1crtali ty Da:y--3C: t-'.I'::"T Populatic:-,

Table 14 . 14 Mortality Day-60 t-ETT ?opulat.i,..,..,

Table 14.2.15 Mo::::r:.ality Day-90 ME? Population

Table 14. 2. 16 Mortality 8ay-3C PP Population

TabJ.e 14.2.11 Mortality Day-6C PP?cpulatior,\_

able 2.4. 2.18 Mo::::t:alit:y Day-9G ?P Pop's.:.lat:ion

## T2ble H.2.19 Si"T>Ir,ary of O•ierall Survi,,-al 171' ?cpulation

| | ::ont.rol | Low CX-01 | Hi.gh CX-01 |
|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| | <b>n</b> (%) | n (%) | n (%) |
| Patients Died | ;,:xx xx.x%) | XXX XX. | xxx .;,d) |
| ?atie:1:::s S-cill alive | xxx $zx.xS$ | $\mathbf{z}\mathbf{x}$ . $\mathbf{z}\mathbf{x}$ . | xxx xx.xS) |
| Ti;r,e tc 'Jeath (days) | | | |
| <u>.1 r≤' œo</u> r <u>r''''</u> 1 | xx.; | | ZX.X |
| 95So Cor,f.idence :nterva: for 2'.edian [a) | -::-:.x, xxx.xJ | [x:,:y x, xxx.x) | [xzx.x, ;,:xx.x; |
| 25% and 75% (?ercentilesl | xx.:-:}:, :-:x. xx | x:,: :-:x, xx zx | x:-:. xx, ;-:y. ;-:x |
| Range 'b" | XZZ, XXZ | :-:,::,:, xx;, | X:-:X, ;-;;,;; |
| Vers'-'s Cor,::rol | | | |
| ?-vc.l;;e (Log-Rank 'lio·S:::·, | | ;{. :-:xx | XXX |

No e: Den:xninatoYs fo... perce:1t2ges are based on the rn1..7ber of patients ir:. tf;e

Pop\1la;::ion

[2. r:cpl2:r:;-t,ieier estior,ates.

[b Inc::.J.Oi::g censcreC obser7ations.

?:cograr:-, Name:

D2c.2 Generated:

Page :-: of

Lis tin,; so,.irce: Repeat for t:--,e following displays:

Tab.le 14.2.20 S·c1, -r.rr, ary of Cverall Sc:rvival 1.I TT Po,::n:..; a::i.on

Add:

FCIOt::.cte: Note: De:-wwir,a-::ors for percer-:.tages are baseC on t'...e nu.,Tsber of patieu.ts "-, the 11:ITT Popu:ation

Delete:

Foo::::.o-::e: Note: Deno,::-,ina-;::o:::-s for percer,tages c.r-e based or, the nUEber of ;::c.tients in t'.ne ITT ?opulation

Table .2.21- St:.""TET,ary of Overall Survival PP Popu2-ation

Add:

Foo-:note: Note: Denomina:.::o::s for percer,tages are based on the nUEber of patients ::.n the PP Population

De.lete:

Footnote: Note: DE-nor::cin.-:,tors :t:or percentages are based or. t:le ni\_."; \_c-r-:ber of patien-ts in the ITT Populatior,

Table 14.2.22 Ssccrr,ary of Overall Sur,ri 9-a l :Ss-::.ima-::.e ITT Population

| | | ( . ] = xxx | (N X>'.X) |
|---|---|---|---|
| 0 | ½Z½ | ;: <b>z</b> ;-: | XXX |
| to | ;:Z:,: | XXX | XXZ |
| 8 to 13 | ZXX | xx:-: | XXX |
| 1 4 :::c 21 | x;::, | XZX | ;c-:z |
| to 30 | ZX:,• | XZX | XXX |
| 31 to 90 | XXX | XXX | xxx |
| 91 co 120 <cort-;'''ii'''d></cort-;'''ii'''d> | XXX | ;:XX | xxx |

Progras Name: Listir.g Source: D2te Generated: Page x of

Repeat =or the following displays: Table ::.4.2.23 ScllLLEiar" of c-v-e::-all SurviTal -1 :Ss:::i ace tHTT Pop1..:l2ticr,

Table 14. ~. 24 s,.;..-rfary of o·verall Su::vival tc.,, :Sstir:-,ate PP PopI.<laticn

| | Cont::ol XXX) | Lo;-; CX-01<br>(N = Z:,:X;, | High cx-c:<br>'e, - ;;;; |
|---|---|---|---|
| | xxx | Z:-S:X | XX:, |
| No.::.,"7'.0er of pa::ien::s event free | XXX XX.:,• | xxz xx.x';;) | ::xx x:•:. >:', |
| r-:uri.::,er o:: patients cer:sored | zxx xx | XXX $XX.X.$ | XXX :-: <b>x</b> . |
| 2 ·· <u> :-"""</u> e | x;-;:. X | xx | .X |
| ;,·ec_a | xx. | xx. | XX.X |
| 75· pe centile | xx. | xx.;.; | XX.X |
| ?ar,ge inclc.,ding ce:1scred ·v·alues \ | xxx, ;-:x | xxx, zxx | xxx, ;,;-:x |
| Ra:-:;ge withO'Jt censored. ·values) | xxx, {;{ | xxx, xxx | xxx, x;;: |

Program Earrie: Jaire Geilerated: Page of y

Lis ti.r.g Source:

Repea:: for the following displays:

'cable 2.26 Time to Zvent Free Survival - Says LfiTT Pop·c1::.ation

Table 2.27 Time to Leuk.er:',i.a free Sur:7:..',,al - Days {::':::-o;-r, rando:;;-;\_ization) :TT ?opulat.i:-:in Add:

::,:ote to P:::ogram:ne:::: ?.eplace ever.t free ,,iti"", leukemia free

Table 2.4. 2. 28 Time t:::: Leukerr\_ia ree Sur-,,i-.;c.l - Ja.ys (frorce ::-a:.do:-s.';.;:ation) I•T?':: Pop:ilatio-, Add:

:1ote to Programmer: Replace evect free v:iti": leukemia f:::-ee

Table .2.29 Ti:ne tc Ne;;trophil ?.eco7e::'.'y \>5CO) - Days (from ::.-and.omizat.ion) :T':: Populatio:1 .A.dci:

i:::Ote to Prograrr,mer: Replace event free wit.!'. net.:trophil recc-,,e:::y

```
Table 14.2.30 Ti",e tc platelet Recovery (>20000\ - Days (f:::or:, rar;.dorr,ization) ?opu.latior. Add:
    ;,..;ote tc Prograrr.ser: ?..eplace eve:r;t free Ki"'.:h platelet reco-,.rery

Table · .--31 :'i::te tc., Neutrophil Recove:-:-y (>l.CCO) - Days ;fro-.:: randomization) ITT Popu2.ation Add:
    :::ote to ?rograrc.r:10r: Replace event free with neutropf".il recove::-y
```

Ta8le 14 Time ts platelet Recovery (>100000) - Days (froz, rar,domizatior::) Pvp...lo...:o.-Acid:

: ate "".:.o P:-:-ogra:;,,,'r,er: ?..eplace evect free \•:.: t:1 platelet recove:-:-v

Table 14.2.33 .t::::z,e::c relapse (duration c:::::rr:orphologic CR) - Days ITT ?opula.c:io:, Add:
 c'!.iote to Program:-.:r,em: ?.eplace event free . .;;ith relapse

Tc.ble : '..4. .34 Tir:, e -::0 relapse (du.ratio,, of composite CR) - Days :::T:- Population

Table c 4. 2. 35 Ti::r,e E1:er.t E"ree Survi-:, ,al - Uays (fron <u>-a...d.---....</u>; p-99ul2tic::-:

Ta:0}.e 14.2.36 T.:'\_r:-,e ::e Leukemia ?ree Survival - Days P? ?opulatio:: Add:

Ncte to Prograrr;:-ner: ?..e;,lace event free with 2-eukemia free

ic.u.j\_e 14.2.37 Tirr,e tc- '«:::-t:::-opn Recov-ery (>SGC) Days (:'.::::-c;n .rando;r:izatior,) ?? ?01>u.lation Add:
 c'iote to ?rogra::cmer: Replace event f.ree ,,;ith neutrophil recover.

Table 14.2.38 Tictie to platelet Recovery .!>2GOGG) - Days (f:::-o:rr: ra::idc:r.izac.ior.) ?? ?op-...:.atio;1

Add:

 $\cdot Note \ to \ ?rograrr:.r: -, er: :: Zeplace \ event \ free \ ; d:: h \ platelet \ ::: -ecc;; e:; :-y$ 

Table 14.2.39 Tir;-,e tc- Jei..;trcphi.l Recovery (>1000) - Days {froEt ra.::1domization) ?? ?opi..;la,:ion Add:

Note to ?rograrcmer: Replace event free ;-;i::'.", neutrophil reco;ter--.

Table 14.2.40 Tir.",e to platelet Reco'ter/ {>lOGDGO} Oays (from ra:ndornizationl PP ?opulation Add:

Note to Prog:::-arr;rr-,e::::-: Replace event free 'With platelet recc;terv

Table 14.2.½1 Ti::ree te rel2pse -'.dura-:ion of morphologie CR) - D2ys PP Pop-..;latio;;;. Add:

Note to Progra2.c--ner: Replace even-:: free ,. ith relapse

Table ; c:..1/2 Ii,;;,e to relapse (d:..:rac::ion of corr,pcsite CR) - Days?? Popu2-ation

T2;)le -,i 2 "3 ScJ.bgroup Analysis-CR :::"c':' ?opulaticc.

| | ::ontrol | Low CX-01 | High CX-01 |
|---|---|---|---|
| | (N = XXX) | (N = xxx) | (N = xxx) |
| | n (%) | n (%) | n (%) |
| Ageg.::oup: < !'J | xxx <b>xx.x°f</b> ' | zxx \ xx.x%! | xxx xx.x%) |
| 5 , Confi::ience :::r.t.e.::vc:l | (x.x>: , x.zx·, | \Z.XX , X.xx;, | ; x.xx, x.xx) |
| age group: 2 c .:, | xxx ·-·x.x-e, | XXX ( XX. ,,:':s | xxx ( xx.x%:, |
| 5? Confider,ce :::,,c.e.::vo.::. | (x.z ;-:.x:-::, | (x.xx, x.zx.) | (x.xx, x.xx) |
| '::: Ve govo | xxz xx.xS | :-:XZ <b>xx. x</b> 81 | xxx ( xx.x%/ |
| % ConfiCe,1:::-2: :::.e.::, :c: | (x.xx , x.xx\ | (x.x x. | ::;,:. <b>xz</b> , x.xxi |
| i•L: Secoredary | xxx( xx.x%; | xz:-: (xx.xSi | · <xx td="" xx.x%)<=""><td></td></xx> |
| ½ Cor::fiO.er::ce ""~e::::,-2 | (x.xx , x.xz·: | (x.:o: , x.x:<\ | (x.xx, x.xz) |
| OG: ::;; | ××× x:-:.z'o> | xxz X;-; .X"o'• | xx:-:: ( xx.x\i·r |
| 5% ConfiCence :::n-::.e.::val | (x.xx, x.xx:, | (x.xx , x.xx) | (x.xx , x.x:-:l |
| COG: 2 | XXX(xx.xS' | xxx ( x;-,.x%; | :,;xx ;-o-:.x·t |
| 5% Confidence :rc::e:c,,al | (z.xx, x.xx) | (x.xx , x.xx:, | ,:X.ZX ;,:.xx) |

::a-::e Ger,erated:

c:;; is based or: Clopper ?earsor. S:-act L...L ?rogra::n r.Jar;e: ::a-::e Ger,e Listing Sou.::-ce: ?..epeat ::or t.he followi.ng displays: Table- 1. 2. 44 S::;)g.::i-o::;p An2lysis-Corq:::osite CR :TT ?op::..2.2-:.ior

?age x cf y

Table 14.3.1.1.1

Overall Swe.rr,.ary of Adv,-erse Events

Safe::y ?opu:..ation

| | ::ontro | | Low C | | High ( | | Overal | |
|---|---|---|---|---|---|---|---|---|
| | (N = XX) | * | (N = x) | | $\{N = xxx\}$ | • | $\{N = x\}$ | • |
| | n (% | ) | n (%) | ) | n (%) | | n {9 | <b>(6)</b> |
| Patients with A:t,y Adverse Eve2ts 'ASs) | x::,:x | xx.x%} | xxx | XX. | x:-;:x | :0:.: | ;,:x;-1 | xx.x?s) |
| Patients ,-,it!l Any T.::eath,ent-Eme:r-gent | XZX | xx.x'l;) | xxx | x:-:.z%} | XXX | xx.;-: ' | ······· | :,:x.·,-, |
| Adverse Ever:ts (TEAEs) | | | | | | | | |
| Patients with A,,}' AE ty r:-:axirm.1.rr, NC::::-CTCAE | | | | | | | | |
| g::ade | | | | | | | | |
| | XXX | XX.X'ii | XXX | xx.x%) | X<'.Z | xx. xc:,: | | xx.xi) |
| 2 | xx:,: | xx.x% | XXX | xx.xS '- | XXX | XX. z 1: 1 | ;,:xx | XZ. |
| 3 | XZX | xx.x% | XXX | xx.x'i: | XXX | xx.xS | ;o::•: | XX.X".; i |
| | XXX | xx.x% | XXX | xx.xi·, | ;,:xx | xz. xli | :,:xx | >D'. :-;:%) |
| S | XXX | XX. | XXX | xx.x% | XXZ | XX.X | x;,:x | x x . z °3; |
| G:::ade 1 or .c:: | | | | | | | | |
| Grade <b>3</b> or 4 | | | | | | | | |
| Grade 3 or above | XXX | xx.z%' | XXX | xx.z't) | :-:xz | xx.x'i: | ;,;xx | xx. y>,) |
| Patients ,,,ith A2yTEAE by axinnr:. NCI- | | | | | | | | |
| CTCl-\.E grade | | | | | | | | |
| 1 | XXX | XX.X.O | XXX | xx.xi& | ZZX | XZ. | ;,;}:X | XX.X |
| 2 | XXX | xx.x%" | XXX | xx.x:;c | : <xx< td=""><td>&gt;'.Z. X'0 ',</td><td>XXX</td><td>xx.x</td></xx<> | >'.Z. X'0 ', | XXX | xx.x |
| 3 | XXX | XX.:S:% | XXX | xx.x%, | ;,:xx | xx.x'c' | | XZ.X |
| | ZXX | xx.:d. | XXX | xx.xi·, | ;-:ZX | ;,:x. | :,;x;-c: | ;,: <b>x</b> . x·o <i>i</i> |
| 5 | XXX | XX.X% | XXX | XX.X <sup>1</sup> / <sub>2</sub> '- | XXX | $XY. X\cdot \} \setminus$ | X:-:X | XX. |
| Gradel or 2 | | | | | | | | |
| Grade 3 er 4 | | | | | | | | |
| Grade 3 or above | xxz ( | x:-:.z\';) | ;,:xx | ( xx.::%) | XXX | (;,:X. | | ;,:x.::-: :) |

The derwminator f:::,r percentages is t:.-'.e r:cJ..c,ber cf patients in the Safety Populat::\_or, Cases with s.,r:kr:.owr, severity ,::e:::-e assLL-r,ed to be severe.

Program l\a:me: Date Generated: Page of Listii:1g Source:

'Zable "'1.3.1.
::::verall S ":W,a:::-y of Adve::se Events
Safety Popi..;lation

| | ::antr | x} | Low C | (x) | $High CX_{(N = xxx)}$ | | Overal $(N = XX)$ | |
|---|---|---|---|---|---|---|---|---|
| | n (% | o) | n (%) | | n {%} | | n (%) | |
| Patients with A:,•:/ A::":s leading to treatr:-,ent | | | | | | | | |
| nte:-rupti -,<br>Patients th Ar::y 7E.n.Es leading to | XZX | h.•,.f | XXX | xx.x"o | xxx | xx.x:, | X}'.X | xx. xi) |
| ec:ice : | XXX | XX, X0, | XXX | 1/.X. | xxx | XX.X½:, | XXX | Y.>:. <b>X'S</b> |
| eductinn<br>Patients with;,-, 'I'EAEs leading to | XXX | ;-;x.X'2 | xxx | ;,;;-:. >: | xxx | xx.x'i,) | xx | XX.X,, |
| -"""a-:-1·"'.". """"du,-t; | XXX | xx. x:- | x:-sx | xx. x"o i | x:-:x | xx.·,C·' | | xx.x%) |
| sco:-it.i;.;uatior.<br>atier:.ts ·.1i tr: An.,, TE.'''.Es leading to | xx:-: | S. ,., | ;-;x;-: | xx. x'i∖ | xxx ( | xx.x%} | ZZX | ·-:.%) |
| eatmer.t C.iscontinua-;::ion | ZXX | XX. | XXX | xz. xt; | :,;;.;:x | xz.x%) | ;,;,;;; | xv vSc' |
| ients with AnySeve::e Adverse E1;e:;;:.s | XXX | X X . X . 0 | XXX | xx.x';.,) | XZX | ××.× \'• | :-:X:•: | X:-: |
| tients with Any Treatmen"t-Emergent vere Adverse Events (TES.fl.Es) | XXX | xx,.).\ | ZXX | XX •.iCC | XZX | xx.x%) | | xx. |
| atier,_ts •,;i ti Any SAEs leading to dea:.h | X:-:X | xx.∷s·, | XXX | :•:x.x'i) | ;-:xx | xx.;{:±; | XZX | XX.X':0) |
| tients ••:ith A::1y TE:SAEs leading to death ::ien::s with Any S."\Es 1eading to | XXX | XX | xxx | xx. x'::) | :-:xx | XX.Z;•:; | X}:;-; | xx.x,) |
| eatment disco:-itinuac:ion<br>tt.ients witr'A:-iy TES.AEs leading to | XXX | xx.x | >:X:-: | xx. | XZX | xx.x%) | XX>-: | <b>X::</b> : :,:?;) |
| _y-;:,atment disco:;.tin.1.;at'.io:, | XXX | xx.xi' | zxz | ;.;;;,;;,;;) | XXX | XX.X | ZXX | XX.X% |
| tients with any st·Jd)' drug :-elated -"-Es | XXX | xx.x%l | ;-:xx | xx.x'i:) | xxx | XX.X | XXX | xx.x"t |
| tienc:s with any study drug related TEAEs | X;,;:S | xx.x%) | XXX | X. ;t) | XXX | XX.X | Y.XX | XX.X% |

?he denominator for percer..tages is the nu,.--n.ber of patier.t.s :,,.r, the S2fety Fopulati.cn Cases -:.,·i th unkr,o,.,n seve::ity were assu.7,ed to be severe.

Program Nar:-,e: Listing Source: Date Ger:.erac.eci.:

Page of y

Table ·," 3 sel; JL-r, ary of Treatment related Ade; er se Event (Idarubici::-i) Safety ?cpula-::=ion

| | :::ontr<br>(N = XX | | $ \begin{array}{c} \text{Low C} \\ \text{(N = X)} \end{array} $ | | $ \text{High C} \\ (N = XXX) $ | | Overa:<br>(N = xx | |
|---|---|---|---|---|---|---|---|---|
| | n (% | (b) | n (%) | | n (%) | | n (% | 6) |
| Patients '. i .I:iarubicin re:.ated Adverse Ever,ts (AES | :,:xx | xx.x%) | XXX | xx.x ,) | ZZX | *** | :x | xx.:d) |
| Patients wi Iciar,ibicin related Treatmer,t-<br>Err:ergec::: Adverse Ever:ts (TEA:'::s)<br>Patie::-,ts wifr, Idarubicirl rela':ed A:S by | XXX | Z}:::-r'''' | XX'.{ | ·-··· | x; x | zx,.·" | | xx.x%) |
| | XXX | XX. | xzx | x:,;. xSc | XXX | xx. | zxx | zz.z,}) |
| 2 3 | XXX | X};. X"" | xxx | :-:x. x> | xxx | XX. | X::X | :-:x. xi'.; l |
| | XXX | xx ,.;· | xx:,: | x:{ | XXX | XX. | :•: ::{ | ( xx. x% l |
| 4 | XXX | xx.x% | :,: <b>x</b> :,: | ·-·,.:{'i;' | XXX | x:-:.x'" | XXX | xx.xi) |
| 5 | XXX | xx.xi' | ;co: | X: .Z'c, | :,;xx | :-:x.x?o | XXX | xx.x%) |
| rade or 2 | XXX | xx.xt; | xxx | XX. | XXZ | Z' | ZXZ | xx.x%) |
| rade 3 or | XXX | xx.x%"; | XXX | xz. x?;' | xxx | ::x,-o''' | XXX | ZX. |
| rade 3 or above | ZXX | xx.xi) | xxx | x:,:. x"'· | XXX | :,:x.x% \ | XZX | xx.x%) |
| ttie:1ts wit.h Ici.ar,.;Dicir. rela'.:ed TEA£ b:,/ximu,.L, NCI-C'.:'C'''.E gracie | | | | | | | | |
| | XZX | X}:.x½; | xxx | x •:. >:'.!i) | XXX | x;,:. x'i: | XXZ | ZX. |
| 2 | xxx | xx. x:: | xxz | :,;x. | XXX | x::,. x'2) | ;,;xx | xx.x%) |
| 2 3 | XXX | XX. | xx::-: | xx.::-:':: | XXZ | xx.z?' | XXX | xx.x'bl |
| | XXX | xx.x%' | xxx | XX | XXX | Z | XXX | ( z::.x";) |
| 5 | xxx | XX. X·c | :u:z | XX.X | XXX | ×× .×''' | ;-::0: | xx.;,;'\) |
| rade or 2 | ;,:xx | xx.xt) | 1/.XZ | x;:.x | XXX | :::,: . | XXX | xz |
| rade or 4 | x:,:x | xx.:-vo' | xxx | ZZ.X | xxx | .x:.z | XXX | ;,:::, . x-3 |
| Gracie or abov-e | ;,:xx | xx.x·o' | xzx | xx.x | XXX | XX.Z | x::x | xx. x'o |

Cases with t.:.Ek::-.01-:n se-,:eri ty were assc.:.-r-.ed to be severe.

I\_'rograrrirri\_ih\_g Not.es::
Change, drug na..cH? to, !d2r't:i.bicin related.
Program Name:
Listing Source:

Date Gerierated:

?age x of J

Tab2.e 14.3... a
Su,,c:t.a:.::y of Treat:.c,er:t related t'.dverse Event (Ida:.::s.,bicir-,)
Safety Populatior.

| | ::antra<br>(N = x | | Low C | | $ \text{High C} \\ \{N = xxx \} $ | | Overa<br>(N = XX | |
|---|---|---|---|---|---|---|---|---|
| | n (% | 6) | n (%) | , | n (%) | • | n (%) | , |
| Patients 1s-ith Idarubicin related _;:::s | | | | | | | | |
| eading to treatmer;t inte::::n:.ption | >:x:,: | ZZ. | xxx | - ;>'- | XXX | xx.x%) | | zx.Y" |
| Patients ;·i th Idarubicin re2.ated 7E.;:i::s | | | | | | , | | |
| eadir,g c:o treatmer:t inte::::cJ.ptic:-:. | XXX | x:.,:. | xxx | XX.X''o'i | xxx | :-;: -•;: :<'"• | ;.;;-;): | xx.;,:'i |
| Patients ·wi tl": Idarubicin ::::elateci ASs | | | | | | | | -,,,- |
| eadir,g to t:::eatmer,t :::eductior, | XZ;,; | :-;:x. x 1 | XXX | XZ. X <sup>0</sup> 0 | XXZ | ZX.X½;, | XXX | :-;:x |
| atients with Idan: bicin ::::elated 7EA:Ss | | | | | | | | |
| eadir,g to treatment r ductior:. | x:.,:;: | $ZZ.X^{1/2}$ | x;:x | :-:x | xxx | xx.;.:'t '. | X:-:;•: | :,:.x |
| atients with Idar'.lbic n related _;;_ss | | | | | | | | |
| eading to t::::eatmer.t d scontinuc.tion | ;:x;c | X:-: | XXX | XI":.;:-,; | XXX | ( XX.Zf | XXZ | }: ,:• :;-:'.6; |
| 2tients ·,,ith :Cdc.rubic r. relc.ted 'I:S;o.Es | | | | | | | | |
| e.ding to t:::eatment ciiscontinu2tior. | z;,:x | •,:i':) | XXX | x;:,;:'o | XXX | x:,:.xt. | XXX | z:cx ,, |
| tien.ts ,,ri th Idar1;.bicir. ::::e::_ateci Sesrere | ZZX | | XXX | x::. ';) | :-;:x:>s | zx.x%; | XXX | xx.x":/ |
| dverse Events (SAEs) | | | | | | | | |
| tie1;.ts with Idan;,biciL re2.ated Treatme;;t- | XXX | zz.x'· | XXX | zx.x%) | XXX | ;.:x. | ·,:xx | ;,:x.x%-· |
| :ne:rgent Seve:.::e _;c.,.cerse Events | | | | | | | | |
| TESAEs) | | | | | | | | |
| Patients ·,,·i th IdaruOicin ::::elated SAF.s | XZX | ZZ.Y | XXX | XZ. | XXX | zx.xt' | ZZX | xx.xS:' |
| ading to death | | | | | | | | |
| atients ;, i th Idarubicir, relateci. TESAEs | XXX | ZX. <i>iZ</i> \ '- | ;;xx | XY x?,) | n.t'.• | XX.Z%' | XXX | $xx.x^{1/2}J$ |
| ading to death | | | | | | | | |
| tier-,ts with Idarci.bic E rela::ed SAEs | | | | | | | | |
| ading to treat:2ent C scontinuatic-:, | ZXZ | xz.x"∷ | XXX | XX. | x:-;:x | xx.x't. i | xx;: | xx.z |
| tients ·,,.'c t:r; Idarubic n re:2.2,ted TESAEs | | | | | | | | |
| adir,g to treatment d scontinuation, | xzx | X | xx,-: | xx.x':o i | XXX | xx.xt' | XXX | zx.x'; |

Cases :,-:itf'. \.ln>:no-.-;n severity were assu.c.ed t:o te se'.'ere.

f,rcgi::.a--riroiii.g·- -fbtes:

Cha:n9'e:-dr·u\_g -name to· Idar'v.bi:cin· r lated

Program Name: I..isting Sou:.::ce: Date Generate::i:

?. ge x of ,,.-

Repeat for the following displays:

?able 14.3. 3 Su,,cunary of T::eat:-cent related Aciverse Eve:1t (Cytarabin.e) Safe'.:y P:::ipulatior-i .i".dd:

No'.:e ':o Prog-rarnmer: Change drug name to Cytarabi::e re:ated

#### Delete:

Note to Progra:;ru-:;er: Change drug name to Idari.lbici'l related

Table 14. 3.:... s,.:rnr::.ary cf Treatment related Adve::se Event {CXOI) Sa::"'e-:: Pcp....laticr ::'\.dd:

Note -::o ?::og-::amrr,er: C:',ange d:::ug name to CXOl relate...,

# Delete:

No.:e -:.c ?rog:::.-a::rcmer: Cf::ange Crug Lame to Ida::·c1bicir. related

Table 14.3. 5 S·c1.rn,--r:a::y o::: Adve:::se Eve:it Cue to ..:.r:Cerl·, ins disease er o:::te.::: dcC'gs o:: che:r,.icals Safety Po;;mlatio:1 \_\_:i.\_ctc:

1, Jote to Prograrr -r,e.r: Change dx-ug name to Ur, derlyir:g disease or otf::er d::ugs or chemica2.s related

#### Delete:

·Jote to P:::-ogram:.--::-ter: Ctange drug ::-iame to Ida:::c:b.'cci.n related

Table 1.4. 3. 1. 6 Qveral:i.. Cmlnts of Aci.ve::se Es;er:ts Sa.:"e::y Populaticr,

| | ::antral | Low CX-01 | High CX-01 | Overall |
|---|---|---|---|---|
| | (N = xxx) | (N = XXX) | (N = xxx) | (N = xxx) |
| | n (%) | n (%) | n {%) | n (%) |
| AES | x.:-:x | xxx | Zc'.X | ZXX |
| TE.;;.Es | XZX | :0:X | ZXX | X:0: |
| SAEs | XX:•: | z:o: | ZZ: | X%Z |
| TESAEs | z:,:x | XXX | XXX | X:-cx |
| 120120 | 2., | AAA | AAA | ΧСΧ |
| T::::eatment 1'.'e ated AEs | x;.:x | XXX | xz;,: | X:,:;,: |
| T::eatsen re a ed TEAEs | XXX | xxx | x:-:x | ;,::,:x |
| Treat:c,ent re ated SAEs | XXX | xxx | xx: | x C{ |
| 'T'reatrr,ent re ated TESAEs | ZZX | | xxx | xx:,: |
| AEs leading to treatrr,ent inter::uptio:-, | | XXZ | xzx | |
| EAE 2.ead ng to treat-e1t -te:::r-pt-o- | ::xx | xxx | XXX | xxx |
| SAEs leading to treat:r,e:st inte::::ruption | XZX | xxx | xxx | XZX |
| 'iESFEs eaoi"'g to tl'."eat-rre- <u>·</u> -te:::::up | XX:-: | XX>: | XXX | XXY. |
| AEs leadir.g to treat:me:it reci. ctior, | · -·· · · · | XZX | xxx | X:,;X |
| TE.;;.Es leading to -:reatment rec\':ction | Y.X:-C | XXX | XXX | x:r:x |
| SAEs leading to treat;;r,en,:: ::::e'.:: e::ion | 1.AC | :xx | XXX | XXX |
| 'i'ESAEs 2.eading to treatrr,ent reductic-2 | X;-:X | XXX | :-:XX | )CZX |
| 120, 120 2.cuting to treatif, one reductic 2 | л, .л | AAA | ^^ | )627 |
| AEs leaci.ing "o treat.:2en.t ,'it.hd::::a1•:al | xxx | :-:xx | XXX | XXX |
| TEPEs leading to treatment,;::_t:-lcira',,'al | x;,:z | :u:x | XZX | XXX |
| S.1/2.Es leading to ':::reatrr.er::: wi. thd::::awal | :::XX | XXX | XXX | XXX |
| TESAEs leading to t.:::eatRent ,,,:i t!"'.dra,,;al | XXX | xzx | XXX | xxx |

Cases with unKnosir, se,,eri ty ·,.;e:ce assu.,-r,eC. 1:0 be seve::::e.

Progrc.:m Na;-r,e:

Date Ge;:ierated:
I.,isting Source:

?age x of y

## ':'2b:1..e 14.3.1.6 Ove!."2ll CO-:Jr',tS cf Adverse Events S2::':ety Population

| | ::antral | Low CX-01 | High CX-01 | Overall | |
|---|---|---|---|---|---|
| | (N = xxx) | (N = xxx) | xxx $(N = xxx)$ | $\{N = xxx\}$ | |
| | n (-%) | n {%) | <b>n</b> (-%) | n (%) | |
| :-:::eatrr,er.t related AEs leading to tre2t2ent | | | | | |
| nte::::-uption | | XXX | x:-:x | XXX | |
| Trec.tr:ient :::elated TEF>Es :eadir::g::o | | | | | |
| "2"°""P""t ir-t-""rup1-; | XX·•· | :-:xx | xx:,-: | XXX | |
| ::ceatr;ier.t related S.f.Es leadir::g to | | | | | |
| reat2ent interruption | | :,:z:-: | XXZ | XXX | |
| Freatr'.',ent !"elated T S1'.Es 2.eading to | | | | | |
| reat::-,er,t inte:cruptior: | 'O'.X | ·.;;;;; | XZX | XXX | |
| Freat22r,1: related P,Es leading to treatment | | | | | |
| | Z:,•·· | ZXX | XXX | ;-0:X | |
| re2trr,er.t related TEAEs leading:.0 | | | | | |
| re2::rr,e,:t red::ction | :-<;c:,-: | XX:-: | XXX | XXX | |
| Freatc,,enc: related s.n.Es le2ding to related s.n.Es le2ding to related s.n.Es le2ding to | | | | | |
| Freat:;cer,t related TESFEs leading to | | ZXX | XXX | ;,;:,-:X | |
| reatcc:er,t x-ed:ction | | | | | |
| reatce:er,t x-edciion | X:•:;,· | ;,;X:`: | X:-:Z | XZX | |
| Proof to antivolated AFO loading to treatment | | | | | |
| Freat:c.ent related AEs leading to treatment | VV . 4 | ZX:-: | xx:x | ;::,-:x | |
| Freatment :::-elated IE.t.,Es 1,c?ading to | XX:< | ZX | ΛΛ.Λ | ,,^ | |
| reathererated fe.t,,es i,c rading to | X | XXY | XXX | XXX | |
| Treat2e, t related SAEs leacing to | Α | VVI | AAA | ^^^ | |
| :::-ea.t:.,er,t wit:,ctrawal | ;;; | XXX | XXX | ;-;:xx | |
| :::eat:mer.t related TESP,Ss leading to | *** | AAA | AAA | , , | |
| reatrr,ent ·wit:'.'.drawal | ;:xx | :-:xx | XXZ | XXX | |
| , | <b>*</b> · | | | | |
| Cases wit:ti unknow::: severity we::::e ass1uned to | be severe. | | | | |
| rograrr, Name: | ::::ate G,.:me | rated: | | | :?age x of Y |
| Listing Source: | , | | | | - |

Table H.3.1.7 su..,c:nayy of T:-::Ass 8y ;'Jed.D? S System Qyga:1 Class and Fre:'.:, rred Term Sc.fety ?09ulat:ion

| S;/ste::n ():rgar. Class Cco.'Fc.reod """T | ::antral<br>(N = xxx)<br>n (%) | Low CX-01<br>(N = XXX)<br>n (%) | High CX-01<br>(N = xxx)<br>n {%) | Overall<br>(N = xxx)<br>n (-%) |
|---|---|---|---|---|
| ?c.:.ients ,;:ith Ar,y TEAI:, | xxx xx. xi\:, | >:xz xy.x%) | XZX XX. | Z>:X xx.x |
| Sys·::em Organ Class | x:-;:x :-:x.X'S | XXX XX.X'o | :-co: xz.x | xx;: xx. |
| ?re erred Terrr, | XXX XX.X% | XX}: ;:Z.X <sup>1</sup> / <sub>2</sub> | XX.X | xxx xx. |
| 2:re erred :e:rm 2 | xzz x:-:.x% | XXX XX. X;, | XXX ::X.Z | >:xx xx.x':>1 |
| P::::-e erred Term 3 | x:,:x ( xx.xS' | X;-;:Z X:-:. | x:o: xx. | xx:,;: xx.x% |
| ec:c. | | | | |
| System Orga::, Class | x:,:x xx.x | x;,;:z xx.xS) | :,:xx | :,:xz xx.>' |
| Preferred Term | xxx xx.xi | x:o; x.:,. x".;) | zxx :G:.;-::'.\ | XXX :-:x.x% |
| P;::eferred Ter:n | ;-:XX XX . X 0/; | xxx x.:,•• xS) | :-;:{;,;: <b>x:-::</b> . | xxx :,:x.xo) |
| <u>o.::e"r• e.· Tern</u> | xxx xx.x% | xxx $xY. xS)$ | ZX:-;: :-:x | xx.:,;:";\ |
| etc. | | | | |

te denominator for pe::ce?Ttages is t:he r,u.,c-ber of patienc:s in t:-,e Safety ?opu.latior,

Jote: This table cor, tc.ircs counts c:f patien::s. :£ a patient experienced more tha::: 0:12 episode of an ad rerse e7er,t, the patient is cosmted only or, ce -within a pre: erred ter:::i. =t a patient experienced :x.o::e than one adv-erse event ,;; ithin a syste:::-:. organ class, the patie,:\_t is counted or.ce for each prefeyr,=C terr.-, anci once for the sysc.em organ class.

Progo'.'a::t Na:::te:
Listing Source:

Date Generated:

Pc.ge x of

Repeat for ;:be fo2.lo;;ir,g displays:

TaO.le 14. 3. 1. 9 Sur:1.nar::/ of:1CI-CTCAS G::::ade 3 or higher TE:ASs by EedD?..A Systeo;n Crga., c:.ass and ?refer:::ed Ter.;n Safety Population

7able 14.3.1.10 S;.1..:ccmary of N:::I-CTc....:; Grade 2 or lm•.'er TE.l:..Es by l"ledDRA Syste,,"c Organ Class a2d Preferreci Terr:-; Sa::':ety Pcp-c.12.atior Delete:

Footnote: The de:1c:nir1ator for 9erce:1tages is the ;-;,-1J.--::-be;;- of patients in the sa:=ety Population

Footnote: Nocie: ":-:is table contains cm;;r-,ts of patier-,ts. :::: a patient exper1.enced more t!-,ar: 02e e;;;,isccie of ar, adverse event, the patient is cou; ted once for each prefe:-:-red ter:... ar,d o,.ce ::or tie system; o:::::a::i a patient exper1.enced more t!-,ar: 02e e;;;,isccie of ar, adverse event, the patient is cou; ted once for each prefe:-:-red ter:... ar,d o,.ce ::or tie system; o:::::a::i class.

Table 3... Il Su., J.cw.ry of Treat:nent-?..elated TEP.Es by ;;edDRA System Orgar, c:..ass and Preferreci :e::::- Safet" ?op; ; lation

TaD:e 14.3.1.... I SU:""'.rn.arv of TESA-2:s/Serio. : s ':'EA'::s b::i 1::ec:::::::... System Orgar. C2 ass ac:d Prefer::::ed '::-err. Safet: Population.

Table 14.3 ....18 Surr,l;)\_ary cf NCI-CTCAE Grace 3 er hi-:;her TSSAE:s/Serio;is TEP-.Es n,, MedD?..l'-. Syster:. C·rgar. Class ar-,d ?:r.eferred Term Sa:'..ety S1..-Population

Tab2.e 14.3.1.19 ;,rmmary cf NCI-CTCAE: Grade 2 or l.o;,re:::::::SAEs/Serious ?EA;;;;:s by I•ledD?)l.. Sys,;:er:. c,rgan Class and ?refer:::-ed 7e:::=Safety

## Ops.t:: ac. o.•

Delete:

'foot2ote; The Ce::crr,inator for perce, tages is the r,Uc-rcber c-f patier:ts in tt-e Sa:!:e::y ?opulatj on

Footnote: t ote: ';"his table contains cou.nts of patients. --= a patie2t experier.ceC. nore t:-"a::1 one episode of a,, adverse eve::t, t!", e patie::::t ;, s cou::ted only once ,,,it!", ir, a preferred ':::er2. a ;;;,atie"-.: expe:-ie:--:.ced more than one a::iverse ever.t ,,-it:-, ii:--, sys-:::e:n or;ar: c.::.ass, tr.e patient is co,; ated o:lce for each ;;,referred tene alld ::,oce for Lie s ys-:::ero, organ class.

:able "" 3.1.21 S0.nmary of TEA:::s Lea::iing to =:ea.tr. c-., I<edD A Syster:-, Orga,, Clccss <mci. ?re:'.:er.red T"errr, Safety Pcpulatior::

'Iable 4.3,\_ 8 Su.,-:-z.ary of TEJ:l..:Ss by ?referred Terrr, Safec:y Pcpula.t.:or,

| | :::ontrol | Low CX-01 | High CX-01 | Overall |
|---|---|---|---|---|
| 0.6. 11:1 | (N = XXX) | (N = xxx) | (N = xxx) | (N = XXX) |
| ?refer;:-ed '.i:'er:m | n (%) | n (%) | n (%) | n (%) |
| ?at.:ents witt. A:r:y `_::,:s_;;;; | xxx <b>xx.x%)</b> | ××× <b>xx.x</b> , | xxx xx.x".s) | x;-:z xx.x?,) |
| ?referred :er:n | xxx ;,:x.;-:(;:: | xxx xx.x:S} | ;-:xx xx.x?;) | XXX XX.X".i |
| Preferred .!:er;:n | :o:x xx.x%) | x:-::; ( :::-:.x - | x;c: xx x'oi | xxx x:-:.x", |
| ::e "'dc | xxx xx.x%) | ZXX XX.X°" | :-:xx ZY. x'i;c) | $xx;=: x:s.x\{;$ |
| ?re erred '!'err:-, | xxx x:.x%) | x:-:x xx. | XX.X'S) | xx:-: x:-:.x%) |
| Pre erred 1er- 5 | xxx (xx.x%) | xxx :-ex. | xx.:-:%) | xxx xx.::%) |
| Pre err:ed ?er::, 6 | xxx xx. xs) | zxx :.:x.::<:' | XXX xx.x'.3) | XXX ZX. |
| Prefer:::-ed Ter::-,<br>e-:c. | ;,:;-:x xx.xi) | xxx xx.x"o) | ::x;: xx.x%) | xxx zx.zt,) |

The Cenc,dn.ator for pe::.-centages is the :r.u.,J::er of patients -c.:-',e Safe-::y Popc.Jlatior:

lote: This ,:able co,.ta.ins co.mts of.pa::iem:s. If a patient ezperi.er,ceci :ncre -::l',a;;; one episode of an adv-erse event, the patient is courcted only once within c. pre:Z:erred t'erm. ?rogra,r, ;"ame:

.-.3-!-:7a s :ir e-

Date --- Ger: er-a-::, ed:

?age of

?able 14.3.1.12

'o'oo-rt,rr,ary o= ?EAEs by Relationship to Study Treatment by :"iedD?.P... Systerr, Crgar, ::lass ar.d Preferred Term Safety· Population

| System Organ Class | ::antral | | Low C | CX-01 | High ( | CX-01 | Overal: | 1 |
|---|---|---|---|---|---|---|---|---|
| Preferred Te= | (N = XXX) | | (N = N) | (XX) | (N = xx) | <b>c</b> ) | $_{(N} = _{XX}$ | X) |
| Relationship to Study Drug | n (%) | | n (% | %) | n (%) | | n (%) | |
| ?atients with J:ny T:::AE | ;.:;,;x x | x.z"s | XXX | XX.X | ZXX | xx. ;-d;: | XZ;; | ;s:x.x%) |
| Idarubicin related | ;,;xx x | x.xS | XXX | XX.X | xx;,: | xx.x'i | XXX | XX. |
| Cytarab ne relac:ed | XXX | z'i | XXX | XX.X | :•:;,:;,( | xz.x' | ;,:xx | XY.X's) |
| CXOl re ated | ;,:xx X | xx.;,:% | XXX | XX.X | XXX | xx. | :•:XX | ;•:x. ;s::;,) |
| Underly ::i.g disea.se o:: cthe:::- ci.ru;s or chemicals related | ;,:xx x | xx.x's | XXX | XX | :•:.:cs: | XY . <b>x'i,</b> , | XXX | x:-:.x%) |
| Not Related | <b>xx</b> :.: | Σ;∷.Ζ:;,· | XXX | x:s. x o) | XXX | ,,,,=, | xx;, | ZX:•·'.' |
| System Organ Cl ss l | xx:<'. × | ::{. Y'''' | XZX | xx.x%) | ;,:::;( | ZX. | | x;,:. x':;' |
| Idarubicin re ated | XXX X | xx.xii | XZX | xx.:,:\'.' | XXX | ;{;,;. x'c | :-,::{;< | >:. x ,) |
| Cyta:cabine re ac.ed | XXX X | x.xS:i | XXX | xx.x% '- | XXX | ZX. X <sup>0</sup> 0·: | ;-::-,:x | xz.x'o) |
| CXOl releted | >:XX X | XX.X·S | XXX | xx.x'i'-) | x:xx | $zx.x\cdot3'$ | XXX | XX. X, |
| Onderl ir.g disease or ether 0.n.::gs c:c cherr,ical related | xxx x | "×.x"> | XZX | xz.x;) | xx;.: | xx.x"': | ·,:x:•: | ;,;x.x'i:) |
| NotRe ated | X/'.X X | х,.;,., | XXX | xx.;,:;;;) | x;:x | XZ. | XXX | xx. ::"t) |
| Preferred TerE 1 | XZ:-' ; | {X.Z'C | XXX | xx.x%) | XX;,: | XX. | | :::x.;s: |
| Idarubicir, related | x:-cx | ×t) | ;.:xx | ( xx.x% | ;:;-,:x | x;-,. ;.:" ' | x:, | ::x.x%'. |
| Cytarabine related | x; x x | (X.X':S' | X)SX | XX. x';; | ZXX | xx.x - | xx;,: | :,-:x.x |
| CXDl related | XXX X | xx.x":o} | ;,:xx | (xx. xS: | XXX | ;,:x.x';,,; | | XX.X |
| Ur.derlying diseese o.:: other dn:gs or chemica.:s related | xxx ( xx | x.x"c' | XZX | ( zx.x% | X | xx.x%,; | XXX | xx.x |
| Not ?.elated | xx:s: x | xx.xc:,·, | XXX | :s:x.x%) | X.:S:X | xx.x:: | XXX | xx. x%-) |
| etc | XXX X | x.::'c\ | XXX | xx.x%) | ;,:xx | :-:x.xs; | | xx.x%; |

The der.ominator for pe:-centages is the :::.L,Tu)er of pat.ie2ts in t:1.e Safety ?op,,-,latiori

Note: This table contair,s cou:ats o:: pati,,nc:s. 2 patier:t e:-:perienced more '...lo',c.n one episode of a 7-;;:\_n\_s, the patier,t is CO"...lnted only once ...,ithi:;1 a preferred te::JT, ac.d o::ce for c:he system organ class.

?rogra:n Na:r'.e: Dete Ger;.erated:

Listing Source:

:2age x of

Table :C.4.3.1.13

SUc.v:-cr.ary of TEA:Ss ;;,,,; :-,Jaxi ,,...:.,, IiCI-C':'CAE Severity, System Oz:-gan Class and Preferred :e::::::\
Safety ?opul2-:::ion

| Syster::, Crg2:1 Class<br>?refer::eci Te::-m | ::ontrol<br>(N = XXX) | Low CX-01 $ (N = xxx)$ | High CX-01 $(N = xxx)$ | Overall {N = xxx) |
|---|---|---|---|---|
| <u>l.C-'*'-"" .:0 ,.ec</u> j | n (%) | n (%) | n (%) | n (%) |
| ?atient.s w:'t.h Any TEAE | xxx | ZXX XY X':',' | xxx <b>xx. x%'</b> . | :-:xx ×)'.x>) |
| Overall | xxx :.;z.·.· | <b>x</b> :,:. x | xxx xx.xS | :,:x :,:x.;,:'.5) |
| 1 | x:,:z zx.:::'.' | ZZX XXX'<;, | xxx xx.zo.:, | xxx xx. x':c |
| | χ:-:χ X>'.xi' | xzx zx. x%1 | :s:xx xx.x%: | · · · - · · |
| 3 | $xx.x$ : {x.:r | ZXX XX. | >:xx xx.x'2 | :c-:z :•:x.x"1;) |
| 4 | XXX XX.X" | zx;-:: | xx.;,:% | xxx xx. x':c |
| S | xxx ;,;;{. | xxz x:-:. x'c) | :-:xx zx.x% | XZX XX. X:-, |
| Syst.ecc, C::::gan Class 1 | xxx zx.z | xx:•: | $\mathbf{x}\mathbf{x}$ $\mathbf{x}\mathbf{x}$ . $\mathbf{x}'$ | x:.;;;; zx. x'i' |
| Overall | xxx :-: <b>x</b> .:,·" | ZXX X/:. | :-:xx ( x%) | $_{\rm XXX}$ ${f xx}.$ |
| | xz;t xx. | .:-:xx xx : {-\ | :-:xx x;x'o | XXX } •• '- |
| 2xxx | :s:x. ·,'C \ | XXX XX.X | XXX xx.xS;, | ZX: :-:X );/;- |
| 3xxx | xx.x'c' | xxx xx. z | xxx ;o:.x ; | x:-:x xx. x% |
| 4 | X:.;X ZX.Z'°c∖ | xzx xx.x | XXX X;,:. | :-:xx |
| S | xxx | ;.:: <b>xx</b> | ;.;xx xx.x½) | :-:xx x:-:. x?,;. |
| ?.referred Terce, | xxx xx. | X:-0, ::o:.x | xxx xxx%) | xxx $xx.x$ |
| o,rerall | XXX ( x;;. ;;-l | xx;{ xx.:-: | XXX (:{X.;.:\;;, | :,:xx X}:. Z |
| | ××× :-::x.x | :,:XX XX.Y | XXX XZ. X'i | :0Z:-: XZ.X |
| 2 XXX | >D•:.x'±' | XXX XX.X%' | XXX XX.X'S | XXX ; $Z.x$ |
| 3 XXX | XX.X": | XXX Z:X. X-'' | XXX xx.x% | xx.:-: ××.×5 |
| • | xxx xx. | XXX XX. X",' | xxx $x::.x'$ , | zxx xx.x'.'; |
| 5 | ××× :-:x. | xxx xx.xS, | xxx xx.x% | xx:,: z; Z'Si |
| etc | <b>XXZ</b> ;-:z.:,:··, | x;-:x xz.z* | xxx xx.x%1 | xx:,: /;x.z ;) |

The denc::-,in2::or fo:::- percentages is the nursber 0=... patients in the Safety Popc.:lation

?rog:::-am N'ame:

Lis::ing Source:

?.epeat for the fellowing displays:

Date GeD.era"c.ed:

?a,;e of

Note: Patients with :r,issir:g "laxi:r,u.Te. se-.cerity are co,.mted in L;.e Jve:::-212- category only. l = t-:rild, 2 = ;:,Joderate, 3 = Severe, 4 = Life Threatening, 5 = Dea"::!",.

Note: This table contains counts of patients. a pa::::.ent e:-:perienceC more th2:1 or.e episode of ar, adverse evenc., ;:h.e patient is cm.:nted o:lly-once witLi.n a preferred tern and for ::he episode ,1:::h ::he r.:a;;ionc:.c-n seve:::-i::y. If a patient e:<perienced more ::han one acive:::-se eve:1t witi'.in a system organ class, the patient is counted or,ce fo::.- each preferred term ar,d or.ce for the system erg a;,, cl.ass.

Tab:..e 14.3.1.::\_.:; SLL.'Tu.--::-,a:cy of Treatme::.t-?.elated TEF>,Es by ;;,;aximw,, I c:::-CTCAE Seve:city, Syster:"c O:cgan c::\_ass ar,d ?reference Term Safety Pope:.lation Acid:

Note to ?::::og:carr:!T,e:::: Replace TEAE by T:::-eatne;:i.t-Related TEAE

Table::.4.3.1.15

,\_\_Tu":',ar)" O=: ?EAEs Ca,;.siTJ.g Uiscoc,tinuation from, S-;:udy Treatment Dy CTCF-.E and ,mrst C CAE grade
Safety Pop·c1lation:.

| c::CAE ca tegor""y<br>(alphabetical order) | 'a2-p::abetica.l<br>a.c.s,it-l-:<br>C?CA:S category:, | <u>T″ C₁C::::</u> ;<br>grade | ::ontro<br>(N = x<br>n (% | xx) | $ \begin{aligned} &\text{Low } 0 \\ &\mathbf{N} = \mathbf{x} \\ &\mathbf{n} \end{aligned} $ | - | High C<br>(N = xx<br>n (%) | | ()-,1era<br>(N = xx<br>n (% | ×) |
|---|---|---|---|---|---|---|---|---|---|---|
| Nu:tber i>.;) of subjects | | | | | | | | | | |
| A2-l C'I·CA:C:: categories | Any | Gracie | x:o: | xx. x'i i | XXX | XX. | ;,;x;: | | XXX | x:,s.z,;; |
| | | <u>. ∵::a</u> , | XXX | x-:.x | XXX | :s:x. | ZXX | ZX | ·,:ZX | xx.x\' |
| | | Gracie 3 | XXX | xx.x; | xx;-: | ;,:x.x',· | XXX | xx.:·"·' | XXZ | $\times \times . Xi$ |
| | | Grade | x: <x< td=""><td>ZX .X</td><td>XXX</td><td>xz. ·, 0,</td><td>XXX</td><td><math>xx.x' \leq S \setminus</math></td><td>XXX</td><td>xx.:,s(:</td></x<> | ZX .X | XXX | xz. ·, 0, | XXX | $xx.x' \leq S \setminus$ | XXX | xx.:,s(: |
| | | Gracie | х:, | ;:X | XXX | ;,:z. | xx;,: | .:,d | :{XX | zx.x's |
| ' 'A Cc•- gov | Pn.y | Grade | ;,c,:x | x;,:. x%) | XXX | xz.;-;º · | xxx | :ZX. | C{ZX | xx. |
| | | Grade | XXX | Y.X. | :•:xx | ;-n:. | ;,:zx | xx.x-s' | XXZ | XY .xf;) |
| | | Gra6e 3 | x:o: | Y.X. | XXX | xz.x,,·, | XXX | xx.x:) | ;,:zx | x:s:.x{,' |
| | | Gl'.aC.e 4 | XXX | ZX. ;,·>·- | XXX | xx.x".:, | XXZ | zx' | ;-:zz | xx. x\'i' |
| | | Grade 5 | ZXX | xx. x'c; | XX;-;: | <u>u: x'.</u> | XXX | z:,:.Y | | xx.x-:, |
| | <u>c·\ i -· · CAE</u> <b>err</b> :-, | Gra6e | x;-::x | xx.;,; | XXX | xx.•.,::, | xxx | ;,-:x. x::; | :,:zx | |
| | | C;l'.aCe | XXX | XX.X | XXX | xx.x | xxx | xx.x') | xxx | xx.xi; |
| | | Gracie 3 | :-:xx | x;,:.x | XXX | xx.;,-: | XXX | xx. | XXX | zx.x;) |
| | | Grace 4 | XXX | XX. | XXX | x_;x | xxx | xx.x%) | xx:<: | ·•·x. xs1 |
| Z::c | | G:rade 5 | XXX | xx. :-:-Z1 | XXX | xx.z"o'. | XXX | :n:. × <sup>0</sup> 0 \ | ZX;-: | ;-::;-:. x%1 |

The deno:r.ir.a.toY foY percentages is the nu.,.Llber cf patier,ts in the Safety ?opc:lation

::ote: Tt.is table contains counts c:f patients. If a pa-;:ient experienced r:.\Orf, than one episode 0f an adverse ever:t, the patient is coc:r,ted onl.
once within a prefel'.red ter:r, a patient expel'.ie::ced r:corF> than one a.dverse event within a syste:r, ol'.gan c2-ass, t le patient is cointed cnce
for each preferred ter::I acci. once for the systeB organ: class.

?rograr:: ?::a;∴,e: D2t:e Generated: ?age z of

Listing S01..:rce:

 $Table\ 14.3.1.15\\ S,;;"eL-n.ary\ of\ TE.D, Es\ Causing\ : Jisecntinuation:\ frort:\ Study\ T.reatment\ n\cdot.,\ CTCAE\ and\ worst\ CTCAE\ grade\ Sc.fet\\ ?op:...la::ion$ 

| | :ontro | (XX) | Low C | cx) | High C | | Overal<br>(N = x | cx) |
|---|---|---|---|---|---|---|---|---|
| | <b>n</b> (% | ⁄o) | n (% | ) | n {%) | | n {% | 5) |
| ?atien::s w'. t:h Any AEs leaciing to treatment | | | | | | | | |
| | XXX | xx.:-cs' | xxx | z:,:. x%' | xxx | zx. xf,) | x:-:x | XZ. |
| Patient.s ,;;ith Specifie::i TEA:Ss .leading to c:.reat2ent | | | | • | | , | | |
| ; nc'''- ''-t-''' | XXX | x:-:. xS', | xxx | xx.z':i | xx:,: | xx.x'-5) | | ;,:x .x%) |
| ?atie:1ts W.:th Any AEs leadin9 to treatment reduct.:on | XZX | xx. x'c' | xx;-;: | xx.z% | XXX | xx. | | ;,:x.x\) |
| ?atie::ts ,-,ith Specified TEAEs leading to ':.reatrr,en:: | | | | | | | | |
| ,ed1,;.ct.::.c.: | XZX | xx.:-:"" | XXX | zx.:,%) | :-:xx | ZX. | zx:,: | X:,;.X::,J |
| ?atier-,ts 1-;ith Any AEs leaC:in;; to treat.me | | | | | | | | |
| a : s" : <b>L.<a< b=""></a<></b> | XZX | XX X'.O i | XXX | xx.x'.i;) | XXX | XX.X'O | | XX.XS) |
| Patients c-;i th SpecifieC TE.AES leading to treat:nent | | | | | | | | |
| ri.is co:,ti::::a ti on | XXX | :cs:. x':s': | xx:,: | xx.zSJ | ZX:-;: | <b>XX</b> . (C) | Z{X | xz.:·d;) |
| Patients -1itD Pny se,h:cre Fd·,,erse Svents (SAEs) | XXX | xx. x, | /:x;,: | };;:.x'/;) | ZXX | i":x. z'S) | Z:-:Z | XX. X'o i |
| Patients ; •: ith Speci-::ied ?reat::r:.en:::-i::merge:-i.t Severe | | | | | | | | |
| Adverse Events (TESAEs) | XXX | X}:. | XXX | xx.X's) | XXX | XX. | xx:-: | xx.x%) |
| Patier:ts - '- Any S.AEs leading to death | XXX | X:Z. X; °' | xx:;: | xx. x"o) | XXX | xx.x0) | XXX | xx. x°s) |
| <u>P-3+-i e'''':S ::-o Sp''',; -!-i e; 7'''\$:'\Sc,</u> lead.1:.g to death | XZX | z:-: ,,, | | ;.;x. x'h) | ;;xx | ;,:x.x%) | z;-:z | X>:. x".,) |
| Patier:ts ,.;.ith P.:1y SAEs leadi:,;; to treat:r,ent | | | | | | | | |
| ciiscor'.!tinuation | xx:<: | /o'x.xx | xxz | XX. | xx;-: | xx.x0 | ZXX | zx.x"o) |
| ?atiects with Specifed TSSAEs leading to treatment | | | | | | | | |
| dis ontirn.;ation | %XX | 30 -1. X -1 1 | XX)'. | x:,;.xS' | :;.:x;z | xx.x': | XXX | :e:x. x%) |
| Pat e:-i.ts ·,•:ith 2"-Y study Cn:g related AEs | xzx | xx.xi': | zxx | xx.xi | XXX | xz.x%) | XXX | xx.x •'• |
| Pat e:-i.ts wit:1 any study Cr g :::-elated specified TEAEs | x:-;:x | XX.X°. | xzx | xx.x-\::\ | XXX | x;x%) | z,:x | xz.x%] |

The der:.orr,::r:.at:Jr fa;:: per:-centages is t:-.e nuw.ber cf pat.i.ec.ts ir:. the Safety ?opulation

Page z of

Prog::a:s 1\ar:-,e:

Date Generated:

Listing Source:

Repeat for the follo,, •ing displays;

Table :4.3. 16 Su.--:i.mary of TreatE",ent-Related TSAEs Causing Disco:,-;::inuat.i.on frorr-, St,.;.dy T:::-eatmer.t Dy CTCAE and wc.::-st C?CAE g.cade Safe-:::y

<sup>\*</sup>cte; This table contains 20......its of patients, If a patie:ct experienced :w.ore than one episode or:ce ;; ithin a p:::eferreC ".::em. a patie'lt experienced :w.ore tr?.ar.. or,e ad-,re:::se ever.it •,;it:,in a system organ class, the patient is coc::-,ted once for each preferred ter.:., ai.C. or..ce for the system, organ class.

Table 14.3.2.1 Death Listing Safety Population

| Control<br>Patient/Age/Sex/R | AWL at<br>baseline | "" or" > "" t,1 r.; E1,-< ri; m" f)]] · r1 | Study drug<br>Start Date<br>Day) /End Date<br>(Day) | Last dose<br>(unit) | Date of<br>Geath |
|---|---|---|---|---|---|
| XZXX/39/48/XXX | 0.<br>.,<br>0<br><br><b>III</b><br>5 | | | | t:<br>:<br>:<br>:<br>:<br>:<br>:<br>: |
| Programming Notes: Repeat for each Treatment group Program Name: Listing Source: | ch Treatment group | "11<br>7 7<br>""<br>C | in General State of S | | >,<br>""<br>0<br>""<br>0,<br>"" |

Table 1 .3.2.2.1
SG.\Ena::::; of Labore.to.::-,,- Test Results and Change f:::o:r, Baseline by Visit-3one Marro,..:
Safety Populatior,

| : <u>v</u> Vi"i c- | ccr.t:::ol<br>""XXX | () | Lo·,· CX -01<br>= ;,:xx) | :iigh CX<br><sub>'}</sub> J = x;{x: | -Ol | Ove:::all<br>:-:xx1 | |
|---|---|---|---|---|---|---|---|
| | { %) | | | n | | n | |
| aseli'.1<2 | | | | | | | |
| | кхх | | xxx | x;,:x | | xxx | |
| :mean (s.d.) | ;,o:.x | xx.xx) | xx.x (xx.xx'. | ·:-:.xx | ( xx.;;s:) | xx.;,:z | x:::.xx) |
| median | ½2X . X | | ZX* | | | xx.z;.: | |
| :;:iin | : <x. td="" x<=""><td></td><td>x:, .z</td><td>xx.z</td><td></td><td>xx.xx</td><td></td></x.> | | x:, .z | xx.z | | xx.xx | |
| :nax | XX.X | | XZ. X | .:-:z .x | | V ∆X | |
| ∥ sit> | | | | | | | |
| r: | :-:xx | | ;,:xx | XZZ | | ;.:zx | |
| :71.earr (s.c:.: | ;-::-:.x | x;-:. xx:, | $xx.x (xx.x:\{\cdot,$ | XX.XX | xx. xx', | xx.xx | xx.xx) |
| cnediar:. | ו:. × | | x | ;,:x.z | | :,:x. | |
| ;:n1n | x;,:.>-: | | x:-:.x | xx.;.: | | XX.XX | |
| max | :,:x.x | | XX.X | XX. | | x;s.;,o: | |
| Change £:::o:r, 3aselir,e | | | | | | | |
| rr | xx;.: | | ;,::0:. | xxx | | ;.:XX | |
| mean (s.d.) | :,:z.z | xx.xx) | xx.x (xx.xx) | xx.x:,: | XX,. | <u> </u> | xx.:-::-:) |
| median | ;,:z.x | | xx.x | XX.X | | :-ex.xx | |
| m.1.n | x'x | | xx.:-: | ;-:x.;.: | | xx.x:-: | |
| c2ax | .x | | XX.X | :o:.;z | | XX.XY. | |

### [C6ntinti'e fOr;'-rE!maining post-baseline time poin.tS]

:'iote: For cha::-ge £:::ori :Jaselice cal,::ulatio2s, this tables 0,.1,, preser,ts :::esults fo::: 9atiects with non-::;-.iss:.ng data 2t ;:)aseli:1e a::1ci time po.:nt of interest

Page x of

Listiu.g Source:

Table 14.3.2.2.1
S:Z'etary of LaDoc:atory Test Resc:.lts ar,d Change frorre Baseline by \'isit-3one Mar:cow Safety Pepell at i or,

| dy Visit | :ont | rol<br>xx::;:. | $_{(N} = )$ | CX-01 | High C ;::;:= x n ('!; | | Over. | 3.ll<br>xx;{} |
|---|---|---|---|---|---|---|---|---|
| si c.> | | | | | | | | |
| Auer rods | | | | | | | | |
| ľ.J | ,::,:x | | xxx | | XXX | | :,::0: | |
| Yes | >:x:-: | | XY.X | xx.x'.s' | XXX | :c:.x%) | x;-:;, | xx.:,· |
| :-le | ;{;"'.x | Y.X. | XXX | xx.x% | XXX | ;-cx.x'"\ | :S:X:-:: | xx.x":) |
| Response | | | | | | | | |
| | Y.:•:X | | XXX | | XXX | | x;,:x | |
| Mo::::-phologi:::: corr.plete rerr,issicr, (C?.) | Y.:<:x | XX.Y.0' | XXX | XX.X'c' | XXX | ( ZX. | ·•:xx | xx.x%; |
| Co::!:tplete re:nis2ion without reco-ery o-f | | | | | | | | |
| platelets (CRp;,<br>Complete :::-ecTLission withct:.t ne,,;:::::-ophi2.s | XY.X | XX. | xxx | XX.X | XXX | XX. ∺ <sup>7</sup> c) | | XY.X |
| and/or platelets rc?i) | '{XX | ;,:x. x't' | :{×× | XX.X | XY.Z | X:•: | X>:z | xx.x% |
| ?a::tial emissio:1 {?R} | s:xx | XX. | XZX | );x.x | xx;-: | XX.X, | '.C{X | z:-:. x';- |
| Progress ve dis as (PD) | :<:XX | 7.X. Xi;: | XZX | xx.x | XXX | <b>xx</b> "".!/, | ;:XZ | |
| Stable D sease SD | :,:;:X | ., : 'c | XXX | XX.X | XXX | xx.z% | XXX | xx.;:% |
| Relapse c:crr, C?. C?. /PR | ,::S:X | >:x. x'c | x;:x | XX.X'O | XXX | xx.x?i | ZX:,: | xx.x':,: |
| In.deter;:n !:ate | ,:xx | x :. <b>x</b> :;,• | :-:xx | xx.x\"0) | XXX | xx | | x;:. |
| U:iknown | ,:zx | xx.xo;;; | :s:xx | xx.x%) | XXX | xx.x% | :,:xx | zx.x%" |

[C6nti'nile: £Or remaiii.ihg post-: ba·s·e1"i -ne tim·e- -pointsj\_

;;;ote: lo::: char:ge from, baseline calculations, -chis tables o::-,l--- p:::esents :ces;;;.lts for patients ;::ith non-r::-,issl::lg data at baseline a.r"d tit.me point of interest

?ro-;::aon:-lane: Pate Ger,e::a.tei: ?age x of

7.'5...-: :- s " C""

# Table '4 3.2.2.2

Su.'Ilc;a:r:::-' of Laborato::::-y Tes:: Results and Cl"",ange ::'::::-:r.. Baseline by Vis.::.\_t.-:-ie:;r,atology wi::h CBC Safety ?cpulation

Hematology -;...;-i t.: l CBC: f.err:ogl.obir, ,: u:-ii t)

| dy Visit | :ont:col<br>{N = x;•:x)<br>n (%) | LO\*! C,-v.<br>xxxl<br>r, | $\frac{1g''''}{(1-, = XXX)}$ | Ove::::-all '.l.(= xxx) C, | |
|---|---|---|---|---|---|
| eline | | | | | |
| n | xxx | XXX | XXX | XXX | |
| | XC{.Z XX .: z'. | xx.x XY.XX) | x:,:.x>c (xx.x;:) | | xx.xxj |
| ' <ed.::_ar,< td=""><td>XX.X</td><td>xx</td><td>xx.x</td><td>x:::</td><td></td></ed.::_ar,<> | XX.X | xx | xx.x | x::: | |
| D1:1 | XX.X | XX.X | xx.x | xx.x:-: | |
| r:-,ax | xx.x | XX.X | :=;;= | ;,:;,:: | |
| sit> | | | | | |
| n | XXX | ZXX | xz:-: | ;-:xz | |
| r:;ea.n \s .d. | xx.x ixx.xx | xx.x ( x;-:.xx:· | xx.xx (xx.xx) | ;; ,:. ;-:z | xz.zz) |
| Dedian | XX.X | xx.:-: | XX.X | :,:z.xx | |
| r::in | xx.x | xx.x | Z}:.;: | xx. x;,: | |
| max | XX.X | X | .··,:.x | x:-:.xx | |
| :J.ar:s:;e from :Sase::.ine | | | | | |
| n | /:xx | | XXX | XXX | |
| r:-,ean (s.d.·· | xx.x ( xx.xx) | <b>xx.x</b> x:-:.x:-:} | XX. ;,:;:. ZX) | :-:z.zx | xz.xx) |
| :-edia'''.' | XX.X | :,:x.x | <i>x</i> ∴ x | :,;:z.xx | |
| XITI | xx.x | XX. | };; z | :,;:;,:::-:z | |
| :::ia;: | x;:.x | XX.X | :{. ): | xx.;,o: | |

t-t::ont:LnUe £or remaining pos t --:baSeline time 'poihtSJ

Note: Fe:::- cha;:-;ge: E::corr: baseline calculation.s, this ::ables only presents result:s :::ol:" patier,ts wi::.r". no,,-r:--.issin:; data at baseline and tirr,e point: of inter:-est rOgr -rimi,hg, Notes,:

Repe-at- fOr each c'oritinuous fab pai:affieter

Program Name: Date Generated: Page x of Y

List.ir::g So,.\_;\_rce:

Repeat fo:c t.:"?.e followc..ng displays:

Table 14.3.2.2.3 su., Ilriery of ::.aboratory Test Results and Change fron, Baseli:1e by Visit-Coagulation Safety Population

Table 14.3.2.2. Signal y of Laboratory Tes:: Results and Change from Ease:cine by Visit.-Se:ru!ri. C'."",emistry Safety ?opulatior:

Table 14.3.2.2.5
Shift. ?able of :,anoYa o::::: ?est Results icm.;.nts:, b:, :-:::\_CTC.".E g:::::ade: He"latology ,,,ith CBC Safety ?opulatio:-:

| HeBatology with CBC: He:r,oglobir, | Control {N = xxx} \';'erst Occu::-rence | LOK CX-01<br>= xxz·<br>Worst Occc,:::re:-:,::;( | High CX-0'<br>(N = :-:xx)<br>:·Jo:rst C·cc,1:::-rence |
|---|---|---|---|
| | 2 3 ' | ?Ј | N 3 • |
| Change f.::::0c:-, ,,:erst grace to last grade: | | | |
| 0 | xz}: xxx xxx xxx xxx | XX}: XXX XXX ZXY XXZ | xx:{ x; <z :="" :,:;,:x="" x="" xxx="">:</z> |
| -1 | XXZxxx xxx x;u: xzx | xxz xzz XXX :,;x:,: :-:z;,; | XXX XXX Z:{x xx;{ xxx |
| | xx_;.:xxx xxx xxx xxx | :-;:;,:_;:: xxx | XXX XXX };:,:x ;{:-::{ :,;xx |
| -3 | zxx :co: XXX xxx XXX | x: x xx:,; :-:xx ;,::, x xxx | xxx xxx x: <x xx="" xxx="">:</x> |
| Only o:1e :c.easure,r,er,t e::c | XXX x:,;;z zxx x}:x xzx | :zxx :-:x:s zx;,: z:,:;,: xxz | XX:< XX:< X:C*: XXX XXZ |
| | xxx :n::z xxz zzx xxx | X>:x xxx xxx x}::, :,:x:{ | ZXX XXZ '.{xx xxx xxx |
| +2 | }D:X ;,;XX XXX XXX XXX | :-:ZX XX:: XXX :•:XX :,;;;X | XXX ;:XX XXX :-:XX X:<:i: |
| +3 | XX): ZXX XXX XXX :SO:X | xxx xxx xxx }:xz _;.:z;: | ',:XX %X:% X;-::X :-::XX X:-:X |
| .Only or,e!1'.easure,:tent etc. | ·-:XX ZXX XXX XXX XXZ | x:::z xzx xxz xzx }:x | ;;; XX>; XXX XX}; XXX |

Note: This table p:::ese:1:::s "o:::st to last va:Cc;e fro::-t A?:.;ia;es, by definitior, Ai'::is desig:ied to :::ecc:::::ds 1nto;;;-ard clinica::. eve:-its, so im:x::o,;e::ne:1ts are usu:ally not reco:::ded tr'£ database, this limi-cation of data is ic;rportar.t for t:'..e i::terp::etatior, of this ::able.

P,r; /gr'.a,ffimin-g Note-s

Repei:it "for eaCh lab -parameter

Program Ncne: Date Ger,era::ed:

?age of

Listing Source:

Repeat fo:c the foJ.. lowi:1g displays:

Table 14.3., 2,6 Shift Tab:Ce of Labora-::o::-y Tes:: Resc.:.2.ts (co;;;\_nts) by NC: C:TCA-2: grade: Coaq,\_;\_latic:r, Safety ?opulation

Table 11.3., .2.7 Shif:: 'table of Lr.borator,- Tes:: 'esec:.lts (counts) by NCI\_C:TCA2: grade: Ser T Cherr,istry Safety Pop;,,lation

Table '4.3.2.2.8 Shif-:: Table of ::.,aborat.ory Tes-:: Resc:lt.s \%) by NC: CTCA -;rrade: Hema-:::olcgy ,:it:/ CBC Safe-:::y ?opulatior,

| Eematoiogy with CBC.Hemoglobin | Cor.trol<br>,;i,.;, = xx:-::<br>Korst <u>GC(T: Pre</u> | I.o·,,· 0:-01<br>(N = xxx)<br>C\o::st_Occu::::RT:CR | E.igh CX-Gl '}) "" xxxj ::-Jors-::: Occ of r -:::::::: e |
|---|---|---|---|
| | l'J 3 4 | N 2 3 4 | 2 3 4 |
| Cha:1:;e frorr, wo.:::st g.:::acie to lase: grade: | | | |
| C | ;-:xx :-:zx xxx zxx xx;,.: | xxx xxx xxx xxx xxx | XX',::O:X XX:;;: XXX XXX |
| | x;-;x xxz xxx xxx ;::-:z | XXX ;-;;,:;.,: :<'.XX XXX XXX | ·,;x;-: xx;,; ;.,;xx x;.:x xxx |
| | xx:-::-::-:;< xx;-· xxx ;,:;-:x | XXY ;O:X X:-:X XXX XXX | $x;; xx:{ \times \times = x; -: }(\times \times$ |
| -3 | xxx xxx xx:< xxx :•:xx | xx;{ xxx xzx xxx zxx | XZ}; ;-:z:-: XZX xxx xxx |
| cn.:y one :u.easureZ<1er,::: ec:c. | xxx }:xx xxz xxx xxx | xxx xxx xxx x;o: xxx | ZXX :<::-S::{ xxx |
| | xxx x:{x xxx xx;-: xzx | xxx xx;,: ;-o:x ;,:;,:x xxx | :-:xx xx;: xxz xxx xxz |
| | ::-0:X XXX | xxx :{xx xxx xxx xxx | zz;.; Xz:,; XXX XXX XX:{ |
| :.3 | ;:;{x ;;;:;, X:-:X X:-::,: | xx:: xx:: xxx xxx :<:xx | ;o::-; :-:ZX XX;: XXX XXX |
| . Oiiy one :c.easurezr.en.t etc. | XXX XXZ XXX ;,.:XX | xxx ;-:x:-: :-::-:z ;:xx ;,:xx | :-:xx xxx xxx x:,:z |

: ote: ihis taCle presents worst to last valc,e fro;r, A.S pages, by definitior AE is designed to record ,\_;\_::t0h'ard cl.irLi.cal ever.-'.:s, so irr,proveu,ents are use.ally not recor"cied ir:: the database, t'.", is limitation of data is irnportar, t for '.:he i::terpreta""...io:: of c.r'.is tabl.e. ?:to(Jramming-:ii6:tes::

REPE: "a'.t fo\_r. -iat:h .lab\_ - pa.tB.rneter,\_ % fo.i:'- the denominato'r \_is\_bi!sed on the - t6tal - wi"t:bin- .each: - rBC\_tarigle - cell. :'..v-: ca., t-:a1c.8. :Jate Generated:

Listing Source:

?ag-e x cf y

?..epeat fo:::: the followin; displays:

Table "L 3. Shift Table of Laborato::::,, Test Res'.llts t:-y 1:CCI CTCAE grade: Coagulation Safety PopcJ.la-:::ior.

ab::.e .3.2.2.10 Shift Table of Laborato::::i Test Resu.: "'.:.s by UCI CTCP..E g::::ade: SerGTc Cf',emistyy Sa:::"ety PopcJ.l.abo::

 $\label{eq:table_ros_3.2.2.1l} Table \ cf \ Laboratory \ R < csc:lts \ (co'..lnts) \ He.satology \ with \ C3C:Her:,oglobi::-: \\ Safet'.f\cdot \ Popu.lc.tion$ 

?age ::-: of

| Hematology with CBC | Control<br>(N = XXX)<br>Baseline<br>C-N Baseline | | | | Low CX-01<br>(N = xxx)<br>Baseline | | | | High CX-01 (N = xxx) Baseline | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -IN | Ε. | _0_0 | | | | Aot | | \ <b>J</b> | E | Tot |
| <visit></visit> | | | | | | | | | | | | |
| Lo;,· (L; | xx;-:: | XXX | x:,:x | xzx | XXX | xx;,: | x ::<: | XXX | XXX | :,-:x;-: | xxz | ;,;:,:x |
| Nore.al ( :;,) | XXX | XXX | XXX | XXX | XXZ | :-co-: | x;;z | ;-:x:-:: | x;-:x | L:xz | xx:-:: | z:-::x |
| Eigh (1'1) | xxx | XXX | XXX | XXX | x;:x | ;-:: <b>x</b> ;: | | | XXX | ;,::xx | XXX | x:-::x |
| Total ::Tot) | :{XX | xxx | | xxx | XXX | XXX | ;:;SZ | :-::,-;;: | :,:x;-: | | ZXX | XXX |
| <visit></visit> | | | | | | | | | | | | |
| i,C; (l. i | ZXX | XXX | :n:x | :s:xx | XXX | ;,:x:,: | | xxx | xxx | ZX;-:: | ;-:;,;x | XXX |
| <u>\:</u> 1 | ZXZ | zz:X | xxx | XXX | xzx | ;-::zx | :,:;-::x | : :-:x | xxx | ;-::xx | xxx | XXX |
| Eigh {:-i) | zx:-:: | XXX | XXX | xxx | xxx | :-:: <b>x</b> x | XXX | xx:-: | x'.x | XZX | XXX | XXX |
| Total ,:rot) | XXX | XXX | XXX | xxx | xzx | :-::xz | ZXX | :-::xx | xxx | XXX | XXX | XXX |

< continue for 'an: \risi ts,>

:'late: 'Phis ;:able or:ly 9Yese:1ts :results for pat.ien.ts with !"lon-rr;issing da;:a a:: base2.ine a:l'.::, the tirr:e poir::t o:!: ir::terest. FrOgr-a,.--mr,ing - Not.es:

:R.epeat:):cr. ea'Ch l:ab·-para-n':lt:er

?rog:::artc Na!T!e: iJate Ger::era.ted:

Listi::-:.g Soc.:rce:

Repeat for the following ciisp.1.ays:

Table "4.3.2.2.12 Shi:'.:t :a;:)le cf Lcaborato:::y ?,esc.lts (counts:,: Co2.gu.latio:c:A::-;\_ti-Factor Xa Safet" ?opulati.on

7ab.l.e 14.3.. 2 11 Shift '.ra:Ole of Labo::::ato:::y Results {counts} · Se:::-""-" C:lemistc,-:Albu,,-r,in Safety Pop:;;\_laticn

Table 14.3.2.2.14
Shi::'t Table of Laborat:cry Resc2lts {%\: H.e:ri.atclcgy \cdot,;:'\_\_th 23C:rte::-,og2.o:Ci,.
Safety Population

| Hematology with CBC | | Low CX-01<br>(N "" XXX)<br>Baseline | | | | High CX-01<br>(N"" XXX}<br>Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | e:: | | Tot | L | N | Н | Tot | | | 5: | Tot |
| <visit></visit> | | | | | | | | | | | | |
| Lo:,: | X:G: | :,:x | xxx | zx;,: | x:-::x | xxx | XXX | xz;: | :G:x | XZ:-;: | XXZ | XXX |
| Nor-ma (Nl | *************************************** | XXX | XZX | XXX | XX | XXX | XXZ | XZX | -,::-::;-;: | Z/:X | :-'CXX | XXX |
| Hic;r'. rt) | xxx | XXX | XXX | XXZ | XXX | XXX | XXX | XXX | z:-;:;-; | ;,;x;-:: | ZXX | XXX |
| Total (Tot) | ZXX | X:-:::-: | /:xx | ;,:x:-: | XXX | ;,:xx | xx:-:: | XXX | | :,::,:z | XXX | x: x |
| <visit></visit> | | | | | | | | | | | | |
| Lo:,· \LJ | XXX | XXZ | XZ/: | xxx | XXX | XXX | XXX | ZXX | x:, | :-:xx | z:-;:x | :-:: <b>xx</b> |
| No::-:real (N) | x;o; | xxx | | XZX | XXX | ZXX | XXX | XXX | ;.::,n· | | | XXX |
| Higr', (:-i;, | xxx | x:o: | xxx | xxx | XXX | XXX | XZX | xx:-:: | ;s;:, Z | XXX | :s:xx | XXX |
| To-:::al '.Tot) | ;.: ·'.X | XXX | XZZ | XX/". | xx:-;: | XXX | XXZ | xx:-;: | XXZ | XZX | XXX | XXX |

<Cont±nue ·,£6.b ··all - Vis'its>

;;;oc:e: This table only preser;ts res,ilts ::or patients ;,·it:'. non-:;;:issing data at baseline a:-,d t:-1.e tirr,e poi::-,:: of i;;te;:est. Progra\_mii'ng-1 otes:c.

R€Pea,t :.Jo,r eaC11: lci.b parameter:,

for the denoffiin ater is based on tliELtOtaJ.: 1/4"ithin each -sq,Ji;;;i'.e cell.

Program !: 0ame:

Dat.e Generated:

?age :-:: of Y

Listing Source:

?.epeat for the follov,ing ci.isplays:

'7ab.'...e 'L.3.2.2.15 Shift <;: able of Labora.to:::y S.esc:... ts

Coag\....lation:J:..nti-Factor Xa Safety Populatior.

?able 1 . 3 . . 2 . 16 Shift Table of Lal::oratory ?..es;;lts (": · Seruc.I Che:m.istry:Albc1<--::l:i.D sa:::et;/ Pop:.i.latio,,
Figure 14.3.2.2.LI PT/IN? ove;:;:ir::-,e Safety ?opc:la;:ion



Pc:ogc:am Name: Listir:g Source:

Date GenerateC:

Page z of

epea-::fol'.:the followi::.g displays:

| Figure 14.3.2.2.18 | APT'' 0'7@r ti:me Safe-::y POF-Jlation |
|--------------------|----------------------------------------|
|--------------------|----------------------------------------|

Summary of dest at Screening and Vital Signs at Screening and Start of Footoliogic; F.Y.'s Safety Population

| | | ,,<br>00<br>PO<br>08 | G | o i | ,⊸<br>%<br>%<br>%<br>,5 |
|---|---|---|---|---|---|
| T | | ¥ II | <br>[j | [;] | :<br>: K |
| *** ********************************* | | r: | r. | <b>-•</b> cf,≎ | |
| | 0. i.?,<br>0. w<br>0. w<br>0. iii<br>f.1 0. 4-1 | | | | |
| | (a) | | | | |
| 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 | 1: d d d d d d d d d d d d d d d d d d d | | | | |
| O TO THE STATE OF | ~!!!<br><br><br>!! | | | | |
| -0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 | | | | | |
| See of the see of the | | 7999 | XX | :<<br>X<br>:,: | 2003 |
| Signate of the part of the par | | ;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;; | ××.× | x. | XX.XX |
| XX | median | | ××.× | : <b>&lt;</b> : | 2x.xx |
| ANN NAME OF THE PROPERTY OF TH | cin | | XX.X | | ZX.XX |
| MANN NEW YORK NEW YOR | | X<br>X | > >> | | 22.32. |
| C C C C C C C C C C C C C C C C C C C | 0<br>!!! | | | | |
| X. | , | XX | MMM | | '.<<br>X> |
| | p.e :; <b>==</b> ! | | x x x | X.<br>:< | R |
| X X X X X X X X X X X X X X X X X X X | median | 22.22 | XX:X | :<<br>:;:<br>:< | R<br>KX |
| X | min | M. X. | XX.X | :<<br>X<br>X | • |
| Y | | 20.00 | 2.33 | :<::::::::::::::::::::::::::::::::::::: | x |
| X X X X X X X X X X X X X X X X X X X | | | | | |
| X X X X X X X X X X X X X X X X X X X | | ; X<br>X | XXX | Y.<br>X | XXX |
| X X X X X X X X X X X X X X X X X X X | | ::<: | 83.3 | tje | 22.23 |
| <del>X</del> X | r.:: =================================== | X :::: | x.xx | X<br>:V'. | ZX.XZ |
| ÿ | | | XX.X | Ÿ | XX.XX |
| | | | X . X X | ::<br>X | XX.XX |

H O

c = % Generated

u f.d H o MXBEELINS

| | d Carried Street | Trocarie - | . 1 b, r? | r:<br>;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;; | HE'A 1 :: 10 H → TP MC (1 H) A (10) MC (10 M) (1 A (1) A (1 |
|---|---|---|---|---|---|
| | | - R - r. | | c-1<br>.:X: :<<br>u >:<br>gll : ""<br>:1; ;;; | """""""""""""""""""""""""""""""""""""" |
| SBP (mmHg Screening) | | | - | | , |
| , t: | | >: | XXX | XXX | :<; |
| 0<br><11<br>!:i i | | >( | XX,X | xx.xx | XX. |
| r:<br>"S<br>:i fi | | ,'s<br>:< ; | XX, X | ×.×. | N;;; |
| r,<br>d | | | XX.X | XX.X | ××× |
| N. P. C. | | ,, | X X X | * ** | 22 |
| DBP (AmAg) (Screening | | | | | |
| r. | | N.KO. | XXX | X | KAS |
| mean (s.d.) | | XX.X | XXXX | :•:<br>>:<br><b>i</b> | X :: |
| median | | ×. ×. | 22.22 | R | |
| nin | | XX.X | 22.2 | R | × × × × |
| NEG | | 20.00 | 22.22 | | |

0 :<

Date Generated

! ITI <UG | n . .-I | O m | y . -I | n, ,..i

Table 14.3.3.1 Su.Tu--nary of 2:COG S-:::atus at Sc.:::-eening and Vital Signs at Scree?:J.ing ar,d Start 0::. Cc::1solidation Cyc.:.e Safety ?opulati::Jn

| | :cr:trcl<br>= xxx) | | :,o'.'-' D'<br>{!'i = ?:zx | | High CX- $(N = XXX)$ $E(;)$ | 01 | Over2ll<br>CJ xx<br>r. :S:, | |
|---|---|---|---|---|---|---|---|---|
| Weight i/;g} (Ccnsolidatio:-:: cycle} | | | ,, | | E.(,) | | 1. 101, | |
| c | XXX | | xxx | | XXX | | xxx | |
| :,,ean (s.C) | | :X.XZ} | ·-:x. | xx.xx) | XX.:-:X | xz.:,;x) | xx.· | ·,···,-·· |
| median | xx.x | , | xx.x | , | xx.x | ,, , | xx.xx | ,,, |
| 17,ln | }:X.X | | ""(,:,: | | xx. | | XX.XX | |
| c:iax | x::-:.x | | ;=: | | xx.:,: | | ;-:x.x:,:: | |
| Height ter.) Co:csolida-:::ion cycle) | | | , | | ,. | | ,, | |
| C | :, z:- | | | | xxx | | xxx | |
| ,near, (s.d. | xx.}: z | y .xx1 | }'.Z, ∨ | xx.xz} | :-:-,; 2X | xx.xx) | xx.xx | ·.•;,:.:c-::; |
| .:c:edian | XX. | | XX.Z | | XY | | xx.:-:x | |
| '.c'.in | XX.Z | | x:•:. x | | :-:x.x | | xx.xx | |
| :max | xx.;,• | | xx.;-: | | xx.:,:: | | xx.xx | |
| lea.:::::: ?2.te (beats/min) Cor:solidation | | | | | | | | |
| ycle} | X:::X | | x::-:x | | XXX | | xxx | |
| | xx ::- | -:x. xx! | :-::-:.;-1 | xx.:=::x | XX.XX | x;-: xx) | ZX.ZX | X:-::, |
| ::r:.ean (s.d. | XX. | | XX.'>' | | :o:.x | | :x.xx | |
| d: an_ | ;,::,:, <b>x</b> | | xx. | | ZX.X | | xx.x: | |
| Tc,in | XX. | | XZ. | | xx.x | | ··-,· vv | |
| IT;2X | | | | | | | | |
| B? (.:1,;c: g) Consolidation cycle) | | | | | | | | |
| | :-:XX | | x:-:x | | XXX | | XXX | |
| ::-::cear. ,:s.d.· | | ;-:. XX) | XX. | xx.xx} | XX.ZX | ( xx.xx) | xx.xx | x.xx', |
| s.edia-:1 | XZ Z | | XX,'>' | | XX.X | | XX.XX | |
| :n.ir, | XYX | | X;,Z. X | | XX.X | | XX.XX | |
| :2.ax | XX.X | | X:-::. | | XX.: | | XX.XX | |
| OBI? (rur:Hg) Co:1solidation cycle) | | | | | | | | |
| n | XZX | , | XXX | | XXX | | XXX | , |
| :nean (s.d. | | x.xx) | XX.X | xx.x:-:} | | x ( xx.xx) | X}:.xx | ( xx.xx:, |
| :median | xz. :{ | | xx.x | | XX.X | | XX.XX | |
| min | XX.X | | XZ. | | xx.x | | xx.xx | |
| max | :x:x.x | | xx.x | | XX.X | | xx.x:,:: | |

?rograrc, Name: :.,is::ing Sou.::-ce: Page x of y Date Generac:ed:

Table 14. 3. 3 2 Shi::'t of ECG Resollts Safet:y- Population

| | ::antral<br>{N"" XXX)<br>n (%) | Low CX-01<br>(N"" xxx)<br>n (%) | High CX-01<br>(N = xxx)<br>n (%) | Overall<br>(N"" xxx)<br>n {%) |
|---|---|---|---|---|
| <visit></visit> | | | | |
| :'rorr. r-,ot clinically signi:'icant<br>abno:r;r,al | X} | XXX | X:0: | xxx |
| res,lt at baseline to abrormal and clicically sig:lific2r.t:-es'.llt | xx>! xx.x%) | x:c-: xx.x"' | X:,:X XX.:{'''' | xzx ;-:z.;{\;) |
| ?rorr, abnonr:.al and C:inicai::.y<br>signif ca::,t<br>res'J t at baseline c;o nc-t clinic2lly | | | | |
| sign ficar:t abnormal :resc.1.l':: | xx xx.x%;, | x:s:x <b>xx.x%</b> ) | x;-:x = "0, | xzz x:s.Y''' |
| <u>t]· h e<sup>rot</sup>d</u> | xxx <b>xx.x%)</b> | XXX <b>XX.X·3</b> : | xxx x':c\ | XXX XX.X'2 |

. Rej;:ieat for all ,visits where ECG performed >

Note: N: ?Jormal; ANCS: A.Dno:rrr,al, Not C:linica.!..., Significant; f.CS: P-..D:,o:-::mal, Clir,ically Signi:':icant Prograo:1:'1ame:

Listing Source:

?age x of

## Lisc:.i:1g 16.2.1 Subjects Screened

T:reatr.:.ent g:roup: Treatment

| Site | ?atier.t/ Race<br>Sex/A'.ie | Date of<br>Info:rrr.ed<br>consent | Scree:-: Fai.'c.:re |
|---|---|---|---|
| XX | xxx/M/ 4 5 XXX | D':-ir:Mv\·vv | Reason Reasor: 2 Reason |
| XX | xxx/F/35 xxx | DD:-JMMYYYY | |
| .xx | xxx/M/25 xxx | DDi'IMM'.:"YYY | |

P·r·o9 -ra.'r.ming Nb:te\_S:

Repeat: "for all T-reaL--nent groups: \_Sort by Treat\_ment ·gr:o\_up, ·sfte·. and\_pat"ient
Pro-;:ram Name:
Listing Sou:rce:

Date Ge:le:ra pri

?age x of

### Lis::ing 16.2.2 S:.ibject Disposi tic:-.

Treat::ne1;.t group: Treat:;;e;1t

| Site | ?atieEt/<br>Se:,:/Ale | ?.ace | Co:::.pleted<br>St;_;_dy | ?rimary Reason ::or<br>'iiiti:drawal | :ate ofWithdrawal<br>Day)'.a] | ate of ast Dose of<br>tudy :'reatmerIt gro-c1p<br>Dal) {a] |
|---|---|---|---|---|---|---|
| XX<br>X: | xxx/M/ 4<br>xxx/F/3<br>}:>:X/[•1/2 | xx2'<br>xxx<br>xxx | '-0<br>:-;0<br>Yes | Ree.so.,<br>Ree.son 2<br>Reasor: | C::·Dm,11-:'.YYYY {XX<br><u>O</u> , :[*·i.*'t: | DmJMMYYYY (xx<br>DDMMM'IYT:'. (zx<br>DDt-!M.MYYY:' (xx |

[a] ?,elative to the da·, of r2.ndomizatio:1 P:r\_og·ra."r,ming:.Notes

R'ep-eat for. ,all 'f:ceati:ne·nt groups · Sort by T\_i:Ji:ci£itte11t·gr\_oup, site. ind  $Padent = \frac{\text{"-o-r--}}{\text{Lis}} \cdot \frac{\text{L-n--}}{\text{Lis}}$ :
Lis ;::ing Source:

?age x of y

### Listing 1E.2.3 Sc1bject :reatmer;tAllocation

| Site | ?atient/Sex/.n.qe | Race | Random:zed ?reatrr-ar,t Grcclp | Date cf Rand:::mization |
|---|---|---|---|---|
| XX | xxz/11/45 | xx;; | XZ;,-: | DJ11:":::'YY |

P\_ic,g'ra.-n.7"<\_iil\$\_-\_:N t---\_:
-Re,Peat for all tr-eat.c--nent. roups. Sort'b:':i' site- a'nCl patient
Progract, Name:
Listing Source:

Sate Ge::erated:

:?age x of y

### Listir,g 16.2.4 ?ro":.::ocol Deviat:ions

| Sit:e | ?atie:1t/Sex/Age | Race | P.ny<br>Protocol<br>Deviations? | Date | ;:>ro;:ocol Deviatio::1<br>Catego:::-y | Details of ?:::-ctocol<br>Deviatio:1s |
|---|---|---|---|---|---|---|
| xe: | :;:/M/4S | xzx | Yes | J:)>.'eMcJ:VVVY | z;:xxxz;s:xxxzxxzx; | x:-:i{XXX:•:xxxxxxxxxx :xx |

:""cl da '-"":""s" lock. ?ac:ier,t:s rreay ha-ve may have more than or,e Deviatic-:-; ]..e2.ding to No-::.e; Jevia;:ions were ider,tified a,:d categorized prior e:-<:clusio:1 fro:c, Prog:r:a,,"nTili\_ri.g Ncit es:

Repea:t..foi all .Treatment··tjio.u:ps·. -sort by ,T:rea:tm .nt:.group, site; and patient PYogra;r, l:Jame: Date Ger:erat:ed:

Page x of Listing Sou.rce:

| | | >,<br>•••<br>0 |
|---|---|---|
| <b>11</b> Н | | |
| H 상기 | | Control of the Contro |
| ;•;<br>11 | | |
| H<br>Ook | x x x x x x x x x x x x x x x x x x x | 16-1<br>5-1<br> |
| ו בול לי פר;<br>יי וו יי עי ת עית עיק עיק ר. אינ שית עיק ר. אינ עיק עיק ר. | ,#,n<br>< | Programming Westers<br>/ Soft by eath and patient<br>Program Name: |
| ,;;<br>{/) | X X | Profits |

## Listing 16.2.6 Excl;\_.;\_sior. Criteria

| Site | ?ac:ie:1t/Sex/AB:e | ?ace El | E2 | E3 | :'4 | E5 | 6 | s7 | £8 | E9 | ElG | ::C:ll | cl2 | e,13 | E14 | E15 | El6 | El7 :'18 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XY. | ;.:x: h-:/45<br>:xx//35 | XXX | | | Yes | | Yes | | | | | | | | | | | |

Progratmning NOte's:
Sort- by";\_si'te and \_patii:=-nt
Fc-,ha\_c\_,io".e.
Listing So'J.rce:

Date GenerateC.:

?age x of y

#### Listing 16.2.7 Study Pop,; lation

Treatment a ...-oun: Treattrie t

| IIEati | пенс <u>ч</u> ои | D. Treum. | 5.,t | | | |
|---|---|---|---|---|---|---|
| Site | Pc.tie:it/<br>Sex/A2:e | Race | Completed Study | :T? | 1?? | So.fet· |
| xx | x;;x/:-1/45 | XXX | Yes | •-'es | :es | Yes |

?age x of y

Progra; :n Name:
Listing Sci..;rce:
P:r(igrarhthing-: Notes:,

Repeat fOr all Treatment grOup\_s Sort by Trea:tmBn:t,-g'i-6Up;, s'ite -'aild :patient
Program i'arr.:e:
Date Geuerated:

.22.ge x of Y Listing Sour:ce:

### Listing 16.2.8 Demographics and 3aseline Characteris::ics

Treat::',ent grc·clp: Treat:nent;

| 11000. | / one gro orp: | , | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Site | ?atient/Sex/.Age | ?ace | 3MI<br>Cetegory | 3'.fi | Wei.gr,,_<br>:g) | SSP<br>/:JBP | Hea:.::t<br>Rate | ,.,:,-f'.nicity | Time<br>since F>2.L | pJ.;l., | ;.;-:-ese """"<br>of 2:-,y | ECOG<br>status | B.aseli,,r-> peri?l":era::. | 3aseline<br>3one |
| | | | | | <u>!c•'c'''</u><br>(CT:',;; | | {beats,?er rr,:-:.ni | | <u>c : co"'::"</u><br>("::'ear) | | r elega:.t | | blas::s •;Yes/r.;c' | Marro:,·<br>blasts |
| xx | :-:xx/M./4S | x:-:x | xxx | x;-:x | :-: <b>x</b> /:-:;.; | :-exh:;s: | x>: | xxx | xxx | :Je<br>r,ovo | Yes | tettegjet | xxx | xx:-: |

1?ro9"r&lli"ning \_rfo't;,\_es·

Re'peat f6r a:Ll' T.reatmen·t ·groups. Sort by Trecatm':!i:tt: groUp, site am:l.patient
Nar'.'£:

Date Genera"::ed:

Prograic, Nar'.'£: Lis::ing Source:

ege of

### List:ing 16.2.9 '."iedical History

?reatment group: Treat,'Tie,-:t

| Site | Pac:ient/Sex/."'.fe | R.a.ce | Systerr: Orga;:-i Code (SOC)/<br>?:::-eferred ·Terc'7![a] | Verbati:r, | Date cf<br>Resc:. u:cicn |
|---|---|---|---|---|---|
| xx | xz:,:i'i:-i/45 | x:-:x | z:xxxxxxxxxx;,:xx::xx/<br>xx:,:x:,:xxxxxxxxxxxxx;, | XXXXXXXX;,:XXXZ:X:-:: | JDtfr:t, YY':"Y. |
| | | | zxxxxxx>:xxxxx:s:xx/<br>xxxxxxxxxxxxx,-:xxxxx;,: | :-:xxxxxxxxxxxxxx | , E <sub>CPP 2</sub> -C. |
| xx | x:-:x | xx:,: | tior:e | | |

<sup>[</sup>a} HedDRA Dictionary (Versie,, xz.x) ,-;as used :'.:or coding. [b] Relati7e to t:'"le da::,- ci: rar.dcrc,ization '.i?'i.c/gral'l'.niiri'9. Note'.sf

Lis;:ing Source:

?age z of

 $p\_e['eat: for.:a11 \dots -T.ceat: ffier-, t \ groups.:SO,.rt; \ by \ Treatm:ent-:-.9'.i'6\_1ipi. \ i;:'ite.,: \bullet \ pa\cdot t \ i \in n\_t., \ SOC \ and \ preferred \ te-tm. \\ Program::-122,e: Date Generated:$ 

| Treatment group Treatment 1 | | | | | |
|---|---|---|---|---|---|
| n:<br>m:<br>pat/sex/Aga | 0,:1, u 0,:1, u 0,:1, u 0,:1, u 0,:1, u 0,:1, u 1,:1, u 1,: | Dose/Unit/<br>Fraquency/<br>Pouts | Lndication | Corresponding<br>term for<br>concomitant<br>disease or<br>adverse event | $\begin{array}{c} \begin{array}{c} \\ \\ \\ \end{array} \end{array} \end{array} \\ \begin{array}{c} \begin{array}{c} \\ \\ \end{array} \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \\ \end{array} \\ \begin{array}{c} \\ \\ \end{array} \\ \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \\ \end{array} \\ \begin{array}{c} \\ \end{array} \\ \\ \end{array} \\ \begin{array}{c} \\ \\ \\ \end{array} \\ \\ \end{array} \\ \\ \end{array} \\ \begin{array}{c} \\ \\ \end{array} \\ \\ \\ \end{array} \\ \\ \end{array} \\ \begin{array}{c} \\\\ \\ \\ \end{array} \\ \\ \end{array} \\ \\ \\ \\ \end{array} \\ \\ \\ \end{array} \\ \begin{array}{c} \\\\ \\ \end{array} \\ \\ \\ \\ \end{array} \\ \\ \\ \\ \\ \end{array} \\ \\ \\ \\ \\$ |
| XXXX/XX/45 | ARRENDENE<br>RRCCMENDENEND:<br>(PRIMARCHEME | ш<br>Р<br>Г.<br>Б.<br>Б.<br>Э. Э., ≤<br>Э. Э. | | | DD:QCXTXYX<br>(XX)<br>(XX)<br>(XX)<br>DD:QCXYYYY<br>(XX)<br>H4:XX / XX |
| Max/2/35 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | , m<br>d<br>, f, h<br>.>∴ X :<br>× × × | Prestment or<br>Adverse Sweet | | Development of the contract of |

'cl III P aj U II ;: II

> g! \$1 f: ::) 8 UJ fd ||T 1-d| ||m f1,,\_\_,

ö⁻¹

#### Listing 16.2.ll Concorr,itant ('Jed.ication

#### Treatmer.t <;\_!?U\_F: *Treatxenr*:

| Site | ?a'.::ie7it/Sex/Age Rc.ce | T::-ie.:-apeutic Class Cher::ical Subgroup c:2:1;;,ri C Term '.a] | ose/Dr:i:./<br>.:ut ,.cy/ | I,1dicatio:1 | Co:rresponding<br>ter:n fo:e<br>cor,co:nitant<br>disease or<br>a::5.s;erse e-,,en::: | Se;.;rt Date 'day_ AIT.8 Sto9 Date (day/[bJ '.Cime/ DuratioH (da_;[S) |
|---|---|---|---|---|---|---|
| xx | xxx/M/45 | XXXXXXXX:-;;X<br>XXXXXXXXXXXXX<br>1XXX:-;XXXXXXXX:;1 | xx/ur,i ts/<br>xx/<br>xx | ANL | | DD:+11-11-11-11-11-11-11-11-11-11-11-11-11- |
| | | XX:-;:XXXXXXX XXY.X):;:zXXXXXXX (xxxxxxxxxxxxx) [cj | xx/uni:::s/<br>xx/<br>xx | ·J:reat:r,ent o:::<br>P.d,,-erse Sver:t | X:-;;;-: | DDI/,I-IMYY-'!.Y<br>(xx) /<br>001"11-:MYYVY<br>(xx) /x>: |
| xx | xxx/F/3S | No:e | | | | |

?rogram r:ame: Date Generated: Page x cf Y
Listing S01::rce:

#### Listir:g 1E.2.12 ?ost Medicaticr,

#### Treat.rr,er:t group: Treatment

| Si-ce | ?atier,t/Sex/Age | Race | The::apeutic Class C:',esica:C S1.1bgrcup G'''.''''' r -""" [:o. | Dcse/Dr,it/<br>Frequer,cy /<br>?o;.1te | :n::.e.eion | Corresport:ditig term:-forO;_CO* c2: dise2se o:-adv-e::-se event | Sta.rt Date (day) Ti::r,e <u>Sc.o:</u> <i>Uac</i> ;; :::iay; ID 'T"irr.e/ =:uration (d2}_'S) |
|---|---|---|---|---|---|---|---|
| x:x: | x:-:x/ U 45 | xxx | xxxxxxx:c-:x<br>xxxxxx:,:xxxxxx<br>'.xxxxxzxxxx:-:x} | xx;':,ni ts/<br>xx/<br>x;,: | .",,ML | | C•"'·C"", '.XZ', c.;;;-l'-11" Drn;;1;'!YY;v |
| | | | xxxxxxxxxx<br>xxxxxxxxxxxxxxxxxxxxxxxxxxx | xx/ur:its/<br>zx/<br>xx | Treatment of<br>Adverse Event | х | E:::1'.M /xx O:bi+.l' i \;-::-:)/ De:':1." i -:<:)/xz |
| XX | xxx/E'/32- | | •lone | | | | |

Listi:ig Source:

Fage x of

a WEO;)rug Dic-::ior,a:cy (Versior. xx)·,,as used for codir.g.
b ?.elative to t:'le day o-f .::::-ando,nization r
grt,u\t.t.i\_ni;(\_Notes:

·.Repeat fer all Ti€:citme\_nt groups. Sort by Tr.eatmE:n:t ."gr 6 up ₁s\_ite, patient, ·.s·tai:f date:'<Otnd.d.r:u9, clas·s:,
Progra:n Name:

Date Ger:cerater:

## -isi::ing 16. 2. 3 Stud:i-' Drug Gsage a:1G. 2:zposu:::-e

1reat:rr,ent g:::-oc1p: Treat;£1en+-

| Site | Patient<br>/Sex/Age | eye.le | Initial ez:-Cl | Id.arc:.biciD<br>usage rate | Cyta::::abine<br>usage<br>rate | CXGl<br>;_sage<br>ra::e | ,,,,,atsent<br>Sxpcsu;P<br>'.Jays; | l'J-c.<1.cJ:::er o:t<br>days on<br>a.ar_;::,~c~- | ;JtL""iUJer of<br>days on<br>Cytarabine | N ,cber<br>of<br>da ,s<br>o'1 CZ-<br>en | Any Dose "to:!;-"'-ens." |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XX | xxx/1•1/45 | Ind:.J.ction | | xxx | XXX | xzx | :".:-:::x | x:,,:x | :-::: <b>z</b> x | ZXX | N |

P:io r-ir&n\_ing Not!!:s::

Repec.t for all T-ticttmeht \_g'rou)?s .. :\$'q-\_:ii'+,:, ·-oy. \_'!',r'e;atm&ri.t -g'±:ouPr-:•:Site· and patient

2-0: aru llarc:
Listing Source:

Dae: \_\_e''''''-''--e.\_:

Page x of Y

### :Sisting 16.2.14 Efficacy pa.:::t

TreatBent g:::-oup: T:::eatment |

| Site | Patie:t<br>/Sex/Age | Race | Achieved<br>C?,? CRi?<br>Cor.,pos:i.te<br>:R? | Dead? | ?rirr,ary ca;se o-f: death | st,,;dy<br>day of<br>Death | Last<br>study<br>day of<br>fol lot, -<br>up | sve:1::<br>T:::-ee? | Study day<br>to which<br>pac:ien::<br>experiewced<br>e-Jerct free | Leukecnia<br>Tree? | St:_;,dy day<br>to c,·h.i.c::',<br>patient<br>expor:;< | ?,elapse? | Stsdy day<br>to K:lich<br>patiecic:<br>experier:ced<br>relapse |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xx | xx;-:/l-1I45 | xxz | t:/i'i/N | xx | XXX | xx | xx | i(X | xx | xx | xx | xxz | xzx |

tro:9":c'ariimi:r1 r.·1'Tote\_S2:

Repeat for 'a\_U:. Tieatrhent -; rroups. Sort by Treatn\en'::. -<; rro}. IP -. "o.i\_te::\_and pa,\_:ti'e:nt Prograr; i. t-::ane:
Listing Sou:::-ce:

rege z of y

## ::.,ist::.ng 2.6.2.15 Efficacy pa:::-t 2

Treatzr:.er,t <a href="mailto:groc19">groc19</a>: Treat:nern::

| Site | 22::ient<br>/Sex/Age | Race | CR? CR<br>Ccr:',posite<br>C?.? | Dead? | ?rirr,ar:,,<br>ca'-lse o:'.<br>de, -:::h | St:,;dv<br>day of<br>Geatr', | Last<br>sc:idy<br>day of<br>:Ec-2.lo:: | Necc.trophil ?.ecovery? | S':cldy day ".::o whic:: patient ex:_::,erienced ne trophil | ?la-:::elec.<br>Reco-very? | St",dy day to whict: patient |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | x;,;x/1•1/45 | ::: <b>xx</b> | Nit-:/::-; | :-::X | xx | xx | ;.:p<br>xx | XX | reco,ser.'i | xx | platelet<br>receve:::-z |

?r\_ogranuni:ri'g Notes-;
Repeat '.for a.l.l T-l::eatmE'nt grpUps;;;\_ Sod: bj. T,ieatment gr-tiuP site iind patient
?rogram Name:
Lis;:ing Source:

Date Genera-:::ed:

?age ;<:of y

#### List:ir.g 16.2.:: o AC:verse s-,,en;::s Safety ?opu.latin7

Treatment g:::ou:e : Treat.:ne;;t

| Site | ?atier::t<br>/Sex/Age/<br>?ace | Systecci O:::ga.;,. Class/<br>Preferreci Ter::rJ<br>Ver:Oati:7, :2J | Cc ':'i e S,::q:, Date (day'-'.b) Time/ Juratio::c ,da_ys: | <u>ca-r&gt;…n</u><br>E:nergent? | AE is due to<br>:ir::der2-ying dc_sease or<br>ether drs.1gs? | Probable Sh, -1-a causeci. AS? | Action 'laker; with stuciy drog [c; | Oc:.tcose | NC!<br>CTCAE<br>Gracie | SA2 |
|---|---|---|---|---|---|---|---|---|---|---|
| xx | xxx/l•l/45/<br>xx:-: | xx>:xx:-:x,::,;;,::zxx: <xxx,::x ::-:xxxx;:::,::x;:,:x;:,:x;:zz="" <="" td="" x:,::;o:xx::*:xx,::x;::,::xxxx=""><td>(xx'&gt;<br/>H ;i·/,I•:</td><td>No</td><td>Yes</td><td>Yes,</td><td>XXX</td><td>Re-<br/>solved</td><td></td><td>: o</td></xxx,::x> | (xx'><br>H ;i·/,I•: | No | Yes | Yes, | XXX | Re-<br>solved | | : o |
| | | XXXXXXXX;ZZXXXZXXZX XX:O:XXXXXXXXXXXXXXX X;;;;XXX;-:XXX XX;;;;XX:*:/ | (xx) E: rv;;;: /xx DJId•.r v.·, (xx)/ DD)E,JMYYY'i.' (xx) /xx | Yes | No | No | xxx:-: | 3'ata:. | 5 | ··es |
| | XXX | $\begin{aligned} &\text{xx:-:,:-;xx;, zxxzz:-:x:;,x:-:xx} \\ &\text{;,:::,::xxxxxxzzx:-:xx:,:xxx/} \\ &\text{xxxxx;-:x.:-:x:{xxx;*:x}} \end{aligned}$ | DDMMMYYY·::··<br>{xx)/<br>Or.going | Yes | Yes | Yes,<br>o.a.c"• c, | ZXXX | Re-<br>solved<br>h·ith<br>sequela<br>e | 3 | Ne |

<sup>[</sup>a] Coded using MedDRA Dictionary (Version xx.xx:

Progr, -arorrii:rig, - 1:fote8:
-Repeat:", -:£'..or: \_all 'tt,E!at;, i ht',g\_roups, sQ\_\_i,t>by. T,reatment:, 9±'(',ll,fF, -- i:te', \_-pai-i,mt', .:sta\_rt ',da\_te .an,a. SOG:
F-or: 'ACtion: 'tak,en',', ith ...study, 'drug,\_\_,-l s.t;, l\_l dru\_gs: tha\_t 'app;y;, i\_ arae'.ff.:th\_\_.pr b:& lee\_s\_t;u,\_dy:drug - 'caused :AE coiu,-un.
:7his 1-is\_ting includes:.,a.l\_l ,AEs:\_captured i\_n the. study, suc\_h as -p\_r\_e-trea:tm nt..P.Es:?r:ogram Na:ne:
Date Gener2ted:

Listing Source:

Page x of

b] Relative to ::he day of randocnizaL.on

Delete: :'Jote to Programmer: Repea'.:. for all T.:::-eatment gro,..ps. Sort b::,r Treatcc,ent group, site, pac.ient, start dc.te and S.JC. Fo.:::- Action: taken with study, drc.;g, list all circug that apply, sa.me ...;ith probable study dirug ca.t..sed AE colu...,«n. Note to Prag ammer: This list.:i.r:g includes al ;:..Es ca.pts1red in s;:he study, such a.s pre-t::-:eac:ment AEs. Footr, ote: :a Coded using t edD?A!)ictionary Ve.::-sior: :<x.x::-:) [b] Relative to he day of rarrdorr, ization Listing 16 ..c..18 Adve::-:se E;rer,ts ca,:;sir,g Ir,terr,.1ptior. ::rom St: ;dy ':::rea::::-,e::t Safety Po;n,;lation Delete: Note to Programm.er: Repeat fc::: all Treatmer, t gro; 1ps. Sort 10,... ?reatc; te::t groc, p, site, pc.tier.t, stc.rt date a:..d SOC. ?o:r Accier: taker., v.;ith study, drug, list all cirugs t:'lat apply, sa,;:e \\*;ith pro:Oa::)le study, d.::-ug caused AE col:..1...Tfl.!7.. rote to 2:::cg a.mrner; This listing includes all A:Ss capt., 1red in ::.he study, sc.:ch as pre-treatrr.er,t AEs, Footr:ote: :a Coded using MeciDRA Dictiona.c" {Ve:::-sic:i ;o:. xxJ [bJ Relc.ti,,e to he day cf ::-:ar'.dosization Lis ting 16. . 1.9 Adverse Events :::ausing Dose Reciu.ction £rorn St"J.•:iv ?reat:r.ent Safety ?opu.lat::.on De2-ete: l ote to ?:::ogra=e::-:: Repeat for c.ll Treatment gro;;,ps. So:::t by Trea::.;nent group, site, patier.t, start date and So::... For Action ta;:en with study, drug, list all drugs that apply, sa;;;-,e ,,,,i::h probable study drug caused AE colu.:::-..rl. Note to ?:::cg arr --:-er: This listing i.ncludes c.ll. AEs captu:::ed i::: the study, s...-.ch as pre-t:::eatment ?.Es. Foctr,,ote: [a Coded using 1%ciDR.A Dictionary \'.Te:rsi0n xx.xx) [bJ Relative tc he day of rar-.domization Treatmen-c-Re::.ateC Adverse Eve;. s Causing Dose Reductior: :Eron Study Treatment Safety Populatior:. Listing 16. . 20 Delete: Note to Pii-ogiiiias,-neir, ?,epec.t for all Treatment ;-roups, Soirt by ':'reatiner.c: giroup, site, patient, stc.:rt date and s-ix.iii. For P.ction t.-'-"ken :,;;;..th stLldy, drug, list all drugs tr',at apply, s2.ccte with ;,;roDable study dru.g caused AE colu..-n.n.

Note to Prog a:r-.:ne:r: This listir1g r,cludes c.ll .n.ss capt.c:red in the study, such as pre-treatrn.ent AEs.

Foo.:.ncte: [a Coded using ::--led ?.A ictior,ary (Ve::-sicc. :<:x.xx)

.o: Relati:re to he day of rando:nizat or:

Ad,rerse :::venc:s Causir,g Discontir.uat:ion f.:::o;;r, Study T.:::-eatmer.t Safety Population

Repe ': fc-::: the £ollowi::1g disp:avs:

List r.g 2.6...'..l.i

## Listing 16.2.21 Serious Adont se Eve:it.s

#### \$af'a+.v ::. :::.u' a-...: "'

| <u>Ireat me</u><br>Site | <u>go'-' p: Treat.:</u> <u>p</u> /Sex/Age/ Race | <pre>lent System Organ C.1.ass/ Preferreci Term/e:cbatir:, :a;</pre> | Sta:::t Date (day.\) Tiffie Stop Date (day; [b) Tiffie/ D -C-ac-'v' (day_s) | <u>'I.i.ae</u> ,<br>:-cc.e ge, | AE is due to <u>F.e</u> disease or <u>C</u> | =':cobao:.e<br><u>\$rI-'I'</u> :<br>cac:sed AE? | Action<br>Taken<br>wit!"':<br>St.Ll.dy<br>drug | Ou.tcorr,e | NC:-<br>CTCAS<br>Grade |
|---|---|---|---|---|---|---|---|---|---|
| xx | xxx/1•'./45/<br>xxx | xxx:,;:xz:- x:-:zxxx;,:xxxxx<br>xxxx:o:;,;:x:-:xxxxvxx/<br>xxxxz;;:xxxxx;,::::x/ | iJD:":c"J1'lvvvy<br>(z :)<br>'-E':M"-'<br>-' <d\imh\'v'fv< th=""><th>r;o</th><th>':'es</th><th>Yes,<br/>c:2::::- o_,_c</th><th>xx;,:</th><th>Re-<br/>solved</th><th>;</th></d\imh\'v'fv<> | r;o | ':'es | Yes,<br>c:2::::- o_,_c | xx;,: | Re-<br>solved | ; |
| | | <u>vvxx</u> xxxxxxxxxxxx:-:>:x:0;:x/zzvv• v:vxz/ | (ZX) i-i :Mi"'. /xx DDM11i,1YYT (xX)/ D''M:-'\V\"V (XX) /xX | Yes | r;;c | Fi: | ;-:;;;; <b>zz</b> | :atal | 5 |
| ::-:х | X:- <z< td=""><td>xzz:-:zxx;::xzxxzxxx);xx<br/>xxxxxxxxxxx:s:xxxx/<br/>x:-::xxxxxxxxx:s:xxx/</td><td>sIDM!-1lr,, '.:n:)/ Ongoing</td><td>Yes</td><td>Yes</td><td>Yes, "<u>''cc-</u>: ::::::::::::::::::::::::::::::::::</td><td>X:-:XX</td><td>Re-<br/>solved<br/>,-,it ,<br/>sequela<br/>e</td><td>3</td></z<> | xzz:-:zxx;::xzxxzxxx);xx<br>xxxxxxxxxxx:s:xxxx/<br>x:-::xxxxxxxxx:s:xxx/ | sIDM!-1lr,, '.:n:)/ Ongoing | Yes | Yes | Yes, " <u>''cc-</u> : :::::::::::::::::::::::::::::::::: | X:-:XX | Re-<br>solved<br>,-,it ,<br>sequela<br>e | 3 |

<sup>&#</sup>x27;.aj Coded using Me6DRA Dictiona:::-:: (Vel'."sion xx.xx) [bi Relative to the day of l'."ar,dor;-;i::ac.:i.o"

P,rog\_r-a.imni,ng\_N\_oteS:

-?-e\_p at- f\_or a:11 Treatment· gio1lps. \_1fort'"by --\_Treatm,mt,\_-gr,,9up/--Sf t'e-;\_,,\_\_patient, -\_st<(:tt -\_a<i te\_- and, s,ac. F,oi'-,Action taken with study, drug. list all drugs that ,:apply:-;\_--,pame-with pro\_bable s,t"lidY drug caused' AE colµ:inn.

Program Name: Listing Source: Date Gene::-ated:

Page x of y

#### Listing 16.2.22 Laboratory FinCings - Bone Marrow Safety ?op..:.la ion

T:reatmer\_t group: Treat.«ent

| Site | .::atient'<br>/Sex/;:,.ge<br>/Race, | eye.le | ':isit | <u>C"7' e" S"'</u><br>Date (de: [aj | Type of e;,:amination | b.1as::<br>in 3one<br>11arro,,· | .Auer<br>Rods | Respo;:;se |
|---|---|---|---|---|---|---|---|---|
| ZX | :,,,:::x/M/ 45<br>/xxx | Ir,d;_,ct.ion | 3aseline | DJ::01-:'.l'-ri·::·yy ( l) | ::.i:! | xx | xx | |
| | | | x:,x;.: | DD11El::'.Y'-'iY (xx·, | Bi::::_psv | XX | XX | C? |
| | | | | | | | | <u>rO"":-" "" - = -</u><br>remissionj |

[a] Relative to the day of rando:.,ization

Program Name:

Program Name:

Repeat of or vail .T.reat!'n,c;nt groups, Soit oby\_\_.-r-reatni:::ht group, osite, postion"t: :and. "tris:'3.--t"-:

Date Ger, erac;ed;

Progran Nane: Listing Sci..:rcf>.

Page x 8£

#### Listing 16.2.23 Laboratory Fir,dings :-',e,T-atology i>.'itl'. C3C Safety Popula'''.:ion

T:ceat:r,ent group: Treat:Teer;t

| Site | ?atient<br>/Se;z/Pge<br>/?-ace | Cycle | 'hsit | Col2.ection<br>Date !day) [a] | <u>"</u> | W3C | Platelet<br>Cou:-:t | Neutrop::ils Absolate Count (ANC'.) | Seg. Nec,trophils ,/3ands c.:uc-apr.:'s |
|---|---|---|---|---|---|---|---|---|---|
| xx | xxx/'c-1/45<br>/;-:; x | <u>"'ci"-:::r'</u> ,, | Baseline | DDMM'.·IYYYY | xx | | xx | xx | |
| | 7,, 30 | | z:xx | nrn1::,1r-:YYYY (xx) | xx | ZX | xx | xx | xx |

[a] Relative ::.o t:ne Cay of ;:"a:-:cio:mizatiou Pr'cigrammi:r1g Note \_-:-

Repeat-:for al-.l T.reatmefrt groups·, S6it )?Y.' Trea:t:inib:f:.. 9":Coup, site, patiei-rt·k:Ud 'Visit. Date Generated:

Prograrr: Kame: Listir,g- Source:

Page x o.:'

#### Listing 16.2.24 Laborato::-y Fir, dir, gs - Coag, ...1.latior, Safet.,, ?opulation

T:::eatment group: Treat::1eict:

| Site | ?atient<br>/Sex/Age<br>/Race | Cycls | VISI"C | :::o.llection Date (day)[a] | An,∷i-factor<br>xa | ?1' | aP:T | :NR | t ····' 0·vse:-::. | D-diner |
|---|---|---|---|---|---|---|---|---|---|---|
| xx | xxx/M/45<br>/xxx | , <u>na'" : GY</u> . | saselh1e | <u>o::-:u</u> | XX | ;n: | xx | X:-: | ;=::,: | :•:X |
| | / XXX | | X: <xx< td=""><td>1.;C;,;;,:: ffYYY (<b>xx</b>)</td><td>XX</td><td>XX</td><td>xx</td><td>xx</td><td>x:;:</td><td></td></xx<> | 1.;C;,;;,:: ffYYY ( <b>xx</b> ) | XX | XX | xx | xx | x:;: | |

'a· Relative to the da:,r ::Jf Yandomizatior, P:rog'rar!ITtiTlg'-) \_O\_teS·\_:

Repeat Ioc-all· Treatment g·roups. Sort by\_. 7-reatm8nt··g:fo\_up, site;:\_-,pa:t\_i&nt-"--arid visit. ?Ycgram Name:

Lis-::ing Source:

Page x of

# :;;,isti:.:::g 16.2.25 Laborato;:"y ?i:::dings - Sers,: Che:r,istry ?art Safety i?opulatior:.

Treat:.,erit 9 £ou\_p: Treat,11ent l

| Site | Patient<br>/Sex/Age<br>/Race | Cycle | Visit | Collectior. Date (day) taJ | A'b·L7I:" | Tor:al<br>?:::-otein | Total<br>Bilirubi::-i | Blood<br>Drea<br>Nitrogen | Seru.o-n<br>C.r-eatin<br>-ine | Sodiu."'.1 | Pot-<br>assiw-:-, |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xx | xxx/?:-5/45<br>/ xxx | Ir:.di:_ction | Baseline | DD:"IMII:YYYY /I) DDMMNYYYY (J'.X) | xx<br>xx | xx<br>:,:x | xx<br>xx | ;,c;x<br>×× | xx | xx<br>xx | xx<br>xx |

[a] Relative to the day of rando: Ttiza-::ion  $PrOgr\cdot airiJr$ ,.it  $g\cdot$  Notes.:

Repeat: for::a11 •'.l'Teat.-nent groups:. •\_S6\_.rt)i::{,::Treatmerit group,::si-.t.e,::patient.-an,ct: vi.\_S.ft,...

Date Generated:

Program Narae: Listi:1g Sot.:..rce:

Page x of

# Listing ::\_6.2.26 Laboratory Findings Serum Cherr.istry ?art 2 Safety Pop,.:lation

Treatment 9-ro;i:9: Treat:, lent 1

| Site | Patient<br>/Sex/Age<br>/ ace | Cycle | \:.'csit | L/''' '' <u>i -</u> ,<br>Cate :'daJ) [a] | Calciur:: | .Dlkaline<br>Phosphatase | ::Jric<br>Ac.id | SGOT<br>/AST | SG?T<br>{r.L | 1DE |
|---|---|---|---|---|---|---|---|---|---|---|
| xx | xxx/:-1/ 45<br>/xx:-: | <u>'; o</u> | 3ase.line | om,n,1t,1YYYY ( l) | xx | xx | xx | xx | X:-:: | xx |
| | /AA | | xxxx | DD1•ltfc'.,JYYYY {xx) | xx | XX | x;,:; | xx | xx | xx |

[a] Re.1.ati·v·e to the Cay of randorr:.izatior.

P,io\_g\_timrilin\_g\_-Nbt:eS'!

Rei,e"ci't-£0'1'.' :all "freatment groups.-. ·sort by\_ Treatment .\_grcup\_, s-ite", p-2.tient aii.d· visit.

Prograr,, Name: :Jate Generated: Page x of y

Listing Source:

List in; 1E.2.27 i??(listing Safety ?opulation

T:reat .er.t g:roup: Treatment

| Site Patient/Age/Sex Visit Date (d2y) PK Parar:sete:r Pf. value | | ст, с <u>5.10ар</u> . 17 санист | | | | |
|---|---|---|---|---|---|---|
| a | Site | Patient/Age/Sex | Visit | Date (d2y) | PK Parar:sete:r | Pf. value |
| | | | | а | | |
| zx xzx/xz/F zx zz XX xx | zx | xzx/xz/F | ZX | | XX | xx |

2age x of

# Listing 16.2.28 Vital Signs Safety Population

s'reat:;1e:1t group: T:::eatment

| Site | ?atient Visi;:: /Sex/Age /Race | Date Time (day) '.a] | Systolic BP<br>чы <u>-</u> g: | Diase:olic 32<br>:rmn :-tg) | 'leart Rate<br>(beat/min) | Weight<br>(kg) | Eeight (cm) |
|---|---|---|---|---|---|---|---|
| xx | xxx/1-1/4.S xx :x:,:xx<br>/xxx | JJMMMY.Y:.y HE:ME (xx) | xxx | XXX | xx | xx | xx |

[a] Relative to the dc.y of .::ar,dorcization
Pr69'faTiliiling,-Not'e,'s::

1<:epeat £cr\_,--E.ll T.teatment' gl:'o\_ups\_sOrt by Tie:a:tment:\_g,:i.:-Oijp, 'sfre:, pati'-et-it and: vis-it.

Da"'.:e Generated:

Page x of Y

#### List.ir,g 16 2.29 ECG ?,esu ts Sa::"ety Pope::ation

Treatment group: Treatme t

| | itment group: 176 | | | | |
|---|---|---|---|---|---|
| | s.::.,tePatient | Visit | .i".ssessnent:: | ECG | Z:ny clinically |
| | /Sex/Age | | Date Tir;-,.e | performed? | sigr,.ificant |
| | /?-ace | | (da_;[) taJ | | "br,or:na2-i t::ies? |
| СХ | xxx/t,;/45<br>/xxx | xxx | DDMMMY<br>HH:YJM xx;· | y,33 | Yes |
| | | XX}'. | DDMMMY YY<br>HH:r1M x:-:' | i'io, ?artial<br>refusal | |
| ХХ | xxx/F/45<br>/:-:xx | xx:,: | DDMMI·1YY'!."Y<br>H2:t1M (:-:x) | ::es | -Jo |
| | | XX}: | DDMM.lY:YYY<br>HE.!"iM (:<:x) | Yes | No |

L.stirrg Sou:::ce:

?age x of Y

## :ist.'.r1g 16.2.30 ?hysica2. Examination ?,esult.s Safety Population

Treat.me21t. g:::-oup: Treatment 1

| Site | ?atient<br>/Se:-:/Age<br>/Race | Visit | Assessrrcent Date (day) [a] | Time | Was<br>done? | Body<br><b>Syste2</b> .<br>Examined | ?esults Normal<br><u>o Ah''''O'''''''T'2 7?</u> | Specify if J.:bnormal |
|---|---|---|---|---|---|---|---|---|
| x: | X)'.X/M/45 | 3aS8line | DDIC:MMYYYY HH:t1!-'I | (xx) | Yes | Cardio,-asc | ':Jo:::mal | |
| | /,-:xx | | | , | | ular | | |
| | | | | | | RepiratcJr. | Ab:r;orr,al | ·,•:•::-:X |
| | | | | | | Gastroir,te<br>stinal | ?,JC:::-:na; | |
| | | | | | | Skin<br>(0-ther | :,Jormal | |
| | | | | | | t:l.a:1<br>pri:;;-,.ar | | |
| | | | | | | site o infect on} | | |
| | | | | | | :'luscc.:losh:e<br>let.al | No:::r:2 | |
| | | | | | | E'''or-:,, | '•,:o:::rr,a- | |
| | | | | | | Ne·ccrolcgic | :-Jormal | |
| | | | | | | al | | |
| | | | | | | HEEIsT | Jo.::-sal | |
| | | | | | | Genitourin | No:::mal | |
| | | | | | | ary | | |
| | | Wee:-: x | "DEMMYYYY .EE: 111":: | (v: :) | No | i one | | |

[a] ?elative to the day of rando:nization

Progr, amtr, i-rig' Jfotes:

-Repeat\_-:fcr,\_ ll T\_r,eatme,nt' -= ups.\_'S $\Diamond$ -r-t::- y/I',f "? rnent -\_-group, site pat,ieiit- and ,vi\_sit\_.  $\Diamond$ -fl- Y\_::ptes\_e\_nt abTlortnal bO'dy s:/stems'. If all body systems are,normal at -a visit;. output '\_None'--<-i\_n,-\_Body System iTonorw..a:Uti•es-,cc-lurtm. for the visit-.

... oa.c.-" Ne.me.
Listing Source: Date Generated: Page z of y